CLINICAL TRIAL: NCT01986881
Title: Randomized, Double-Blind, Placebo-Controlled, Parallel-Group Study to Assess Cardiovascular Outcomes Following Treatment With Ertugliflozin (MK-8835/PF-04971729) in Subjects With Type 2 Diabetes Mellitus and Established Vascular Disease, The VERTIS CV Study
Brief Title: Cardiovascular Outcomes Following Ertugliflozin Treatment in Type 2 Diabetes Mellitus Participants With Vascular Disease, The VERTIS CV Study (MK-8835-004)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 8835-004; 2013-002518-11 (EudraCT Number); B1521021 (Other: Pfizer Protocol Number)
Record Dates: First submitted 2013-11-12; First posted 2013-11-19 (Estimated); Results first posted 2021-02-15 (Actual); Last update posted 2022-09-23 (Actual); Status verified 2022-09

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — ertugliflozin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Ertugliflozin, 15 mg (Experimental): Ertugliflozin 15 mg administered orally once daily for up to approximately 6 years
  Interventions: Drug: Ertugliflozin; Drug: Glycemic Rescue
- Ertugliflozin, 5 mg (Experimental): Ertugliflozin 5 mg administered orally once daily for up to approximately 6 years
  Interventions: Drug: Ertugliflozin; Drug: Placebo; Drug: Glycemic Rescue
- Placebo (Placebo Comparator): Matching placebo to ertugliflozin administered orally once daily for up to approximately 6 years
  Interventions: Drug: Placebo; Drug: Glycemic Rescue

INTERVENTIONS:
Drug: Ertugliflozin — Oral, once daily, for up to approximately 6 years
  Other Names: MK-8835, PF-04971729, Steglatro
  Arms: Ertugliflozin, 15 mg; Ertugliflozin, 5 mg
Drug: Placebo — Matching placebo to ertugliflozin administered orally, once daily, for up to approximately 6 years
  Arms: Ertugliflozin, 5 mg; Placebo
Drug: Glycemic Rescue — Doses of background anti-hyperglycemic agents (AHA), medications will be required to be held constant in all participants enrolled for the initial 18 weeks of the trial with 2 exceptions: First, participant will be prescribed glycemic rescue therapy if they meet specific, progressively more stringent, glycemic thresholds based on repeated, confirmed fasting plasma glucose (FPG) measured at a central laboratory. Second, a participant experiencing clinically significant hypoglycemia according to the investigator at any time during the trial is permitted to have the dose of appropriate background AHA (e.g., insulin, sulfonylurea [SU], glinide) reduced or discontinued as per the judgment of the investigator or the treating physician. Choice and dosing of glycemic rescue will be at the discretion of the investigator or the treating physician consistent with standards of care for management of patients with Type 2 diabetes mellitus (T2DM) within the country of the investigational site.

SUMMARY:
An overall study of the cardiovascular outcomes following treatment with ertugliflozin in participants with type 2 diabetes mellitus (T2DM) and established vascular disease. The main objective of this study is to assess the cardiovascular safety of ertugliflozin. This trial includes 3 pre-defined glycemic sub-studies; 1. In participants receiving background insulin with or without metformin, 2. In participants receiving background sulfonylurea monotherapy, and 3. In participants receiving background metformin with sulfonylurea (all fully-enrolled).

Participants enrolled prior to Amendment 1 were in the overall study as well as a sub-study, if they met certain entry criteria. Participants enrolled following the start of Amendment 1 were only enrolled in the overall study. The sub-studies were the initial 18 weeks of the overall study period.

DETAILED DESCRIPTION:
The primary hypotheses for the 4 studies are:

1. Overall Cardiovascular Study:

   The time to first occurrence of the composite endpoint of MACE: cardiovascular death, non-fatal myocardial infarction [MI] or non-fatal stroke in participants treated with ertugliflozin is non-inferior compared to that in participants treated with placebo.
2. The 3 Glycemic Sub-studies:

   1. The mean reduction from baseline in hemoglobin A1c (A1C) for 15 mg ertugliflozin is greater than that for placebo.
   2. The mean reduction from baseline in A1C for 5 mg ertugliflozin is greater than that for placebo.

ELIGIBILITY:
Inclusion Criteria (Overall Cardiovascular Study):

* Diagnosis of T2DM in accordance with American Diabetes Association (ADA) guidelines
* Hemoglobin A1c (A1C) at the start of study participation of 7.0-10.5% (53-91 mmol/mol)
* On stable allowable anti-hyperglycemic agents (AHA) or on no background AHA for at least 8 weeks prior to the study participation
* Body Mass Index (BMI) > or = to 18.0 kg/m^2
* Evidence or a history of atherosclerosis involving the coronary, cerebral or peripheral vascular systems
* There is adequate documentation of the objective evidence that the participant has established vascular disease such as investigational site's medical records, copies of such records from other institutions, or a letter from a referring physician that specifically states the diagnosis and date of the most recent occurrence of the qualifying event(s) or procedure(s).
* Male, female not or reproductive potential, or female of reproductive potential who agrees to be abstinent from heterosexual activity or agrees to use or have their partner use 2 acceptable methods of contraception

Exclusion Criteria (Overall Cardiovascular Study):

* Previous randomization into this trial
* Experiencing a cardiovascular event (myocardial infarction or stroke) or undergoing coronary angioplasty or peripheral intervention procedure between the Screening Visit and randomization
* Undergoing any cardiovascular surgery (valvular surgery) within 3 months of study participation
* Planned revascularization or peripheral intervention procedure or other cardiovascular surgery
* New York Heart Association (NYHA) IV heart failure at study participation
* History of type 1 diabetes mellitus or a history of ketoacidosis

Key Inclusion Criteria for the 3 Glycemic Sub-studies:

1. Insulin With or Without Metformin Sub-study: Stable doses of insulin (>=20 units/day, with variations up to 10% in the daily dose permitted) with or without metformin (>=1500 mg/day) for at least 8 weeks prior to the time of the Screening Visit (V1) and during the period between the Screening Visit (V1) and randomization.
2. Sulfonylurea (SU) Monotherapy Sub-study: Participants receiving a stable dose of SU monotherapy for at least 8 weeks prior to the time of the Screening Visit (V1) and during the period between the Screening Visit (V1) and randomization.
3. Metformin with SU Sub-study: Participants receiving a stable dose metformin (≥1500 mg/day) with a SU for at least 8 weeks prior to the time of the Screening Visit (V1) and during the period between the Screening Visit (V1) and randomization.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8246 (Actual)
Dates: Start 2013-11-04 (Actual); Primary Completion 2019-12-27 (Actual); Study Completion 2019-12-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Background] Cannon CP, McGuire DK, Pratley R, Dagogo-Jack S, Mancuso J, Huyck S, Charbonnel B, Shih WJ, Gallo S, Masiukiewicz U, Golm G, Cosentino F, Lauring B, Terra SG; VERTIS-CV Investigators. Design and baseline characteristics of the eValuation of ERTugliflozin effIcacy and Safety CardioVascular outcomes trial (VERTIS-CV). Am Heart J. 2018 Dec;206:11-23. doi: 10.1016/j.ahj.2018.08.016. Epub 2018 Sep 5. PMID 30290289
- [Derived] Natale P, Tunnicliffe DJ, Toyama T, Palmer SC, Saglimbene VM, Ruospo M, Gargano L, Stallone G, Gesualdo L, Strippoli GF. Sodium-glucose co-transporter protein 2 (SGLT2) inhibitors for people with chronic kidney disease and diabetes. Cochrane Database Syst Rev. 2024 May 21;5(5):CD015588. doi: 10.1002/14651858.CD015588.pub2. PMID 38770818
- [Derived] Pratley RE, Cannon CP, Cherney DZI, Cosentino F, McGuire DK, Essex MN, Lawrence D, Jones PLS, Liu J, Adamsons I, Dagogo-Jack S. Cardiorenal outcomes, kidney function, and other safety outcomes with ertugliflozin in older adults with type 2 diabetes (VERTIS CV): secondary analyses from a randomised, double-blind trial. Lancet Healthy Longev. 2023 Apr;4(4):e143-e154. doi: 10.1016/S2666-7568(23)00032-6. PMID 37003273
- [Derived] Cherney DZI, Cosentino F, Dagogo-Jack S, McGuire DK, Pratley RE, Frederich R, Maldonado M, Liu CC, Pong A, Cannon CP; VERTIS CV Investigators. Initial eGFR Changes with Ertugliflozin and Associations with Clinical Parameters: Analyses from the VERTIS CV Trial. Am J Nephrol. 2022;53(7):516-525. doi: 10.1159/000524889. Epub 2022 Jun 10. PMID 35691283
- [Derived] Segar MW, Kolkailah AA, Frederich R, Pong A, Cannon CP, Cosentino F, Dagogo-Jack S, McGuire DK, Pratley RE, Liu CC, Maldonado M, Liu J, Cater NB, Pandey A, Cherney DZI. Mediators of ertugliflozin effects on heart failure and kidney outcomes among patients with type 2 diabetes mellitus. Diabetes Obes Metab. 2022 Sep;24(9):1829-1839. doi: 10.1111/dom.14769. Epub 2022 Jun 15. PMID 35603908
- [Derived] Wojeck BS, Inzucchi SE, Neeland IJ, Mancuso JP, Frederich R, Masiukiewicz U, Cater NB, McGuire DK, Cannon CP, Yaggi HK. Ertugliflozin and incident obstructive sleep apnea: an analysis from the VERTIS CV trial. Sleep Breath. 2023 May;27(2):669-672. doi: 10.1007/s11325-022-02594-2. Epub 2022 May 20. PMID 35596030
- [Derived] Dagogo-Jack S, Cannon CP, Cherney DZI, Cosentino F, Liu J, Pong A, Gantz I, Frederich R, Mancuso JP, Pratley RE. Cardiorenal outcomes with ertugliflozin assessed according to baseline glucose-lowering agent: An analysis from VERTIS CV. Diabetes Obes Metab. 2022 Jul;24(7):1245-1254. doi: 10.1111/dom.14691. Epub 2022 Mar 29. PMID 35266296
- [Derived] Cherney DZI, Cosentino F, Pratley RE, Dagogo-Jack S, Frederich R, Maldonado M, Liu J, Pong A, Liu CC, Cannon CP; VERTIS CV Investigators. The differential effects of ertugliflozin on glucosuria and natriuresis biomarkers: Prespecified analyses from VERTIS CV. Diabetes Obes Metab. 2022 Jun;24(6):1114-1122. doi: 10.1111/dom.14677. Epub 2022 Mar 28. PMID 35233908
- [Derived] Dagogo-Jack S, Pratley RE, Cherney DZI, McGuire DK, Cosentino F, Shih WJ, Liu J, Frederich R, Mancuso JP, Raji A, Gantz I. Glycemic efficacy and safety of the SGLT2 inhibitor ertugliflozin in patients with type 2 diabetes and stage 3 chronic kidney disease: an analysis from the VERTIS CV randomized trial. BMJ Open Diabetes Res Care. 2021 Oct;9(1):e002484. doi: 10.1136/bmjdrc-2021-002484. PMID 34620621
- [Derived] Cherney DZI, Cosentino F, Dagogo-Jack S, McGuire DK, Pratley R, Frederich R, Maldonado M, Liu CC, Liu J, Pong A, Cannon CP; VERTIS CV Investigators. Ertugliflozin and Slope of Chronic eGFR: Prespecified Analyses from the Randomized VERTIS CV Trial. Clin J Am Soc Nephrol. 2021 Sep;16(9):1345-1354. doi: 10.2215/CJN.01130121. Epub 2021 Jun 18. PMID 34497110
- [Derived] Lingvay I, Greenberg M, Gallo S, Shi H, Liu J, Gantz I. Efficacy and safety of ertugliflozin in patients with type 2 diabetes mellitus and established cardiovascular disease using insulin: A VERTIS CV substudy. Diabetes Obes Metab. 2021 Jul;23(7):1640-1651. doi: 10.1111/dom.14385. Epub 2021 May 5. PMID 33769675
- [Derived] Budoff MJ, Davis TME, Palmer AG, Frederich R, Lawrence DE, Liu J, Gantz I, Derosa G. Efficacy and Safety of Ertugliflozin in Patients with Type 2 Diabetes Inadequately Controlled by Metformin and Sulfonylurea: A Sub-Study of VERTIS CV. Diabetes Ther. 2021 May;12(5):1279-1297. doi: 10.1007/s13300-021-01033-x. Epub 2021 Mar 15. PMID 33721213
- [Derived] Strojek K, Pandey AS, Dell V, Sisson M, Wang S, Huyck S, Liu J, Gantz I. Efficacy and Safety of Ertugliflozin in Patients With Diabetes Mellitus Inadequately Controlled by Sulfonylurea Monotherapy: a Substudy of VERTIS CV. Diabetes Ther. 2021 Apr;12(4):1175-1192. doi: 10.1007/s13300-021-01018-w. Epub 2021 Mar 10. PMID 33694093
- [Derived] Cherney DZI, Charbonnel B, Cosentino F, Dagogo-Jack S, McGuire DK, Pratley R, Shih WJ, Frederich R, Maldonado M, Pong A, Cannon CP; VERTIS CV Investigators. Effects of ertugliflozin on kidney composite outcomes, renal function and albuminuria in patients with type 2 diabetes mellitus: an analysis from the randomised VERTIS CV trial. Diabetologia. 2021 Jun;64(6):1256-1267. doi: 10.1007/s00125-021-05407-5. Epub 2021 Mar 4. PMID 33665685
- [Derived] Cosentino F, Cannon CP, Cherney DZI, Masiukiewicz U, Pratley R, Dagogo-Jack S, Frederich R, Charbonnel B, Mancuso J, Shih WJ, Terra SG, Cater NB, Gantz I, McGuire DK; VERTIS CV Investigators. Efficacy of Ertugliflozin on Heart Failure-Related Events in Patients With Type 2 Diabetes Mellitus and Established Atherosclerotic Cardiovascular Disease: Results of the VERTIS CV Trial. Circulation. 2020 Dec 8;142(23):2205-2215. doi: 10.1161/CIRCULATIONAHA.120.050255. Epub 2020 Oct 7. PMID 33026243
- [Derived] Cannon CP, Pratley R, Dagogo-Jack S, Mancuso J, Huyck S, Masiukiewicz U, Charbonnel B, Frederich R, Gallo S, Cosentino F, Shih WJ, Gantz I, Terra SG, Cherney DZI, McGuire DK; VERTIS CV Investigators. Cardiovascular Outcomes with Ertugliflozin in Type 2 Diabetes. N Engl J Med. 2020 Oct 8;383(15):1425-1435. doi: 10.1056/NEJMoa2004967. Epub 2020 Sep 23. PMID 32966714
- [Derived] Wittbrodt ET, Eudicone JM, Bell KF, Enhoffer DM, Latham K, Green JB. Eligibility varies among the 4 sodium-glucose cotransporter-2 inhibitor cardiovascular outcomes trials: implications for the general type 2 diabetes US population. Am J Manag Care. 2018 Apr;24(8 Suppl):S138-S145. PMID 29693360

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study included participants in 34 countries at 548 study centers (Overall Cardiovascular Study).
Groups:
- Ertugliflozin 5 mg (Overall Cardiovascular Study): Ertugliflozin 5 mg, administered orally, once daily, for up to approximately 6 years
- Ertugliflozin 15 mg (Overall Cardiovascular Study): Ertugliflozin 15 mg, administered orally, once daily, for up to approximately 6 years
- Placebo (Overall Cardiovascular Study): Matching placebo to ertugliflozin administered orally, once daily, for up to approximately 6 years
Period: Overall Study
Arm/Group | Ertugliflozin 5 mg (Overall Cardiovascular Study) | Ertugliflozin 15 mg (Overall Cardiovascular Study) | Placebo (Overall Cardiovascular Study)
Started | 2752 | 2747 | 2747
Treated | 2746 | 2747 | 2745
Participants Enrolled in the Insulin +/- Metformin Glycemic Sub-Study | 348 | 370 | 347
Participants Enrolled in the Sulfonylurea Monotherapy Glycemic Sub-Study | 55 | 54 | 48
Participants Enrolled in the Metformin With Sulfonylurea Glycemic Sub-Study | 100 | 113 | 117
Completed | 2422 | 2401 | 2389
Not Completed | 330 | 346 | 358
Not completed — Death | 228 | 233 | 247
Not completed — Lost to Follow-up | 51 | 44 | 55
Not completed — Physician Decision | 7 | 4 | 6
Not completed — Study Site Terminated by Sponsor | 2 | 2 | 3
Not completed — Withdrawal by Subject | 41 | 60 | 45
Not completed — Subject Moved | 0 | 1 | 0
Not completed — Other | 1 | 2 | 2

BASELINE CHARACTERISTICS:
Population: The analysis population is all randomized participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Ertugliflozin 5 mg (Overall Cardiovascular Study) | Ertugliflozin 15 mg (Overall Cardiovascular Study) | Placebo (Overall Cardiovascular Study) | Total
Number analyzed (Participants) | 2752 | 2747 | 2747 | 8246
Age, Continuous [Mean (Standard Deviation); unit: Years] | 64.3 (8.2) | 64.4 (8.0) | 64.4 (8.0) | 64.4 (8.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 801 | 832 | 844 | 2477
  Male | 1951 | 1915 | 1903 | 5769
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 353 | 347 | 343 | 1043
  Not Hispanic or Latino | 2390 | 2392 | 2399 | 7181
  Unknown or Not Reported | 9 | 8 | 5 | 22
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 13 | 8 | 17 | 38
  Asian | 187 | 149 | 162 | 498
  Native Hawaiian or Other Pacific Islander | 4 | 10 | 15 | 29
  Black or African American | 91 | 75 | 69 | 235
  White | 2390 | 2436 | 2414 | 7240
  More than one race | 67 | 69 | 70 | 206
  Unknown or Not Reported | 0 | 0 | 0 | 0
Fasting Plasma Glucose (FPG) [Mean (Standard Deviation); unit: mg/dL] — Population: The analysis population included all participants with an baseline FPG measurement.
  mg/dL
    number analyzed (Participants) | 2739 | 2737 | 2727 | 8203
    (all) | 176.1 (52.5) | 174.8 (51.6) | 173.6 (49.4) | 174.8 (51.2)
Sitting Systolic Blood Pressure (SBP) [Mean (Standard Deviation); unit: mmHg] — Population: The analysis population included all participants with a baseline SBP measurement.
  mmHg
    number analyzed (Participants) | 2740 | 2741 | 2740 | 8221
    (all) | 133.7 (13.7) | 133.2 (13.8) | 133.1 (13.9) | 133.3 (13.8)
Sitting Diastolic Blood Pressure (DBP) [Mean (Standard Deviation); unit: mmHg] — Population: The analysis population included all participants with a baseline DBP measurement.
  mmHg
    number analyzed (Participants) | 2740 | 2741 | 2740 | 8221
    (all) | 76.8 (8.5) | 76.7 (8.2) | 76.4 (8.7) | 76.6 (8.5)
Body Weight [Mean (Standard Deviation); unit: Kilograms] — Population: The analysis population included all participants with a baseline weight measurement.
  Kilograms
    number analyzed (Participants) | 2750 | 2746 | 2747 | 8243
    (all) | 91.9 (18.4) | 91.6 (18.6) | 91.9 (18.3) | 91.8 (18.4)
Hemoglobin A1C (A1C) [Mean (Standard Deviation); unit: A1C Percentage] — Population: The analysis population included all participants with a baseline A1C measurement.
  A1C Percentage
    number analyzed (Participants) | 2737 | 2737 | 2732 | 8206
    (all) | 8.3 (1.0) | 8.2 (1.0) | 8.2 (0.9) | 8.2 (1.0)
Estimated Glomerular Filtration Rate (eGFR) [Mean (Standard Deviation); unit: mL/min/1.73 m^2] — Population: The analysis population included all participants with a baseline eGFR measurement.
  mL/min/1.73 m^2
    number analyzed (Participants) | 2751 | 2747 | 2747 | 8245
    (all) | 76.0 (20.8) | 76.2 (20.9) | 75.7 (20.8) | 76.0 (20.9)

OUTCOME MEASURES:

1. Primary Outcome: Time to First Occurrence of MACE (Composite Endpoint of Major Adverse Cardiovascular Events [Cardiovascular Death, Non-fatal Myocardial Infarction or Non-fatal Stroke]) (On-Treatment + 365-day Approach) (Overall Cardiovascular Study)
Description: Time to the first occurrence of any of the following adjudicated components of the primary composite endpoint (3-point major adverse cardiovascular events (MACE)): cardiovascular (CV) death (including fatal stroke and fatal myocardial infarction (MI)), non-fatal MI, and non-fatal stroke. The on-treatment approach included confirmed events that occurred between the date of first dose of study medication and the on-treatment censor date. Person-years was calculated as the sum of participants' time to first event or time to censoring (the earliest of participants' end of study date, death date, last contact date, or 365 days after the last dose).
Time Frame: Up to approximately 6 years
Population: The analysis population included all participants who were randomized into the study and who received at least 1 dose of study medication.
Measure: Number; unit: Events per 100 Person-years
Groups:
- All Ertugliflozin (Overall Cardiovascular Study): Ertugliflozin 5 mg or 15 mg, administered orally, once daily, for up to approximately 6 years
Arm/Group | Ertugliflozin 5 mg (Overall Cardiovascular Study) | Ertugliflozin 15 mg (Overall Cardiovascular Study) | Placebo (Overall Cardiovascular Study) | All Ertugliflozin (Overall Cardiovascular Study)
Number analyzed (Participants) | 2746 | 2747 | 2745 | 5493
Events per 100 Person-years | 3.64 | 4.16 | 4.01 | 3.90
Statistical Analysis 1: Comparison: Placebo (Overall Cardiovascular Study) vs All Ertugliflozin (Overall Cardiovascular Study); Test type: Non-Inferiority — 1-sided p-value and the non-inferiority margin is a hazard ratio of 1.3; p < 0.001, Cox Proportional Hazards Model — Model included treatment as an explanatory factor and cohort category as a stratification factor; Hazard Ratio (HR) = 0.97, 95.6% CI 2-sided [0.848 to 1.114]
Statistical Analysis 2: Comparison: Ertugliflozin 15 mg (Overall Cardiovascular Study) vs Placebo (Overall Cardiovascular Study); Test type: Non-Inferiority — 1-sided p-value and the non-inferiority margin is a hazard ratio of 1.3; p = 0.002, Cox Proportional Hazards Model; Model included treatment as an explanatory factor and cohort category as a stratification factor; Hazard Ratio (HR) = 1.04, 95.6% CI 2-sided [0.887 to 1.211]
Statistical Analysis 3: Comparison: Ertugliflozin 5 mg (Overall Cardiovascular Study) vs Placebo (Overall Cardiovascular Study); Test type: Non-Inferiority — 1-sided p-value and the non-inferiority margin is a hazard ratio of 1.3; p < 0.001, Cox Proportional Hazards Model; Model included treatment as an explanatory factor and cohort category as a stratification factor; Hazard Ratio (HR) = 0.91, 95.6% CI 2-sided [0.773 to 1.065]

2. Primary Outcome: Baseline Hemoglobin A1C (A1C) (Insulin With or Without Metformin Add-on Glycemic Sub-study)
Description: A1C is a blood marker used to report average blood glucose levels over prolonged periods of time and is reported as a percentage (%). A1C represents the percentage of glycated hemoglobin. This baseline reflects the Week 0 A1C.
Time Frame: Baseline
Population: The analysis population included all participants who were randomized, participated in the Insulin +/- Metformin Glycemic Sub-study, and had a measurement of the analysis endpoint at Baseline.
Measure: Mean (Standard Deviation); unit: A1C Percentage
Groups:
- Ertugliflozin 5 mg (Insulin +/- Metformin Glycemic Sub-study): Ertugliflozin 5 mg, administered orally, once daily, for up to 18 weeks
- Ertugliflozin 15 mg (Insulin +/- Metformin Glycemic Sub-study): Ertugliflozin 15 mg, administered orally, once daily, for up to 18 weeks
- Placebo (Ins+/-Met Sub-study): Matching placebo to ertugliflozin administered orally, once daily, for up to 18 weeks
Arm/Group | Ertugliflozin 5 mg (Insulin +/- Metformin Glycemic Sub-study) | Ertugliflozin 15 mg (Insulin +/- Metformin Glycemic Sub-study) | Placebo (Ins+/-Met Sub-study)
Number analyzed (Participants) | 348 | 370 | 347
A1C Percentage | 8.45 (0.944) | 8.38 (0.985) | 8.39 (0.928)

3. Primary Outcome: Change From Baseline in Hemoglobin A1C (A1C) at Week 18 - Excluding Rescue Approach (Insulin With or Without Metformin Add-on Glycemic Sub-study)
Description: A1C is a blood marker used to report average blood glucose levels over prolonged periods of time and is reported as a percentage (%). A1C represents the percentage of glycated hemoglobin. This change from baseline reflects the Week 18 A1C minus the Week 0 A1C. A negative number indicates a reduction in A1C level. Participants who met glycemic rescue criteria received glycemic rescue medication. "Excluding Rescue" excluded all data following the initiation of rescue in order to avoid the confounding influence of the rescue therapy.
Time Frame: Baseline and Week 18
Population: The analysis population included all participants who were randomized, participated in the Insulin +/- Metformin Glycemic Sub-study, received at least 1 dose of study medication, and had at least 1 measurement of the analysis endpoint for the specified timepoint(s) from Baseline to Week 18.
Measure: Least Squares Mean (95% Confidence Interval); unit: A1C Percentage
Arm/Group | Ertugliflozin 5 mg (Insulin +/- Metformin Glycemic Sub-study) | Ertugliflozin 15 mg (Insulin +/- Metformin Glycemic Sub-study) | Placebo (Ins+/-Met Sub-study)
Number analyzed (Participants) | 348 | 370 | 347
A1C Percentage | -0.77 [-0.86 to -0.67] | -0.84 [-0.93 to -0.74] | -0.19 [-0.29 to -0.09]
Statistical Analysis 1: Comparison: Ertugliflozin 15 mg (Insulin +/- Metformin Glycemic Sub-study) vs Placebo (Ins+/-Met Sub-study); Test type: Superiority; p < 0.001, cLDA Model — Constrained longitudinal data analysis (cLDA) model with fixed effects for treatment, time, baseline eGFR, stratum, and the interaction of time by treatment. The stratum was (insulin alone or insulin+metformin) and "Time" was a categorical variable; Difference in the Least Squares Means = -0.65, 95% CI 2-sided [-0.78 to -0.51]
Statistical Analysis 2: Comparison: Ertugliflozin 5 mg (Insulin +/- Metformin Glycemic Sub-study) vs Placebo (Ins+/-Met Sub-study); Test type: Superiority; p < 0.001, Constrained longitudinal data analysis — [p-value comment as in outcome 3, analysis 1]; Difference in the Least Squares Means = -0.58, 95% CI 2-sided [-0.71 to -0.44]

4. Primary Outcome: Baseline Hemoglobin A1C (A1C) (Sulfonylurea Monotherapy Add-on Glycemic Sub-Study)
Description: as for outcome 2
Time Frame: Baseline
Population: The analysis population included all participants who were randomized, participated in the Sulfonyl Monotherapy Glycemic Sub-study, and had a measurement of the analysis endpoint at Baseline.
Measure: Mean (Standard Deviation); unit: A1C Percentage
Groups:
- Ertugliflozin 5 mg (Sulfonylurea Monotherapy Glycemic Sub-Study): Ertugliflozin 5 mg, administered orally, once daily, for up to 18 weeks
- Ertugliflozin 15 mg (Sulfonylurea Monotherapy Glycemic Sub-Study): Ertugliflozin 15 mg, administered orally, once daily, for up to 18 weeks
- Placebo (Sulfonylurea Monotherapy Glycemic Sub-Study): Matching placebo to ertugliflozin administered orally, once daily, for up to 18 weeks
Arm/Group | Ertugliflozin 5 mg (Sulfonylurea Monotherapy Glycemic Sub-Study) | Ertugliflozin 15 mg (Sulfonylurea Monotherapy Glycemic Sub-Study) | Placebo (Sulfonylurea Monotherapy Glycemic Sub-Study)
Number analyzed (Participants) | 54 | 54 | 48
A1C Percentage | 8.27 (0.999) | 8.39 (1.019) | 8.21 (1.169)

5. Primary Outcome: Change From Baseline in Hemoglobin A1C (A1C) at Week 18 - Excluding Rescue Approach (Sulfonylurea Monotherapy Add-on Glycemic Sub-Study)
Description: as for outcome 3
Time Frame: Baseline and Week 18
Population: The analysis population included all participants who were randomized, participated in the Sulfonyl Monotherapy Glycemic Sub-study, received at least 1 dose of study medication, and had at least 1 measurement of the analysis endpoint for the specified timepoint(s) at any time from Baseline to Week 18.
Measure: Least Squares Mean (95% Confidence Interval); unit: A1C Percentage
Arm/Group | Ertugliflozin 5 mg (Sulfonylurea Monotherapy Glycemic Sub-Study) | Ertugliflozin 15 mg (Sulfonylurea Monotherapy Glycemic Sub-Study) | Placebo (Sulfonylurea Monotherapy Glycemic Sub-Study)
Number analyzed (Participants) | 55 | 54 | 48
A1C Percentage | -0.91 [-1.17 to -0.65] | -0.78 [-1.06 to -0.51] | -0.56 [-0.84 to -0.27]
Statistical Analysis 1: Comparison: Ertugliflozin 15 mg (Sulfonylurea Monotherapy Glycemic Sub-Study) vs Placebo (Sulfonylurea Monotherapy Glycemic Sub-Study); Test type: Superiority; p = 0.247, cLDA Model — Constrained longitudinal data analysis (cLDA) model with fixed effects for treatment, time, baseline eGFR, and the interaction of time by treatment; Difference in the Least Squares Means = -0.22, 95% CI 2-sided [-0.60 to 0.16]
Statistical Analysis 2: Comparison: Ertugliflozin 5 mg (Sulfonylurea Monotherapy Glycemic Sub-Study) vs Placebo (Sulfonylurea Monotherapy Glycemic Sub-Study); Test type: Superiority; p = 0.063, cLDA model — [p-value comment as in outcome 5, analysis 1]; Difference in the Least Squares Means = -0.35, 95% CI 2-sided [-0.72 to 0.02]

6. Primary Outcome: Baseline Hemoglobin A1C (A1C) (Metformin With Sulfonylurea Add-on Glycemic Sub-study)
Description: A1C is a blood marker used to report average blood glucose levels over prolonged periods of time and is reported as a percentage (%). A1C represents the percentage of glycated hemoglobin. This baseline reflects Week 0 A1C.
Time Frame: Baseline
Population: The analysis population included all participants who were randomized, participated in the Metformin with Sulfonylurea Glycemic Sub-study, and had an assessment for the analysis endpoint at Baseline.
Measure: Mean (Standard Deviation); unit: A1C Percentage
Groups:
- Ertugliflozin 5 mg (Metformin With Sulfonylurea Glycemic Sub-study): Ertugliflozin 5 mg, administered orally, once daily, for up to 18 weeks
- Ertugliflozin 15 mg (Metformin With Sulfonylurea Glycemic Sub-study): Ertugliflozin 15 mg, administered orally, once daily, for up to 18 weeks
- Placebo (Metformin With Sulfonylurea Glycemic Sub-study): Matching placebo to ertugliflozin administered orally, once daily, for up to 18 weeks
Arm/Group | Ertugliflozin 5 mg (Metformin With Sulfonylurea Glycemic Sub-study) | Ertugliflozin 15 mg (Metformin With Sulfonylurea Glycemic Sub-study) | Placebo (Metformin With Sulfonylurea Glycemic Sub-study)
Number analyzed (Participants) | 99 | 113 | 116
A1C Percentage | 8.39 (0.960) | 8.30 (0.963) | 8.27 (0.994)

7. Primary Outcome: Change From Baseline in Hemoglobin A1C (A1C) at Week 18 - Excluding Rescue Approach (Metformin With Sulfonylurea Add-on Glycemic Sub-study)
Description: as for outcome 3
Time Frame: Baseline and Week 18
Population: The analysis population included all participants who were randomized, participated in the Metformin with Sulfonylurea Glycemic Sub-study, received at least one dose of blinded study medication, and had at least one assessment for the analysis endpoint for the specified timepoint(s) at or after Baseline.
Measure: Least Squares Mean (95% Confidence Interval); unit: A1C Percentage
Arm/Group | Ertugliflozin 5 mg (Metformin With Sulfonylurea Glycemic Sub-study) | Ertugliflozin 15 mg (Metformin With Sulfonylurea Glycemic Sub-study) | Placebo (Metformin With Sulfonylurea Glycemic Sub-study)
Number analyzed (Participants) | 100 | 113 | 117
A1C Percentage | -0.89 [-1.06 to -0.71] | -0.98 [-1.14 to -0.82] | -0.23 [-0.39 to -0.06]
Statistical Analysis 1: Comparison: Ertugliflozin 15 mg (Metformin With Sulfonylurea Glycemic Sub-study) vs Placebo (Metformin With Sulfonylurea Glycemic Sub-study); Test type: Superiority; p < 0.001, cLDA Model — [p-value comment as in outcome 5, analysis 1]; Difference in the Least Squares Means = -0.75, 95% CI 2-sided [-0.98 to -0.53]
Statistical Analysis 2: Comparison: Ertugliflozin 5 mg (Metformin With Sulfonylurea Glycemic Sub-study) vs Placebo (Metformin With Sulfonylurea Glycemic Sub-study); Test type: Superiority; p < 0.001, cLDA model — [p-value comment as in outcome 5, analysis 1]; Difference in the Least Squares Means = -0.66, 95% CI 2-sided [-0.89 to -0.43]

8. Secondary Outcome: Time to Occurrence of Cardiovascular (CV) Death or Hospitalization for Heart Failure (HHF) (On-Study Approach) (Overall Cardiovascular Study)
Description: Time to the occurrence of any of the following adjudicated components of cardiovascular (CV) death (including fatal stroke and fatal myocardial infarction (MI)) or hospitalization for heart failure. The on-study approach included confirmed events that occurred between the randomization date and the on-study censor date. Person-years was calculated as the sum of participants' time to event or time to censoring (the earliest of participants' end of study date, death date, or last contact date).
Time Frame: Up to approximately 6 years
Population: The analysis population included all randomized participants.
Measure: Number; unit: Events per 100 Person-years
Arm/Group | Ertugliflozin 5 mg (Overall Cardiovascular Study) | Ertugliflozin 15 mg (Overall Cardiovascular Study) | Placebo (Overall Cardiovascular Study) | All Ertugliflozin (Overall Cardiovascular Study)
Number analyzed (Participants) | 2752 | 2747 | 2747 | 5499
Events per 100 Person-years | 2.36 | 2.33 | 2.66 | 2.34
Statistical Analysis 1: Comparison: Placebo (Overall Cardiovascular Study) vs All Ertugliflozin (Overall Cardiovascular Study); Test type: Superiority; p = 0.108, Cox Proportional Hazards Model; Model included treatment as an explanatory factor and cohort category as a stratification factor; Hazard Ratio (HR) = 0.88, 95.8% CI 2-sided [0.750 to 1.034]
Statistical Analysis 2: Comparison: Ertugliflozin 15 mg (Overall Cardiovascular Study) vs Placebo (Overall Cardiovascular Study); Test type: Superiority; p = 0.150, Cox Proportional Hazards Model; Model included treatment as an explanatory factor and cohort category as a stratification factor; Hazard Ratio (HR) = 0.88, 95.8% CI 2-sided [0.725 to 1.057]
Statistical Analysis 3: Comparison: Ertugliflozin 5 mg (Overall Cardiovascular Study) vs Placebo (Overall Cardiovascular Study); Test type: Superiority; p = 0.188, Cox Proportional Hazards Model; Model included treatment as an explanatory factor and cohort category as a stratification factor; Hazard Ratio (HR) = 0.89, 95.8% CI 2-sided [0.735 to 1.068]

9. Secondary Outcome: Time to Occurrence of Cardiovascular Death (On-study Approach) (Overall Cardiovascular Study)
Description: Time to the occurrence of cardiovascular (CV) death (including fatal stroke and fatal myocardial infarction (MI)). The on-study approach included confirmed events that occurred between the randomization date and the on-study censor date. Person-years was calculated as the sum of participants' time to CV death or time to censoring (the earliest of participants' end of study date or date last known to be alive).
Time Frame: Up to approximately 6 years
Population: The analysis population included all randomized participants.
Measure: Number; unit: Events per 100 Person-years
Arm/Group | Ertugliflozin 5 mg (Overall Cardiovascular Study) | Ertugliflozin 15 mg (Overall Cardiovascular Study) | Placebo (Overall Cardiovascular Study) | All Ertugliflozin (Overall Cardiovascular Study)
Number analyzed (Participants) | 2752 | 2747 | 2747 | 5499
Events per 100 Person-years | 1.77 | 1.74 | 1.90 | 1.76
Statistical Analysis 1: Comparison: Placebo (Overall Cardiovascular Study) vs All Ertugliflozin (Overall Cardiovascular Study); Test type: Superiority; p = 0.385, Cox Proportional Hazards Model; Model included treatment as an explanatory factor and cohort category as a stratification factor; Hazard Ratio (HR) = 0.92, 95.8% CI 2-sided [0.767 to 1.113]
Statistical Analysis 2: Comparison: Ertugliflozin 15 mg (Overall Cardiovascular Study) vs Placebo (Overall Cardiovascular Study); Test type: Superiority; p = 0.417, Cox Proportional Hazards Model; Model included treatment as an explanatory factor and cohort category as a stratification factor; Hazard Ratio (HR) = 0.92, 95.8% CI 2-sided [0.739 to 1.139]
Statistical Analysis 3: Comparison: Ertugliflozin 5 mg (Overall Cardiovascular Study) vs Placebo (Overall Cardiovascular Study); Test type: Superiority; p = 0.494, Cox Proportional Hazards Model; Model included treatment as an explanatory factor and cohort category as a stratification factor; Hazard Ratio (HR) = 0.93, 95.8% CI 2-sided [0.750 to 1.154]

10. Secondary Outcome: Time to First Occurrence of the Renal Composite: the Composite of Renal Death, Renal Dialysis/Transplant, or Doubling of Serum Creatinine From Baseline (On-Study Approach) (Overall Cardiovascular Study)
Description: Renal composite endpoint was defined as a composite of renal death, renal dialysis/transplant, or doubling of serum creatinine from baseline. The on-study approach included events that occurred between the randomization date and the on-study censor date. Person-years was calculated as the sum of participants' time to first event or time to censoring (the earliest of participants' end of study date, death date, or last contact date). The on-study approach included events that occurred between the randomization date and the on-study censor date.
Time Frame: Up to approximately 6 years
Population: The analysis population included all randomized participants.
Measure: Number; unit: Events per 100 Person-years
Arm/Group | Ertugliflozin 5 mg (Overall Cardiovascular Study) | Ertugliflozin 15 mg (Overall Cardiovascular Study) | Placebo (Overall Cardiovascular Study) | All Ertugliflozin (Overall Cardiovascular Study)
Number analyzed (Participants) | 2752 | 2747 | 2747 | 5499
Events per 100 Person-years | 0.87 | 0.98 | 1.15 | 0.93
Statistical Analysis 1: Comparison: Placebo (Overall Cardiovascular Study) vs All Ertugliflozin (Overall Cardiovascular Study); Test type: Superiority; p = 0.081, Cox Proportional Hazards Model; Model included treatment as an explanatory factor and cohort category as a stratification factor; Hazard Ratio (HR) = 0.81, 95.8% CI 2-sided [0.630 to 1.036]
Statistical Analysis 2: Comparison: Ertugliflozin 15 mg (Overall Cardiovascular Study) vs Placebo (Overall Cardiovascular Study); Test type: Superiority; p = 0.258, Cox Proportional Hazard Model; Model included treatment as an explanatory factor and cohort category as a stratification factor. Renal; Hazard Ratio (HR) = 0.85, 95.8% CI 2-sided [0.638 to 1.137]
Statistical Analysis 3: Comparison: Ertugliflozin 5 mg (Overall Cardiovascular Study) vs Placebo (Overall Cardiovascular Study); Test type: Superiority; p = 0.065, Cox Proportional Hazards Model; Model included treatment as an explanatory factor and cohort category as a stratification factor; Hazard Ratio (HR) = 0.76, 95.8% CI 2-sided [0.568 to 1.028]

11. Secondary Outcome: Time to First Occurrence of MACE Plus (Composite Endpoint of Cardiovascular Death, Non-fatal Myocardial Infarction, Non-fatal Stroke or Hospitalization for Unstable Angina) (On-Study Approach) (Overall Cardiovascular Study)
Description: Time to the first occurrence of any of the following adjudicated components 4-point MACE: cardiovascular death (including fatal stroke and fatal myocardial infarction), non-fatal myocardial infarction, non-fatal stroke, and hospitalization for unstable angina pectoris. The on-study approach included confirmed events that occurred between the randomization date and the on-study censor date. Person-years was calculated as the sum of participants' time to first event or time to censoring (the earliest of participants' end of study date, death date, or last contact date). The on-study approach included events that occurred between the randomization date and the on-study censor date.
Time Frame: Up to approximately 6 years
Population: The analysis population included all randomized participants.
Measure: Number; unit: Events per 100 Person-years
Arm/Group | Ertugliflozin 5 mg (Overall Cardiovascular Study) | Ertugliflozin 15 mg (Overall Cardiovascular Study) | Placebo (Overall Cardiovascular Study) | All Ertugliflozin (Overall Cardiovascular Study)
Number analyzed (Participants) | 2752 | 2747 | 2747 | 5499
Events per 100 Person-years | 4.42 | 4.67 | 4.92 | 4.54
Statistical Analysis 1: Comparison: Placebo (Overall Cardiovascular Study) vs All Ertugliflozin (Overall Cardiovascular Study); Test type: Superiority; p = 0.183, Cox proportional hazards model — Hazard ratio, CI, and 2-sided p-value comparing All Ertugliflozin versus Placebo, based on the stratified Cox proportional hazards model that included treatment as an explanatory factor and cohort category as a stratification factor; Hazard Ratio (HR) = 0.92, 95% CI 2-sided [0.823 to 1.038]
Statistical Analysis 2: Comparison: Ertugliflozin 15 mg (Overall Cardiovascular Study) vs Placebo (Overall Cardiovascular Study); Test type: Superiority; p = 0.450, Cox Proportional Hazards Model; Model included treatment as an explanatory factor and cohort category as a stratification factor; Hazard Ratio (HR) = 0.95, 95% CI 2-sided [0.831 to 1.086]
Statistical Analysis 3: Comparison: Ertugliflozin 5 mg (Overall Cardiovascular Study) vs Placebo (Overall Cardiovascular Study); Test type: Superiority; p = 0.123, Cox Proportional Hazards Model; Model included treatment as an explanatory factor and cohort category as a stratification factor; Hazard Ratio (HR) = 0.90, 95% CI 2-sided [0.785 to 1.029]

12. Secondary Outcome: Time to First Occurrence of Fatal or Non-fatal Myocardial Infarction (On-Study Approach) (Overall Cardiovascular Study)
Description: Time to First Occurrence of Fatal or Non-fatal Myocardial Infarction. The on-study approach included confirmed events that occurred between the randomization date and the on-study censor date. Person-years was calculated as the sum of participants' time to first event or time to censoring (the earliest of participants' end of study date, death date, or last contact date).
Time Frame: Up to approximately 6 years
Population: The analysis population included all randomized participants.
Measure: Number; unit: Events per 100 Person-years
Arm/Group | Ertugliflozin 5 mg (Overall Cardiovascular Study) | Ertugliflozin 15 mg (Overall Cardiovascular Study) | Placebo (Overall Cardiovascular Study) | All Ertugliflozin (Overall Cardiovascular Study)
Number analyzed (Participants) | 2752 | 2747 | 2747 | 5499
Events per 100 Person-years | 1.55 | 2.00 | 1.70 | 1.77
Statistical Analysis 1: Comparison: Placebo (Overall Cardiovascular Study) vs All Ertugliflozin (Overall Cardiovascular Study); Test type: Superiority; p = 0.676, Cox Proportional Hazards Model; Model included treatment as an explanatory factor and cohort category as a stratification factor; Hazard Ratio (HR) = 1.04, 95% CI 2-sided [0.861 to 1.259]
Statistical Analysis 2: Comparison: Ertugliflozin 15 mg (Overall Cardiovascular Study) vs Placebo (Overall Cardiovascular Study); Test type: Superiority; p = 0.139, Cox Proportional Hazards Model; Model included treatment as an explanatory factor and cohort category as a stratification factor; Hazard Ratio (HR) = 1.17, 95% CI 2-sided [0.949 to 1.451]
Statistical Analysis 3: Comparison: Ertugliflozin 5 mg (Overall Cardiovascular Study) vs Placebo (Overall Cardiovascular Study); Test type: Superiority; p = 0.416, Cox Proportional Hazards Model; Model included treatment as an explanatory factor and cohort category as a stratification factor; Hazard Ratio (HR) = 0.91, 95% CI 2-sided [0.727 to 1.141]

13. Secondary Outcome: Time to First Occurrence of Fatal or Non-fatal Stroke (FNF Stroke) (On-Study Approach) (Overall Cardiovascular Study)
Description: Time to the first occurrence of fatal and no-fatal stroke. The on-study approach included confirmed events that occurred between the randomization date and the on-study censor date. Person-years was calculated as the sum of participants' time to first event or time to censoring (the earliest of participants' end of study date, death date, or last contact date). The on-study approach included events that occurred between the randomization date and the on-study censor date.
Time Frame: Up to approximately 6 years
Population: The analysis population included all randomized participants.
Measure: Number; unit: Events per 100 Person-years
Arm/Group | Ertugliflozin 5 mg (Overall Cardiovascular Study) | Ertugliflozin 15 mg (Overall Cardiovascular Study) | Placebo (Overall Cardiovascular Study) | All Ertugliflozin (Overall Cardiovascular Study)
Number analyzed (Participants) | 2752 | 2747 | 2747 | 5499
Events per 100 Person-years | 0.92 | 1.04 | 0.93 | 0.98
Statistical Analysis 1: Comparison: Placebo (Overall Cardiovascular Study) vs All Ertugliflozin (Overall Cardiovascular Study); Test type: Superiority; p = 0.663, Cox proportional hazards model — [p-value comment as in outcome 11, analysis 1]; Hazard Ratio (HR) = 1.06, 95% CI 2-sided [0.820 to 1.365] — Hazard ratio, CI, and 2-sided p-value comparing All Ertugliflozin versus Placebo, based on the stratified Cox proportional hazards model that included treatment as an explanatory factor and cohort category as a stratification factor
Statistical Analysis 2: Comparison: Ertugliflozin 15 mg (Overall Cardiovascular Study) vs Placebo (Overall Cardiovascular Study); Hazard ratio, confidence interval, and two-sided p-value comparing Ertugliflozin vs Placebo, based on the stratified Cox proportional hazards model that includes treatment as an explanatory factor and cohort category as a stratification factor; Test type: Superiority; p = 0.415, Cox proportional hazards model — A two-sided p-value compared Ertugliflozin vs Placebo, based on the stratified Cox proportional hazards model that included treatment as an explanatory factor and cohort category as a stratification factor; Hazard Ratio (HR) = 1.13, 95% CI 2-sided [0.845 to 1.505]
Statistical Analysis 3: Comparison: Ertugliflozin 5 mg (Overall Cardiovascular Study) vs Placebo (Overall Cardiovascular Study); [analysis description as in outcome 13, analysis 2]; Test type: Superiority; p = 0.953, Cox proportional hazards model — [p-value comment as in outcome 13, analysis 2]; Hazard Ratio (HR) = 0.99, 95% CI 2-sided [0.736 to 1.334]

14. Secondary Outcome: Time to First Occurrence of Hospitalization for Heart Failure (HHF) (On-Study Approach) (Overall Cardiovascular Study)
Description: Time to the first occurrence of heart failure requiring hospitalization (adjudicated). The on-study approach included confirmed events that occurred between the randomization date and the on-study censor date. Person-years was calculated as the sum of participants' time to first event or time to censoring (the earliest of participants' end of study date, death date, or last contact date). The on-study approach included events that occurred between the randomization date and the on-study censor date.
Time Frame: Up to approximately 6 years
Population: The analysis population included all randomized participants.
Measure: Number; unit: Events per 100 Person-years
Arm/Group | Ertugliflozin 5 mg (Overall Cardiovascular Study) | Ertugliflozin 15 mg (Overall Cardiovascular Study) | Placebo (Overall Cardiovascular Study) | All Ertugliflozin (Overall Cardiovascular Study)
Number analyzed (Participants) | 2752 | 2747 | 2747 | 5499
Events per 100 Person-years | 0.75 | 0.72 | 1.05 | 0.73
Statistical Analysis 1: Comparison: Placebo (Overall Cardiovascular Study) vs All Ertugliflozin (Overall Cardiovascular Study); Test type: Superiority; p = 0.006, Cox proportional hazards model — [p-value comment as in outcome 11, analysis 1]; Hazard Ratio (HR) = 0.70, 95% CI 2-sided [0.539 to 0.902]
Statistical Analysis 2: Comparison: Ertugliflozin 15 mg (Overall Cardiovascular Study) vs Placebo (Overall Cardiovascular Study); Test type: Superiority; p = 0.016, Cox Proportional Hazards Model; Hazards model that included treatment as an explanatory factor and cohort category as a stratification factor; Hazard Ratio (HR) = 0.68, 95% CI 2-sided [0.502 to 0.932]
Statistical Analysis 3: Comparison: Ertugliflozin 5 mg (Overall Cardiovascular Study) vs Placebo (Overall Cardiovascular Study); Test type: Superiority; p = 0.028, Cox Proportional Hazards Model; Hazards model that included treatment as an explanatory factor and cohort category as a stratification factor; Hazard Ratio (HR) = 0.71, 95% CI 2-sided [0.524 to 0.964]

15. Secondary Outcome: Time to Occurrence of Death From Any Cause (On-Study Approach) (Overall Cardiovascular Study)
Description: Time to the occurrence of death from any cause. The on-study approach included confirmed events that occurred between the randomization date and the on-study censor date. Person-years was calculated as the sum of participants' time to event or time to censoring (the earliest of participants' end of study date, death date, last contact date, or date last known to be alive. The on-study approach included events that occurred between the randomization date and the on-study censor date.
Time Frame: Up to approximately 6 years
Population: The analysis population included all randomized participants.
Measure: Number; unit: Events per 100 Person-years
Arm/Group | Ertugliflozin 5 mg (Overall Cardiovascular Study) | Ertugliflozin 15 mg (Overall Cardiovascular Study) | Placebo (Overall Cardiovascular Study) | All Ertugliflozin (Overall Cardiovascular Study)
Number analyzed (Participants) | 2752 | 2747 | 2747 | 5499
Events per 100 Person-years | 2.42 | 2.46 | 2.62 | 2.44
Statistical Analysis 1: Comparison: Placebo (Overall Cardiovascular Study) vs All Ertugliflozin (Overall Cardiovascular Study); Test type: Superiority — Hazard ratio, CI, and 2-sided p-value comparing Ertugliflozin vs Placebo, based on the stratified Cox proportional hazards model that included treatment as an explanatory factor and cohort category as a stratification factor. The on-study approach included confirmed events that occurred between the randomization date and the on-study censor date; p = 0.340, Cox proportional hazards model — Hazard ratio, CI, and 2-sided p-value comparing Ertugliflozin vs Placebo, based on the stratified Cox proportional hazards model that included treatment as an explanatory factor and cohort category as a stratification factor; Hazard Ratio (HR) = 0.93, 95% CI 2-sided [0.797 to 1.081]
Statistical Analysis 2: Comparison: Ertugliflozin 15 mg (Overall Cardiovascular Study) vs Placebo (Overall Cardiovascular Study); Test type: Superiority; p = 0.463, Cox Proportional Hazards Model; Model included treatment as an explanatory factor and cohort category as a stratification factor; Hazard Ratio (HR) = 0.94, 95% CI 2-sided [0.784 to 1.117]
Statistical Analysis 3: Comparison: Ertugliflozin 5 mg (Overall Cardiovascular Study) vs Placebo (Overall Cardiovascular Study); Test type: Superiority; p = 0.363, Cox Proportional Hazards Model; Model included treatment as an explanatory factor and cohort category as a stratification factor; Hazard Ratio (HR) = 0.92, 95% CI 2-sided [0.771 to 1.100]

16. Secondary Outcome: Andersen-Gill Model for Total MACE (On-Study Approach) (Overall Cardiovascular Study)
Description: All events (first and recurrent) of the composite of MACE (3-point major adverse cardiovascular events: cardiovascular (CV) death (including fatal stroke and fatal myocardial infarction (MI)), non-fatal MI, and non-fatal stroke) were assessed using Andersen-Gill model. The on-study approach included events that occurred between the randomization date and the on-study censor date.
Time Frame: Up to approximately 6 years
Population: The analysis population included all randomized participants.
Measure: Number; unit: Events per 100 Person-years
Arm/Group | Ertugliflozin 5 mg (Overall Cardiovascular Study) | Ertugliflozin 15 mg (Overall Cardiovascular Study) | Placebo (Overall Cardiovascular Study) | All Ertugliflozin (Overall Cardiovascular Study)
Number analyzed (Participants) | 2752 | 2747 | 2747 | 5499
Events per 100 Person-years | 4.35 | 4.91 | 4.59 | 4.63
Statistical Analysis 1: Comparison: Placebo (Overall Cardiovascular Study) vs All Ertugliflozin (Overall Cardiovascular Study); Test type: Superiority — Ertugliflozin vs Placebo, based on the Andersen-Gill model for the recurrent events at the end of study. The on-study approach includes confirmed events that occurred between the randomization date and the on-study censor date; Hazard Ratio (HR) = 1.01, 95% CI 2-sided [0.898 to 1.131]
Statistical Analysis 2: Comparison: Ertugliflozin 15 mg (Overall Cardiovascular Study) vs Placebo (Overall Cardiovascular Study); Test type: Superiority; Hazard Ratio (HR) = 1.07, 95% CI 2-sided [0.937 to 1.219]
Statistical Analysis 3: Comparison: Ertugliflozin 5 mg (Overall Cardiovascular Study) vs Placebo (Overall Cardiovascular Study); Test type: Superiority; Hazard Ratio (HR) = 0.95, 95% CI 2-sided [0.828 to 1.085]

17. Secondary Outcome: Andersen-Gill Model for All Cardiovascular Death (CV Death) or Hospitalizations for Heart Failure (HFF) (On-Study Approach) (Overall Cardiovascular Study)
Description: All events (first and recurrent) of the composite of CV death and HHF were assessed using an Andersen-Gill model. Person-years were calculated as the sum of time from randomization to end of follow-up. The on-study approach included events that occurred between the randomization date and the on-study censor date.
Time Frame: Up to approximately 6 years
Population: The analysis population included all randomized participants.
Measure: Number; unit: Events per 100 Person-years
Arm/Group | Ertugliflozin 5 mg (Overall Cardiovascular Study) | Ertugliflozin 15 mg (Overall Cardiovascular Study) | Placebo (Overall Cardiovascular Study) | All Ertugliflozin (Overall Cardiovascular Study)
Number analyzed (Participants) | 2752 | 2747 | 2747 | 5499
Events per 100 Person-years | 2.92 | 2.71 | 3.42 | 2.82
Statistical Analysis 1: Comparison: Placebo (Overall Cardiovascular Study) vs All Ertugliflozin (Overall Cardiovascular Study); Ertugliflozin vs Placebo, based on the Andersen-Gill model for the recurrent events at the end of study. The on-study approach included confirmed events that occurred between randomization date and the on-study censor date; Test type: Superiority; Hazard Ratio (HR) = 0.82, 95% CI 2-sided [0.716 to 0.945]
Statistical Analysis 2: Comparison: Ertugliflozin 15 mg (Overall Cardiovascular Study) vs Placebo (Overall Cardiovascular Study); Test type: Superiority; Hazard Ratio (HR) = 0.79, 95% CI 2-sided [0.673 to 0.935] — Ertugliflozin vs Placebo, based on the Andersen-Gill model for the recurrent events at the end of study
Statistical Analysis 3: Comparison: Ertugliflozin 5 mg (Overall Cardiovascular Study) vs Placebo (Overall Cardiovascular Study); Test type: Superiority; Hazard Ratio (HR) = 0.85, 95% CI 2-sided [0.725 to 1.001] — Ertugliflozin vs Placebo, based on the Andersen-Gill model for the recurrent events at the end of study

18. Secondary Outcome: Change From Baseline in Hemoglobin A1C (A1C) at Week 18 - Excluding Rescue Approach (Overall Cardiovascular Study)
Description: as for outcome 3
Time Frame: Baseline and Week 18
Population: The analysis population included all participants who were randomized, received at least one dose of blinded study medication, and had at least one assessment for the analysis endpoint for the specified timepoint(s) at or after baseline.
Measure: Least Squares Mean (95% Confidence Interval); unit: A1C Percentage
Arm/Group | Ertugliflozin 5 mg (Overall Cardiovascular Study) | Ertugliflozin 15 mg (Overall Cardiovascular Study) | Placebo (Overall Cardiovascular Study)
Number analyzed (Participants) | 2745 | 2747 | 2742
A1C Percentage | -0.70 [-0.73 to -0.67] | -0.72 [-0.75 to -0.69] | -0.22 [-0.25 to -0.19]
Statistical Analysis 1: Comparison: Ertugliflozin 15 mg (Overall Cardiovascular Study) vs Placebo (Overall Cardiovascular Study); Test type: Superiority; p < 0.001, cLDA Model; cLDA model with fixed effects for treatment, time, baseline eGFR (continuous) and the interaction of time by treatment; Difference in the Least Squares Means = -0.50, 95% CI 2-sided [-0.55 to -0.46]
Statistical Analysis 2: Comparison: Ertugliflozin 5 mg (Overall Cardiovascular Study) vs Placebo (Overall Cardiovascular Study); Test type: Superiority; p < 0.001, cLDA model; cLDA model with fixed effects for treatment, time, baseline eGFR (continuous) and the interaction of time by treatment; Difference in the Least Squares Means = -0.48, 95% CI 2-sided [-0.53 to -0.44]

19. Secondary Outcome: Change From Baseline in A1C at Week 52 (Overall Cardiovascular Study)
Description: A1C is a blood marker used to report average blood glucose levels over prolonged periods of time and is reported as a percentage (%). A1C represents the percentage of glycated hemoglobin. This change from baseline reflects the Week 52 A1C minus the Week 0 A1C. A negative number indicates a reduction in A1C level. Participants who met glycemic rescue criteria received glycemic rescue medication.
Time Frame: Baseline and Week 52
Population: as for outcome 18
Measure: Least Squares Mean (95% Confidence Interval); unit: A1C Percentage
Arm/Group | Ertugliflozin 5 mg (Overall Cardiovascular Study) | Ertugliflozin 15 mg (Overall Cardiovascular Study) | Placebo (Overall Cardiovascular Study)
Number analyzed (Participants) | 2746 | 2747 | 2745
A1C Percentage | -0.69 [-0.73 to -0.65] | -0.67 [-0.71 to -0.63] | -0.19 [-0.23 to -0.15]
Statistical Analysis 1: Comparison: Ertugliflozin 15 mg (Overall Cardiovascular Study) vs Placebo (Overall Cardiovascular Study); Test type: Superiority; p < 0.001, Constrained Longitudinal Data Analysis; Model included fixed effects for treatment, time, baseline eGFR (continuous) and the interaction of time by treatment; Difference in the Least Squares Means = -0.48, 95% CI 2-sided [-0.54 to -0.43]
Statistical Analysis 2: Comparison: Ertugliflozin 5 mg (Overall Cardiovascular Study) vs Placebo (Overall Cardiovascular Study); Test type: Superiority; p < 0.001, Constrained Longitudinal Data Analysis; Model included fixed effects for treatment, time, baseline eGFR (continuous) and the interaction of time by treatment; Difference in the Least Squares Means = -0.50, 95% CI 2-sided [-0.55 to -0.45]

20. Secondary Outcome: Change From Baseline in A1C at Month 24 (Overall Cardiovascular Study)
Description: A1C is a blood marker used to report average blood glucose levels over prolonged periods of time and is reported as a percentage (%). A1C represents the percentage of glycated hemoglobin. This change from baseline reflects the Month 24 A1C minus the Week 0 A1C. A negative number indicates a reduction in A1C level. Participants who met glycemic rescue criteria received glycemic rescue medication.
Time Frame: Baseline and Month 24
Population: The analysis population included all participants who were randomized, received at least one dose of blinded study medication, and had at least one assessment for the specified timepoint(s) at or after baseline.
Measure: Least Squares Mean (95% Confidence Interval); unit: A1C Percentage
Arm/Group | Ertugliflozin 5 mg (Overall Cardiovascular Study) | Ertugliflozin 15 mg (Overall Cardiovascular Study) | Placebo (Overall Cardiovascular Study)
Number analyzed (Participants) | 2746 | 2747 | 2745
A1C Percentage | -0.48 [-0.52 to -0.43] | -0.46 [-0.50 to -0.41] | -0.08 [-0.14 to -0.03]
Statistical Analysis 1: Comparison: Ertugliflozin 15 mg (Overall Cardiovascular Study) vs Placebo (Overall Cardiovascular Study); Test type: Superiority; p < 0.001, Constrained longitudinal data analysis — Constrained longitudinal data analysis (cLDA) model with fixed effects for treatment, time, baseline eGFR (continuous) and the interaction of time by treatment. Time was treated as a categorical variable; Difference in the least squares means = -0.37, 95% CI 2-sided [-0.45 to -0.30] — Ertugliflozin vs. Placebo
Statistical Analysis 2: Comparison: Ertugliflozin 5 mg (Overall Cardiovascular Study) vs Placebo (Overall Cardiovascular Study); Test type: Superiority; p < 0.001, cLDA — [p-value comment as in outcome 20, analysis 1]; Ertugliflozin vs. Placebo; Difference in Least Squares Means = -0.39, 95% CI 2-sided [-0.46 to -0.32]

21. Secondary Outcome: Change From Baseline in A1C at Month 36 (Overall Cardiovascular Study)
Description: A1C is a blood marker used to report average blood glucose levels over prolonged periods of time and is reported as a percentage (%). A1C represents the percentage of glycated hemoglobin. This change from baseline reflects the Month 36 A1C minus the Week 0 A1C. A negative number indicates a reduction in A1C level. Participants who met glycemic rescue criteria received glycemic rescue medication.
Time Frame: Baseline and Month 36
Population: The analysis population included all participants who were randomized, received at least one dose of blinded study medication, and had a measurement for the analysis endpoint for the specified timepoint(s) at both baseline and Month 36.
Measure: Mean (95% Confidence Interval); unit: A1C Percentage
Arm/Group | Ertugliflozin 5 mg (Overall Cardiovascular Study) | Ertugliflozin 15 mg (Overall Cardiovascular Study) | Placebo (Overall Cardiovascular Study)
Number analyzed (Participants) | 1590 | 1574 | 1501
A1C Percentage | -0.42 [-0.47 to -0.37] | -0.38 [-0.43 to -0.33] | -0.04 [-0.10 to 0.01]

22. Secondary Outcome: Change From Baseline in A1C at Month 48 (Overall Cardiovascular Study)
Description: A1C is a blood marker used to report average blood glucose levels over prolonged periods of time and is reported as a percentage (%). A1C represents the percentage of glycated hemoglobin. This change from baseline reflects the Month 48 A1C minus the Week 0 A1C. A negative number indicates a reduction in A1C level. Participants who met glycemic rescue criteria received glycemic rescue medication.
Time Frame: Baseline and Month 48
Population: The analysis population included all participants who were randomized, received at least one dose of blinded study medication, and had at least one assessment for specified timepoint(s) at or after baseline.
Measure: Least Squares Mean (95% Confidence Interval); unit: A1C Percentage
Arm/Group | Ertugliflozin 5 mg (Overall Cardiovascular Study) | Ertugliflozin 15 mg (Overall Cardiovascular Study) | Placebo (Overall Cardiovascular Study)
Number analyzed (Participants) | 2746 | 2747 | 2745
A1C Percentage | -0.22 [-0.29 to -0.15] | -0.17 [-0.24 to -0.10] | 0.14 [0.07 to 0.22]
Statistical Analysis 1: Comparison: Ertugliflozin 15 mg (Overall Cardiovascular Study) vs Placebo (Overall Cardiovascular Study); Test type: Superiority; p = 0.001, cLDA — [p-value comment as in outcome 20, analysis 1]; Difference in the least squares means = -0.31, 95% CI 2-sided [-0.41 to -0.21]
Statistical Analysis 2: Comparison: Ertugliflozin 5 mg (Overall Cardiovascular Study) vs Placebo (Overall Cardiovascular Study); Test type: Superiority; p < 0.001, cLDA model — [p-value comment as in outcome 20, analysis 1]; Difference in the least squares means = -0.36, 95% CI 2-sided [-0.46 to -0.26]

23. Secondary Outcome: Change From Baseline in A1C at Month 60 (Overall Cardiovascular Study)
Description: A1C is a blood marker used to report average blood glucose levels over prolonged periods of time and is reported as a percentage (%). A1C represents the percentage of glycated hemoglobin. This change from baseline reflects the Month 60 A1C minus the Week 0 A1C. A negative number indicates a reduction in A1C level. Participants who met glycemic rescue criteria received glycemic rescue medication.
Time Frame: Baseline and Month 60
Population: The analysis population included all participants who were randomized, received at least one dose of blinded study medication, and had a measurement for the analysis endpoint for the specified timepoint(s) at both baseline and Month 60.
Measure: Mean (95% Confidence Interval); unit: A1C Percentage
Arm/Group | Ertugliflozin 5 mg (Overall Cardiovascular Study) | Ertugliflozin 15 mg (Overall Cardiovascular Study) | Placebo (Overall Cardiovascular Study)
Number analyzed (Participants) | 526 | 527 | 477
A1C Percentage | -0.25 [-0.35 to -0.15] | -0.28 [-0.38 to -0.18] | -0.10 [-0.20 to 0.00]

24. Secondary Outcome: Change From Baseline in A1C at Month 72 (Overall Cardiovascular Study)
Description: A1C is blood marker used to report average blood glucose levels over prolonged periods of time and is reported as a percentage (%). A1C represents the percentage of glycated hemoglobin. This change from baseline reflects the Month 72 A1C minus the Week 0 A1C. A negative number indicates a reduction in A1C level. Participants who met glycemic rescue criteria received glycemic rescue medication.
Time Frame: Baseline and Month 72
Population: The analysis population included all participants who were randomized, received at least one dose of blinded study medication, and had a measurement for the analysis endpoint for the specified timepoint(s) at both baseline and Month 72.
Measure: Mean (95% Confidence Interval); unit: A1C Percentage
Arm/Group | Ertugliflozin 5 mg (Overall Cardiovascular Study) | Ertugliflozin 15 mg (Overall Cardiovascular Study) | Placebo (Overall Cardiovascular Study)
Number analyzed (Participants) | 13 | 12 | 9
A1C Percentage | -0.35 [-0.89 to 0.20] | -0.13 [-0.99 to 0.74] | 0.24 [-0.74 to 1.23]

25. Secondary Outcome: Percentage of Participants With an A1C <7% (<53 mmol/Mol) at Week 18 (Overall Cardiovascular Study)
Description: A1C is a blood marker used to report average blood glucose levels over prolonged periods of time and is reported as a percentage (%). A1C represents the percentage of glycated hemoglobin. Participants who met glycemic rescue criteria received glycemic rescue medication.
Time Frame: Week 18
Population: The analysis population included all randomized and treated participants with an A1C measurement for the analysis endpoint for the specified timepoint(s) at Week 18.
Measure: Number; unit: Percentage of Participants
Arm/Group | Ertugliflozin 5 mg (Overall Cardiovascular Study) | Ertugliflozin 15 mg (Overall Cardiovascular Study) | Placebo (Overall Cardiovascular Study)
Number analyzed (Participants) | 2544 | 2520 | 2527
Percentage of Participants | 28.4 | 28.2 | 15.5

26. Secondary Outcome: Percentage of Participants With an A1C <7% (<53 mmol/Mol) at Week 52 (Overall Cardiovascular Study)
Description: as for outcome 25
Time Frame: Week 52
Population: The analysis population included all randomized and treated participants with an A1C measurement for the analysis endpoint for the specified timepoint(s) at Week 52.
Measure: Number; unit: Percentage of Participants
Arm/Group | Ertugliflozin 5 mg (Overall Cardiovascular Study) | Ertugliflozin 15 mg (Overall Cardiovascular Study) | Placebo (Overall Cardiovascular Study)
Number analyzed (Participants) | 2363 | 2347 | 2311
Percentage of Participants | 28.3 | 29.0 | 17.4

27. Secondary Outcome: Percentage of Participants With an A1C <7% (<53 mmol/Mol) at Month 24 (Overall Cardiovascular Study)
Description: as for outcome 25
Time Frame: Month 24
Population: The analysis population included all randomized and treated participants with an A1C measurement for the analysis endpoint for the specified timepoint(s) at Month 24.
Measure: Number; unit: Percentage of Participants
Arm/Group | Ertugliflozin 5 mg (Overall Cardiovascular Study) | Ertugliflozin 15 mg (Overall Cardiovascular Study) | Placebo (Overall Cardiovascular Study)
Number analyzed (Participants) | 1570 | 1541 | 1496
Percentage of Participants | 23.9 | 23.8 | 16.6

28. Secondary Outcome: Percentage of Participants With an A1C <7% (<53 mmol/Mol) at Month 36 (Overall Cardiovascular Study)
Description: as for outcome 25
Time Frame: Month 36
Population: The analysis population included all randomized and treated participants with an A1C measurement for the analysis endpoint for the specified timepoint(s) at Month 36.
Measure: Number; unit: Percentage of Participants
Arm/Group | Ertugliflozin 5 mg (Overall Cardiovascular Study) | Ertugliflozin 15 mg (Overall Cardiovascular Study) | Placebo (Overall Cardiovascular Study)
Number analyzed (Participants) | 1592 | 1578 | 1507
Percentage of Participants | 23.1 | 22.7 | 16.9

29. Secondary Outcome: Percentage of Participants With an A1C <7% (<53 mmol/Mol) at Month 48 (Overall Cardiovascular Study)
Description: as for outcome 25
Time Frame: Month 48
Population: The analysis population included all randomized and treated participants with an A1C measurement for the analysis endpoint for the specified timepoint(s) at Month 48.
Measure: Number; unit: Percentage of Participants
Arm/Group | Ertugliflozin 5 mg (Overall Cardiovascular Study) | Ertugliflozin 15 mg (Overall Cardiovascular Study) | Placebo (Overall Cardiovascular Study)
Number analyzed (Participants) | 876 | 860 | 786
Percentage of Participants | 24.9 | 22.7 | 18.2

30. Secondary Outcome: Percentage of Participants With an A1C <7% (<53 mmol/Mol) at Month 60 (Overall Cardiovascular Study)
Description: as for outcome 25
Time Frame: Month 60
Population: The analysis population included all randomized and treated participants with an A1C measurement for the analysis endpoint for the specified timepoint(s) at Month 60.
Measure: Number; unit: Percentage of Participants
Arm/Group | Ertugliflozin 5 mg (Overall Cardiovascular Study) | Ertugliflozin 15 mg (Overall Cardiovascular Study) | Placebo (Overall Cardiovascular Study)
Number analyzed (Participants) | 526 | 529 | 478
Percentage of Participants | 18.6 | 20.0 | 16.5

31. Secondary Outcome: Percentage of Participants With an A1C <6.5% (<48 mmol/Mol) at Week 18 (Overall Cardiovascular Study)
Description: as for outcome 25
Time Frame: Week 18
Population: as for outcome 25
Measure: Number; unit: Percentage of Participants
Arm/Group | Ertugliflozin 5 mg (Overall Cardiovascular Study) | Ertugliflozin 15 mg (Overall Cardiovascular Study) | Placebo (Overall Cardiovascular Study)
Number analyzed (Participants) | 2544 | 2520 | 2727
Percentage of Participants | 9.0 | 8.8 | 4.7

32. Secondary Outcome: Percentage of Participants With an A1C <6.5% (<48 mmol/Mol) at Week 52 (Overall Cardiovascular Study)
Description: as for outcome 25
Time Frame: Week 52
Population: as for outcome 26
Measure: Number; unit: Percentage of Participants
Arm/Group | Ertugliflozin 5 mg (Overall Cardiovascular Study) | Ertugliflozin 15 mg (Overall Cardiovascular Study) | Placebo (Overall Cardiovascular Study)
Number analyzed (Participants) | 2363 | 2347 | 2311
Percentage of Participants | 9.4 | 10.9 | 6.1

33. Secondary Outcome: Percentage of Participants With an A1C <6.5% (<48 mmol/Mol) at Month 24 (Overall Cardiovascular Study)
Description: as for outcome 25
Time Frame: Month 24
Population: as for outcome 27
Measure: Number; unit: Percentage of Participants
Arm/Group | Ertugliflozin 5 mg (Overall Cardiovascular Study) | Ertugliflozin 15 mg (Overall Cardiovascular Study) | Placebo (Overall Cardiovascular Study)
Number analyzed (Participants) | 1570 | 1541 | 1496
Percentage of Participants | 9.2 | 8.6 | 5.8

34. Secondary Outcome: Percentage of Participants With an A1C <6.5% (<48 mmol/Mol) at Month 36 (Overall Cardiovascular Study)
Description: as for outcome 25
Time Frame: Month 36
Population: as for outcome 28
Measure: Number; unit: Percentage of Participants
Arm/Group | Ertugliflozin 5 mg (Overall Cardiovascular Study) | Ertugliflozin 15 mg (Overall Cardiovascular Study) | Placebo (Overall Cardiovascular Study)
Number analyzed (Participants) | 1592 | 1578 | 1507
Percentage of Participants | 7.9 | 8.0 | 5.8

35. Secondary Outcome: Percentage of Participants With an A1C <6.5% (<48 mmol/Mol) at Month 48 (Overall Cardiovascular Study)
Description: as for outcome 25
Time Frame: Month 48
Population: as for outcome 29
Measure: Number; unit: Percentage of Participants
Arm/Group | Ertugliflozin 5 mg (Overall Cardiovascular Study) | Ertugliflozin 15 mg (Overall Cardiovascular Study) | Placebo (Overall Cardiovascular Study)
Number analyzed (Participants) | 876 | 860 | 786
Percentage of Participants | 8.1 | 9.1 | 7.5

36. Secondary Outcome: Percentage of Participants With an A1C <6.5% (<48 mmol/Mol) at Month 60 (Overall Cardiovascular Study)
Description: as for outcome 25
Time Frame: Month 60
Population: as for outcome 30
Measure: Number; unit: Percentage of Participants
Arm/Group | Ertugliflozin 5 mg (Overall Cardiovascular Study) | Ertugliflozin 15 mg (Overall Cardiovascular Study) | Placebo (Overall Cardiovascular Study)
Number analyzed (Participants) | 526 | 529 | 478
Percentage of Participants | 5.3 | 9.5 | 6.5

37. Secondary Outcome: Change From Baseline in Fasting Plasma Glucose (FPG) at Week 18 (Excluding Rescue Approach) (Overall Cardiovascular Study)
Description: FPG was analyzed after an overnight fast. This change from baseline reflects the Week 18 FPG minus the Week 0 FPG. A negative number indicates a reduction in FPG. Participants who met glycemic rescue criteria received glycemic rescue medication. "Excluding rescue", excluded all data following the initiation of rescue in order to avoid the confounding influence of the rescue therapy.
Time Frame: Baseline and Week 18
Population: The analysis population included all participants who were randomized, received at least one dose of blinded study medication, and had at least one measurement for the analysis endpoint for the specified timepoint(s) at or after Baseline.
Measure: Least Squares Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Ertugliflozin 5 mg (Overall Cardiovascular Study) | Ertugliflozin 15 mg (Overall Cardiovascular Study) | Placebo (Overall Cardiovascular Study)
Number analyzed (Participants) | 2745 | 2747 | 2744
mg/dL | -32.18 [-33.76 to -30.61] | -34.64 [-36.21 to -33.08] | -17.08 [-18.69 to -15.48]
Statistical Analysis 1: Comparison: Ertugliflozin 15 mg (Overall Cardiovascular Study) vs Placebo (Overall Cardiovascular Study); Test type: Superiority; p < 0.001, CLDA; cLDA model with fixed effects for treatment, time, baseline eGFR (continuous), and the interaction of time by treatment; Difference in the Least Squares Means = -17.56, 95% CI 2-sided [-19.49 to -15.63]
Statistical Analysis 2: Comparison: Ertugliflozin 5 mg (Overall Cardiovascular Study) vs Placebo (Overall Cardiovascular Study); Test type: Superiority; p < 0.001, cLDA; cLDA model with fixed effects for treatment, time, baseline eGFR (continuous), and the interaction of time by treatment; Difference in the Least Squares Means = -15.10, 95% CI 2-sided [-17.03 to -13.17]

38. Secondary Outcome: Change From Baseline in Fasting Plasma Glucose (FPG) at Week 52 (Overall Cardiovascular Study)
Description: FPG was analyzed after an overnight fast. This change from baseline reflects the Week 52 FPG minus the Week 0 FPG. A negative number indicates a reduction in FPG. Participants who met glycemic rescue criteria received glycemic rescue medication.
Time Frame: Baseline and Week 52
Population: The analysis population included all participants who were randomized, received at least one dose of blinded study medication, and had a measurement for the analysis endpoint for the specified timepoint(s) at both Baseline and Week 52.
Measure: Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Ertugliflozin 5 mg (Overall Cardiovascular Study) | Ertugliflozin 15 mg (Overall Cardiovascular Study) | Placebo (Overall Cardiovascular Study)
Number analyzed (Participants) | 2352 | 2328 | 2295
mg/dL | -28.63 [-30.52 to -26.74] | -28.97 [-30.78 to -27.15] | -8.76 [-10.75 to -6.77]

39. Secondary Outcome: Change From Baseline in Fasting Plasma Glucose (FPG) at Month 24 (Overall Cardiovascular Study)
Description: FPG was analyzed after an overnight fast. This change from baseline reflects the Month 24 FPG minus the Week 0 FPG. A negative number indicates a reduction in FPG. Participants who met glycemic rescue criteria received glycemic rescue medication.
Time Frame: Baseline and Month 24
Population: The analysis population included all participants who were randomized, received at least one dose of blinded study medication, and had a measurement for the analysis endpoint for the specified timepoint(s) at both Baseline and Month 24.
Measure: Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Ertugliflozin 5 mg (Overall Cardiovascular Study) | Ertugliflozin 15 mg (Overall Cardiovascular Study) | Placebo (Overall Cardiovascular Study)
Number analyzed (Participants) | 1562 | 1536 | 1487
mg/dL | -22.09 [-24.39 to -19.80] | -24.31 [-26.76 to -21.86] | -4.39 [-6.99 to -1.78]

40. Secondary Outcome: Change From Baseline in Fasting Plasma Glucose (FPG) at Month 36 (Overall Cardiovascular Study)
Description: FPG was analyzed after an overnight fast. This change from baseline reflects the Month 36 FPG minus the Week 0 FPG. A negative number indicates a reduction in FPG. Participants who met glycemic rescue criteria received glycemic rescue medication.
Time Frame: Baseline and Month 36
Population: as for outcome 21
Measure: Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Ertugliflozin 5 mg (Overall Cardiovascular Study) | Ertugliflozin 15 mg (Overall Cardiovascular Study) | Placebo (Overall Cardiovascular Study)
Number analyzed (Participants) | 1579 | 1567 | 1491
mg/dL | -19.39 [-21.88 to -16.89] | -22.59 [-24.96 to -20.21] | -3.63 [-6.45 to -0.81]

41. Secondary Outcome: Change From Baseline in Fasting Plasma Glucose (FPG) at Month 48 (Overall Cardiovascular Study)
Description: FPG was analyzed after an overnight fast. This change from baseline reflects the Month 48 FPG minus the Week 0 FPG. A negative number indicates a reduction in FPG. Participants who met glycemic rescue criteria received glycemic rescue medication.
Time Frame: Baseline and Month 48
Population: The analysis population included all participants who were randomized, received at least one dose of blinded study medication, and had a measurement for the analysis endpoint for the specified timepoint(s) at both Baseline and Month 48.
Measure: Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Ertugliflozin 5 mg (Overall Cardiovascular Study) | Ertugliflozin 15 mg (Overall Cardiovascular Study) | Placebo (Overall Cardiovascular Study)
Number analyzed (Participants) | 868 | 861 | 777
mg/dL | -15.28 [-18.66 to -11.90] | -16.16 [-19.50 to -12.83] | 3.59 [-0.22 to 7.40]

42. Secondary Outcome: Change From Baseline in Fasting Plasma Glucose (FPG) at Month 60 (Overall Cardiovascular Study)
Description: FPG was analyzed after an overnight fast. This change from baseline reflects the Month 60 FPG minus the Week 0 FPG. A negative number indicates a reduction in FPG. Participants who met glycemic rescue criteria received glycemic rescue medication.
Time Frame: Baseline and Month 60
Population: as for outcome 23
Measure: Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Ertugliflozin 5 mg (Overall Cardiovascular Study) | Ertugliflozin 15 mg (Overall Cardiovascular Study) | Placebo (Overall Cardiovascular Study)
Number analyzed (Participants) | 520 | 524 | 473
mg/dL | -13.87 [-18.34 to -9.40] | -11.15 [-15.78 to -6.52] | -4.69 [-9.72 to 0.34]

43. Secondary Outcome: Change From Baseline in Fasting Plasma Glucose (FPG) at Month 72 (Overall Cardiovascular Study)
Description: FPG was analyzed after an overnight fast. This change from baseline reflects the Month 72 FPG minus the Week 0 FPG. A negative number indicates a reduction in FPG. Participants who met glycemic rescue criteria received glycemic rescue medication.
Time Frame: Baseline and Month 72
Population: as for outcome 24
Measure: Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Ertugliflozin 5 mg (Overall Cardiovascular Study) | Ertugliflozin 15 mg (Overall Cardiovascular Study) | Placebo (Overall Cardiovascular Study)
Number analyzed (Participants) | 13 | 12 | 9
mg/dL | -2.46 [-31.28 to 26.36] | -84.83 [-127.31 to -42.35] | 14.56 [-23.11 to 52.22]

44. Secondary Outcome: Time to the First Occurrence of a Participant Receiving Glycemic Rescue Therapy Through Week 18 (Overall Cardiovascular Study)
Description: Participants who met glycemic rescue criteria received open-label sitagliptin glycemic rescue medication.
Time Frame: Up to 18 weeks
Population: The analysis population included all participants who were randomized, received at least one dose of blinded study medication, and received glycemic rescue by Week 18.
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | Ertugliflozin 5 mg (Overall Cardiovascular Study) | Ertugliflozin 15 mg (Overall Cardiovascular Study) | Placebo (Overall Cardiovascular Study)
Number analyzed (Participants) | 141 | 102 | 275
Days | 59.0 [36 to 99] | 51.0 [18 to 91] | 74.0 [37 to 97]
Statistical Analysis 1: Comparison: Ertugliflozin 15 mg (Overall Cardiovascular Study) vs Placebo (Overall Cardiovascular Study); Test type: Superiority; p < 0.001, Log Rank; Log-Rank Test for the comparison to Placebo was based on all data (including for those participants who never had the event)
Statistical Analysis 2: Comparison: Ertugliflozin 5 mg (Overall Cardiovascular Study) vs Placebo (Overall Cardiovascular Study); Test type: Superiority; p < 0.001, Log Rank; [statistical method as in outcome 44, analysis 1]

45. Secondary Outcome: Time to Initiation of Insulin for Participants Not on Insulin at Baseline (Overall Cardiovascular Study)
Description: Participants who were not on insulin therapy at the start of study medication.
Time Frame: Up to approximately 6 years
Population: The analysis population included all participants who were randomized, received at least one dose of blinded study medication, and were not on insulin therapy at the start of study medication.
Measure: Median (Full Range); unit: Days
Arm/Group | Ertugliflozin 5 mg (Overall Cardiovascular Study) | Ertugliflozin 15 mg (Overall Cardiovascular Study) | Placebo (Overall Cardiovascular Study)
Number analyzed (Participants) | 1442 | 1499 | 1400
Days | 602 [8 to 1850] | 650 [16 to 1934] | 482 [10 to 1838]
Statistical Analysis 1: Comparison: Ertugliflozin 15 mg (Overall Cardiovascular Study) vs Placebo (Overall Cardiovascular Study); Test type: Superiority; p < 0.001, Log Rank; [statistical method as in outcome 44, analysis 1]
Statistical Analysis 2: Comparison: Ertugliflozin 5 mg (Overall Cardiovascular Study) vs Placebo (Overall Cardiovascular Study); Test type: Superiority; p < 0.001, Log Rank; [statistical method as in outcome 44, analysis 1]

46. Secondary Outcome: Baseline Insulin Dose for Participants Who Were on Insulin at Baseline (Overall Cardiovascular Study)
Description: Baseline reflects Week 0 insulin dose.
Time Frame: Baseline
Population: The analysis population included all participants who were randomized and were treated with insulin at Baseline.
Measure: Mean (Standard Deviation); unit: Units/Day
Arm/Group | Ertugliflozin 5 mg (Overall Cardiovascular Study) | Ertugliflozin 15 mg (Overall Cardiovascular Study) | Placebo (Overall Cardiovascular Study)
Number analyzed (Participants) | 1304 | 1248 | 1345
Units/Day | 63.82 (48.11) | 62.15 (44.46) | 65.74 (46.34)

47. Secondary Outcome: Change From Baseline in Insulin Dose at Week 18 for Participants Who Were on Insulin at Baseline (Overall Cardiovascular Study)
Description: This change from baseline reflects the Week 18 insulin dose minus the Week 0 insulin dose. A negative number indicates a reduction in the insulin dose.
Time Frame: Baseline and Week 18
Population: The analysis population included all participants who were randomized, received at least one dose of blinded study medication, were treated with insulin at Baseline, and had a measurement for the analysis endpoint for the specified timepoint(s) at both Baseline and Week 18.
Measure: Mean (95% Confidence Interval); unit: Units/Day
Arm/Group | Ertugliflozin 5 mg (Overall Cardiovascular Study) | Ertugliflozin 15 mg (Overall Cardiovascular Study) | Placebo (Overall Cardiovascular Study)
Number analyzed (Participants) | 1297 | 1237 | 1304
Units/Day | 1.05 [0.29 to 1.82] | 0.81 [-0.10 to 1.71] | 3.71 [2.72 to 4.70]

48. Secondary Outcome: Change From Baseline in Insulin Dose at Week 52 for Participants Who Were on Insulin at Baseline (Overall Cardiovascular Study)
Description: This change from baseline reflects the Week 52 insulin dose minus the Week 0 insulin dose. A negative number indicates a reduction in the insulin dose.
Time Frame: Baseline and Week 52
Population: The analysis population included all participants who were randomized, received at least one dose of blinded study medication, were treated with insulin at Baseline, and had a measurement for the analysis endpoint for the specified timepoint(s) at both Baseline and Week 52.
Measure: Mean (95% Confidence Interval); unit: Units/Day
Arm/Group | Ertugliflozin 5 mg (Overall Cardiovascular Study) | Ertugliflozin 15 mg (Overall Cardiovascular Study) | Placebo (Overall Cardiovascular Study)
Number analyzed (Participants) | 1103 | 1067 | 1130
Units/Day | 0.84 [-0.15 to 1.82] | -1.69 [-2.83 to -0.54] | 5.57 [4.16 to 6.98]

49. Secondary Outcome: Change From Baseline in Insulin Dose at Month 24 for Participants Who Were on Insulin at Baseline (Overall Cardiovascular Study)
Description: This change from baseline reflects the Month 24 insulin dose minus the Week 0 insulin dose. A negative number indicates a reduction in the insulin dose.
Time Frame: Baseline and Month 24
Population: The analysis population included all participants who were randomized, received at least one dose of blinded study medication, were treated with insulin at Baseline, and had a measurement for the analysis endpoint for the specified timepoint(s) at both Baseline and Month 24.
Measure: Mean (95% Confidence Interval); unit: Units/Day
Arm/Group | Ertugliflozin 5 mg (Overall Cardiovascular Study) | Ertugliflozin 15 mg (Overall Cardiovascular Study) | Placebo (Overall Cardiovascular Study)
Number analyzed (Participants) | 1004 | 966 | 998
Units/Day | 0.45 [-0.72 to 1.63] | -1.58 [-2.95 to -0.21] | 6.16 [4.47 to 7.85]

50. Secondary Outcome: Change From Baseline in Insulin Dose at Month 36 for Participants Who Were on Insulin at Baseline (Overall Cardiovascular Study)
Description: This change from baseline reflects the Month 36 insulin dose minus the Week 0 insulin dose. A negative number indicates a reduction in the insulin dose.
Time Frame: Baseline and Month 36
Population: The analysis population included all participants who were randomized, received at least one dose of blinded study medication, were treated with insulin at Baseline, and had a measurement for the analysis endpoint for the specified timepoint(s) at both Baseline and Month 36.
Measure: Mean (95% Confidence Interval); unit: Units/Day
Arm/Group | Ertugliflozin 5 mg (Overall Cardiovascular Study) | Ertugliflozin 15 mg (Overall Cardiovascular Study) | Placebo (Overall Cardiovascular Study)
Number analyzed (Participants) | 465 | 464 | 419
Units/Day | 1.64 [-0.77 to 4.05] | -1.92 [-4.31 to 0.46] | 7.99 [4.65 to 11.34]

51. Secondary Outcome: Change From Baseline in Insulin Dose at Month 48 for Participants Who Were on Insulin at Baseline (Overall Cardiovascular Study)
Description: This change from baseline reflects the Month 48 insulin dose minus the Week 0 insulin dose. A negative number indicates a reduction in the insulin dose.
Time Frame: Baseline and Month 48
Population: The analysis population included all participants who were randomized, received at least one dose of blinded study medication, were treated with insulin at Baseline, and had a measurement for the analysis endpoint for the specified timepoint(s) at both Baseline and Month 48.
Measure: Mean (95% Confidence Interval); unit: Units/Day
Arm/Group | Ertugliflozin 5 mg (Overall Cardiovascular Study) | Ertugliflozin 15 mg (Overall Cardiovascular Study) | Placebo (Overall Cardiovascular Study)
Number analyzed (Participants) | 387 | 384 | 326
Units/Day | 2.96 [0.41 to 5.51] | -1.87 [-4.80 to 1.05] | 7.28 [3.66 to 10.91]

52. Secondary Outcome: Change From Baseline in Insulin Dose at Month 60 for Participants Who Were on Insulin at Baseline (Overall Cardiovascular Study)
Description: This change from baseline reflects the Month 60 insulin dose minus the Week 0 insulin dose. A negative number indicates a reduction in the insulin dose.
Time Frame: Baseline and Month 60
Population: The analysis population included all participants who were randomized, received at least one dose of blinded study medication, were treated with insulin at Baseline, and had a measurement for the analysis endpoint for the specified timepoint(s) at both Baseline and Month 60.
Measure: Mean (95% Confidence Interval); unit: Units/Day
Arm/Group | Ertugliflozin 5 mg (Overall Cardiovascular Study) | Ertugliflozin 15 mg (Overall Cardiovascular Study) | Placebo (Overall Cardiovascular Study)
Number analyzed (Participants) | 45 | 47 | 38
Units/Day | -2.47 [-9.65 to 4.72] | -1.77 [-11.95 to 8.42] | 9.42 [1.46 to 17.39]

53. Secondary Outcome: Change From Baseline in Sitting Systolic Blood Pressure (SBP) at Week 18 (Excluding Rescue Approach) (Overall Cardiovascular Study)
Description: This change from baseline reflects the Week 18 SBP minus the Week 0 SBP. A negative number indicates a reduction in SBP. Participants who met glycemic rescue criteria received glycemic rescue medication. "Excluding rescue", excluded all data following the initiation of rescue in order to avoid the confounding influence of the rescue therapy.
Time Frame: Baseline and Week 18
Population: as for outcome 37
Measure: Least Squares Mean (95% Confidence Interval); unit: mmHg
Arm/Group | Ertugliflozin 5 mg (Overall Cardiovascular Study) | Ertugliflozin 15 mg (Overall Cardiovascular Study) | Placebo (Overall Cardiovascular Study)
Number analyzed (Participants) | 2746 | 2746 | 2745
mmHg | -2.51 [-3.00 to -2.02] | -2.75 [-3.24 to -2.26] | 0.03 [-0.48 to 0.53]
Statistical Analysis 1: Comparison: Ertugliflozin 15 mg (Overall Cardiovascular Study) vs Placebo (Overall Cardiovascular Study); Test type: Superiority; p < 0.001, cLDA; The model had fixed effects for treatment, time, baseline eGFR (continuous) and the interaction of time by treatment; Difference in the Least Squares Means = -2.78, 95% CI 2-sided [-3.45 to -2.10]
Statistical Analysis 2: Comparison: Ertugliflozin 5 mg (Overall Cardiovascular Study) vs Placebo (Overall Cardiovascular Study); Test type: Superiority; p < 0.001, cLDA; The model had fixed effects for treatment, time, baseline eGFR (continuous) and the interaction of time by treatment; Difference in the Least Squares Means = -2.53, 95% CI 2-sided [-3.21 to -1.86]

54. Secondary Outcome: Change From Baseline in Sitting Systolic Blood Pressure (SBP) at Week 52 (Overall Cardiovascular Study)
Description: This change from baseline reflects the Week 52 sitting SBP minus the Week 0 SBP. A negative number indicates a reduction in SBP. Participants who met glycemic rescue criteria received glycemic rescue medication.
Time Frame: Baseline and Week 52
Population: as for outcome 37
Measure: Least Squares Mean (95% Confidence Interval); unit: mmHg
Arm/Group | Ertugliflozin 5 mg (Overall Cardiovascular Study) | Ertugliflozin 15 mg (Overall Cardiovascular Study) | Placebo (Overall Cardiovascular Study)
Number analyzed (Participants) | 2746 | 2747 | 2745
mmHg | -1.84 [-2.35 to -1.32] | -2.41 [-2.92 to -1.89] | 0.75 [0.23 to 1.26]
Statistical Analysis 1: Comparison: Ertugliflozin 15 mg (Overall Cardiovascular Study) vs Placebo (Overall Cardiovascular Study); Test type: Superiority; p < 0.001, cLDA; The model had fixed effects for treatment, time, baseline eGFR (continuous) and the interaction of time by treatment; Difference in the Least Squares Mean = -3.15, 95% CI 2-sided [-3.85 to -2.45]
Statistical Analysis 2: Comparison: Ertugliflozin 5 mg (Overall Cardiovascular Study) vs Placebo (Overall Cardiovascular Study); Test type: Superiority; p < 0.001, cLDA; The model had fixed effects for treatment, time, baseline eGFR (continuous) and the interaction of time by treatment; Difference in the Least Squares Means = -2.58, 95% CI 2-sided [-3.28 to -1.89]

55. Secondary Outcome: Change From Baseline in Sitting Systolic Blood Pressure (SBP) at Month 24 (Overall Cardiovascular Study)
Description: This change from baseline reflects the Month 24 SBP minus the Week 0 SBP. A negative number indicates a reduction in SBP. Participants who met glycemic rescue criteria received glycemic rescue medication.
Time Frame: Baseline and Month 24
Population: as for outcome 37
Measure: Least Squares Mean (95% Confidence Interval); unit: mmHg
Arm/Group | Ertugliflozin 5 mg (Overall Cardiovascular Study) | Ertugliflozin 15 mg (Overall Cardiovascular Study) | Placebo (Overall Cardiovascular Study)
Number analyzed (Participants) | 2746 | 2747 | 2745
mmHg | -1.80 [-2.42 to -1.19] | -1.82 [-2.44 to -1.19] | 0.90 [0.27 to 1.53]
Statistical Analysis 1: Comparison: Ertugliflozin 15 mg (Overall Cardiovascular Study) vs Placebo (Overall Cardiovascular Study); Test type: Superiority; p < 0.001, cLDA; The model had fixed effects for treatment, time, baseline eGFR (continuous) and the interaction of time by treatment; Difference in the Least Squares Means = -2.72, 95% CI 2-sided [-3.57 to -1.86]
Statistical Analysis 2: Comparison: Ertugliflozin 5 mg (Overall Cardiovascular Study) vs Placebo (Overall Cardiovascular Study); Test type: Superiority; p < 0.001, cLDA; The model had fixed effects for treatment, time, baseline eGFR (continuous) and the interaction of time by treatment; Difference in the Least Squares Means = -2.70, 95% CI 2-sided [-3.56 to -1.85]

56. Secondary Outcome: Change From Baseline in Sitting Systolic Blood Pressure (SBP) at Month 36 (Overall Cardiovascular Study)
Description: This change from baseline reflects the Month 36 SBP minus the Week 0 SBP. A negative number indicates a reduction in SBP. Participants who met glycemic rescue criteria received glycemic rescue medication.
Time Frame: Baseline and Month 36
Population: as for outcome 21
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Ertugliflozin 5 mg (Overall Cardiovascular Study) | Ertugliflozin 15 mg (Overall Cardiovascular Study) | Placebo (Overall Cardiovascular Study)
Number analyzed (Participants) | 1593 | 1580 | 1505
mmHg | -1.55 (14.56) | -1.21 (15.05) | 0.84 (14.63)

57. Secondary Outcome: Change From Baseline in Sitting Systolic Blood Pressure (SBP) at Month 48 (Overall Cardiovascular Study)
Description: This change from baseline reflects the Month 48 SBP minus the Week 0 SBP. A negative number indicates a reduction in SBP. Participants who met glycemic rescue criteria received glycemic rescue medication.
Time Frame: Baseline and Month 48
Population: as for outcome 37
Measure: Least Squares Mean (95% Confidence Interval); unit: mmHg
Arm/Group | Ertugliflozin 5 mg (Overall Cardiovascular Study) | Ertugliflozin 15 mg (Overall Cardiovascular Study) | Placebo (Overall Cardiovascular Study)
Number analyzed (Participants) | 2746 | 2747 | 2745
mmHg | -2.07 [-2.84 to -1.31] | -2.26 [-3.03 to -1.49] | 0.53 [-0.27 to 1.33]
Statistical Analysis 1: Comparison: Ertugliflozin 5 mg (Overall Cardiovascular Study) vs Placebo (Overall Cardiovascular Study); Test type: Superiority; p < 0.001, cLDA; The model had fixed effects for treatment, time, baseline eGFR (continuous) and the interaction of time by treatment; Difference in the Least Squares Means = -2.60, 95% CI 2-sided [-3.68 to -1.52]
Statistical Analysis 2: Comparison: Ertugliflozin 15 mg (Overall Cardiovascular Study) vs Placebo (Overall Cardiovascular Study); Test type: Superiority; p < 0.001, cLDA; The model had fixed effects for treatment, time, baseline eGFR (continuous) and the interaction of time by treatment; Difference in the Least Squares Means = -2.79, 95% CI 2-sided [-3.87 to -1.71]

58. Secondary Outcome: Change From Baseline in Sitting Systolic Blood Pressure (SBP) at Month 60 (Overall Cardiovascular Study)
Description: This change from baseline reflects the Month 60 SBP minus the Week 0 SBP. A negative number indicates a reduction in SBP. Participants who met glycemic rescue criteria received glycemic rescue medication.
Time Frame: Baseline and Month 60
Population: as for outcome 23
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Ertugliflozin 5 mg (Overall Cardiovascular Study) | Ertugliflozin 15 mg (Overall Cardiovascular Study) | Placebo (Overall Cardiovascular Study)
Number analyzed (Participants) | 525 | 529 | 479
mmHg | -2.18 (15.39) | -1.87 (15.01) | 0.62 (15.85)

59. Secondary Outcome: Change From Baseline in Sitting Systolic Blood Pressure (SBP) at Month 72 (Overall Cardiovascular Study)
Description: This change from baseline reflects the Month 72 SBP minus the Week 0 SBP. A negative number indicates a reduction in SBP. Participants who met glycemic rescue criteria received glycemic rescue medication.
Time Frame: Baseline and Month 72
Population: as for outcome 24
Measure: Mean (95% Confidence Interval); unit: mmHg
Arm/Group | Ertugliflozin 5 mg (Overall Cardiovascular Study) | Ertugliflozin 15 mg (Overall Cardiovascular Study) | Placebo (Overall Cardiovascular Study)
Number analyzed (Participants) | 13 | 12 | 9
mmHg | 1.28 [-7.63 to 10.20] | -3.46 [-10.91 to 3.99] | 2.72 [-5.95 to 11.40]

60. Secondary Outcome: Change From Baseline in Sitting Diastolic Blood Pressure (DBP) at Week 18 (Excluding Rescue Approach) (Overall Cardiovascular Study)
Description: This change from baseline reflects the Week 18 DBP minus the Week 0 DBP. A negative number indicates a reduction in DBP. Participants who met glycemic rescue criteria received glycemic rescue medication. "Excluding rescue", excluded all data following the initiation of rescue in order to avoid the confounding influence of the rescue therapy.
Time Frame: Baseline and Week 18
Population: The analysis population included all participants who were randomized, received at least one dose of blinded study medication, and had at least one measurement for the analysis endpoint at or after Baseline.
Measure: Least Squares Mean (95% Confidence Interval); unit: mmHg
Arm/Group | Ertugliflozin 5 mg (Overall Cardiovascular Study) | Ertugliflozin 15 mg (Overall Cardiovascular Study) | Placebo (Overall Cardiovascular Study)
Number analyzed (Participants) | 2746 | 2746 | 2745
mmHg | -0.99 [-1.29 to -0.70] | -1.08 [-1.38 to -0.79] | -0.12 [-0.42 to 0.18]
Statistical Analysis 1: Comparison: Ertugliflozin 15 mg (Overall Cardiovascular Study) vs Placebo (Overall Cardiovascular Study); Test type: Superiority; p < 0.001, cLDA; cLDA model with fixed effects for treatment, time, baseline eGFR (continuous) and the interaction of time by treatment; Difference in the Least Squares Means = -0.96, 95% CI 2-sided [-1.37 to -0.56]
Statistical Analysis 2: Comparison: Ertugliflozin 5 mg (Overall Cardiovascular Study) vs Placebo (Overall Cardiovascular Study); Test type: Superiority; p < 0.001, cLDA; cLDA model with fixed effects for treatment, time, baseline eGFR (continuous) and the interaction of time by treatment; Difference in the Least Means Squares = -0.87, 95% CI 2-sided [-1.28 to -0.47]

61. Secondary Outcome: Change From Baseline in Sitting Diastolic Blood Pressure (DBP) at Week 52 (Overall Cardiovascular Study)
Description: This change from baseline reflects the Week 52 DBP minus the Week 0 DBP. A negative number indicates a reduction in DBP. Participants who met glycemic rescue criteria received glycemic rescue medication.
Time Frame: Baseline and Week 52
Population: as for outcome 37
Measure: Least Squares Mean (95% Confidence Interval); unit: mmHg
Arm/Group | Ertugliflozin 5 mg (Overall Cardiovascular Study) | Ertugliflozin 15 mg (Overall Cardiovascular Study) | Placebo (Overall Cardiovascular Study)
Number analyzed (Participants) | 2746 | 2747 | 2745
mmHg | -0.97 [-1.28 to -0.67] | -0.95 [-1.26 to -0.65] | -0.15 [-0.45 to 0.16]
Statistical Analysis 1: Comparison: Ertugliflozin 15 mg (Overall Cardiovascular Study) vs Placebo (Overall Cardiovascular Study); Test type: Superiority; p < 0.001, cLDA; The model had fixed effects for treatment, time, baseline eGFR (continuous) and the interaction of time by treatment; Difference in the Least Squares Means = -0.81, 95% CI 2-sided [-1.22 to -0.39]
Statistical Analysis 2: Comparison: Ertugliflozin 5 mg (Overall Cardiovascular Study) vs Placebo (Overall Cardiovascular Study); Test type: Superiority; p < 0.001, cLDA; The model had fixed effects for treatment, time, baseline eGFR (continuous) and the interaction of time by treatment; Difference in the Least Squares Means = -0.83, 95% CI 2-sided [-1.24 to -0.41]

62. Secondary Outcome: Change From Baseline in Sitting Diastolic Blood Pressure (DBP) at Month 24 (Overall Cardiovascular Study)
Description: This change from baseline reflects the Month 24 DBP minus the Week 0 DBP. A negative number indicates a reduction in DBP. Participants who met glycemic rescue criteria received glycemic rescue medication.
Time Frame: Baseline and Month 24
Population: as for outcome 37
Measure: Least Squares Mean (95% Confidence Interval); unit: mmHg
Arm/Group | Ertugliflozin 5 mg (Overall Cardiovascular Study) | Ertugliflozin 15 mg (Overall Cardiovascular Study) | Placebo (Overall Cardiovascular Study)
Number analyzed (Participants) | 2746 | 2747 | 2745
mmHg | -0.94 [-1.31 to -0.57] | -0.90 [-1.27 to -0.53] | -0.23 [-0.60 to 0.15]
Statistical Analysis 1: Comparison: Ertugliflozin 15 mg (Overall Cardiovascular Study) vs Placebo (Overall Cardiovascular Study); Test type: Superiority; p = 0.010, cLDA; The model had fixed effects for treatment, time, baseline eGFR (continuous) and the interaction of time by treatment; Difference in the Least Squares Means = -0.67, 95% CI 2-sided [-1.19 to -0.16]
Statistical Analysis 2: Comparison: Ertugliflozin 5 mg (Overall Cardiovascular Study) vs Placebo (Overall Cardiovascular Study); Test type: Superiority; p = 0.006, cLDA; The model had fixed effects for treatment, time, baseline eGFR (continuous) and the interaction of time by treatment; Difference in the Least Squares Means = -0.71, 95% CI 2-sided [-1.22 to -0.20]

63. Secondary Outcome: Change From Baseline in Sitting Diastolic Blood Pressure (DBP) at Month 36 (Overall Cardiovascular Study)
Description: This change from baseline reflects the Month 36 DBP minus the Week 0 DBP. A negative number indicates a reduction in DBP. Participants who met glycemic rescue criteria received glycemic rescue medication.
Time Frame: Baseline and Month 36
Population: as for outcome 21
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Ertugliflozin 5 mg (Overall Cardiovascular Study) | Ertugliflozin 15 mg (Overall Cardiovascular Study) | Placebo (Overall Cardiovascular Study)
Number analyzed (Participants) | 1593 | 1580 | 1505
mmHg | -1.27 (8.94) | -0.92 (8.89) | -0.22 (9.15)

64. Secondary Outcome: Change From Baseline in Sitting Diastolic Blood Pressure (DBP) at Month 48 (Overall Cardiovascular Study)
Description: This change from baseline reflects the Month 48 DBP minus the Week 0 DBP. A negative number indicates a reduction in DBP. Participants who met glycemic rescue criteria received glycemic rescue medication.
Time Frame: Baseline and Month 48
Population: The analysis population included all participants who were randomized, received at least one dose of blinded study medication, and had a measurement for the analysis endpoint for the specified timepoint(s) at or after Baseline.
Measure: Mean (95% Confidence Interval); unit: mmHg
Arm/Group | Ertugliflozin 5 mg (Overall Cardiovascular Study) | Ertugliflozin 15 mg (Overall Cardiovascular Study) | Placebo (Overall Cardiovascular Study)
Number analyzed (Participants) | 881 | 868 | 789
mmHg | -1.45 [-1.93 to -0.97] | -1.42 [-1.90 to -0.94] | -0.64 [-1.14 to -0.14]
Statistical Analysis 1: Comparison: Ertugliflozin 15 mg (Overall Cardiovascular Study) vs Placebo (Overall Cardiovascular Study); Test type: Superiority; p = 0.024, Constrained longitudinal data analysis — cLDA model with fixed effects for treatment, time, baseline eGFR (continuous) and the interaction of time by treatment. Time was treated as a categorical variable; Difference in the least squares means = -0.78, 95% CI 2-sided [-1.46 to -0.10]
Statistical Analysis 2: Comparison: Ertugliflozin 5 mg (Overall Cardiovascular Study) vs Placebo (Overall Cardiovascular Study); Test type: Superiority; p = 0.020, Constrained longitudinal data analysis — [p-value comment as in outcome 64, analysis 1]; Difference in the least squares means = -0.81, 95% CI 2-sided [-1.48 to -0.13]

65. Secondary Outcome: Change From Baseline in Sitting Diastolic Blood Pressure (DBP) at Month 60 (Overall Cardiovascular Study)
Description: This change from baseline reflects the Month 60 DBP minus the Week 0 DBP. A negative number indicates a reduction in DBP. Participants who met glycemic rescue criteria received glycemic rescue medication.
Time Frame: Baseline and Month 60
Population: as for outcome 23
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Ertugliflozin 5 mg (Overall Cardiovascular Study) | Ertugliflozin 15 mg (Overall Cardiovascular Study) | Placebo (Overall Cardiovascular Study)
Number analyzed (Participants) | 525 | 529 | 479
mmHg | -1.82 (8.66) | -1.43 (9.36) | -1.26 (9.38)

66. Secondary Outcome: Change From Baseline in Sitting Diastolic Blood Pressure (DBP) at Month 72 (Overall Cardiovascular Study)
Description: This change from baseline reflects the Month 72 DBP minus the Week 0 DBP. A negative number indicates a reduction in DBP. Participants who met glycemic rescue criteria received glycemic rescue medication.
Time Frame: Baseline and Month 72
Population: The analysis population included all participants who were randomized, received at least one dose of blinded study medication, and had a measurement for the analysis endpoint for the specified timepoint(s) at both Baseline and time point.
Measure: Mean (95% Confidence Interval); unit: mmHg
Arm/Group | Ertugliflozin 5 mg (Overall Cardiovascular Study) | Ertugliflozin 15 mg (Overall Cardiovascular Study) | Placebo (Overall Cardiovascular Study)
Number analyzed (Participants) | 13 | 12 | 9
mmHg | -2.18 [-7.65 to 3.29] | 1.86 [-2.73 to 6.45] | 7.29 [1.63 to 12.94]

67. Secondary Outcome: Change From Baseline in Body Weight at Week 18 (Excluding Rescue Approach) (Overall Cardiovascular Study)
Description: This change from baseline reflects the Week 18 body weight minus the Week 0 body weight. A negative number indicates a reduction in body weight. Participants who met glycemic rescue criteria received glycemic rescue medication. "Excluding Rescue" excluded all data following the initiation of rescue in order to avoid the confounding influence of the rescue therapy.
Time Frame: Baseline and Week 18
Population: The analysis population included all participants who were randomized, received at least one dose of blinded study medication, and have at least and had at least one measurement for the analysis endpoint for the specified timepoint(s) at or after Baseline.
Measure: Least Squares Mean (95% Confidence Interval); unit: Kilograms
Arm/Group | Ertugliflozin 5 mg (Overall Cardiovascular Study) | Ertugliflozin 15 mg (Overall Cardiovascular Study) | Placebo (Overall Cardiovascular Study)
Number analyzed (Participants) | 2746 | 2746 | 2745
Kilograms | -2.03 [-2.14 to -1.92] | -2.32 [-2.43 to -2.22] | -0.40 [-0.51 to -0.30]
Statistical Analysis 1: Comparison: Ertugliflozin 15 mg (Overall Cardiovascular Study) vs Placebo (Overall Cardiovascular Study); Test type: Superiority; p < 0.001, cLDA; cLDA model with fixed effects for treatment, time, baseline eGFR (continuous) and the interaction of time by treatment; Difference in the Least Squares Means = -1.92, 95% CI 2-sided [-2.07 to -1.77]
Statistical Analysis 2: Comparison: Ertugliflozin 5 mg (Overall Cardiovascular Study) vs Placebo (Overall Cardiovascular Study); Test type: Superiority; p < 0.001, cLDA; cLDA model with fixed effects for treatment, time, baseline eGFR (continuous) and the interaction of time by treatment; Difference in the Least Squares Means = -1.63, 95% CI 2-sided [-1.78 to -1.47]

68. Secondary Outcome: Change From Baseline in Body Weight at Week 52 (Overall Cardiovascular Study)
Description: This change from baseline reflects the Week 52 body weight minus the Week 0 body weight. A negative number indicates a reduction in body weight. Participants who met glycemic rescue criteria received glycemic rescue medication.
Time Frame: Baseline and Week 52
Population: as for outcome 37
Measure: Least Squares Mean (95% Confidence Interval); unit: Kilograms
Arm/Group | Ertugliflozin 5 mg (Overall Cardiovascular Study) | Ertugliflozin 15 mg (Overall Cardiovascular Study) | Placebo (Overall Cardiovascular Study)
Number analyzed (Participants) | 2746 | 2746 | 2745
Kilograms | -2.46 [-2.61 to -2.31] | -2.84 [-2.99 to -2.69] | -0.39 [-0.54 to -0.24]
Statistical Analysis 1: Comparison: Ertugliflozin 15 mg (Overall Cardiovascular Study) vs Placebo (Overall Cardiovascular Study); Test type: Superiority; p < 0.001, cLDA; cLDA model with fixed effects for treatment, time, baseline eGFR (continuous) and the interaction of time by treatment; Difference in the Least Squares Means = -2.45, 95% CI 2-sided [-2.67 to -2.24]
Statistical Analysis 2: Comparison: Ertugliflozin 5 mg (Overall Cardiovascular Study) vs Placebo (Overall Cardiovascular Study); Test type: Superiority; p < 0.001, cLDA; cLDA model with fixed effects for treatment, time, baseline eGFR (continuous) and the interaction of time by treatment; Difference in the Least Squares Means = -2.07, 95% CI 2-sided [-2.28 to -1.86]

69. Secondary Outcome: Change From Baseline in Body Weight at Month 24 (Overall Cardiovascular Study)
Description: This change from baseline reflects the Month 24 body weight minus the Week 0 body weight. A negative number indicates a reduction in body weight. Participants who met glycemic rescue criteria received glycemic rescue medication.
Time Frame: Baseline and Month 24
Population: as for outcome 37
Measure: Least Squares Mean (95% Confidence Interval); unit: Kilograms
Arm/Group | Ertugliflozin 5 mg (Overall Cardiovascular Study) | Ertugliflozin 15 mg (Overall Cardiovascular Study) | Placebo (Overall Cardiovascular Study)
Number analyzed (Participants) | 2746 | 2746 | 2745
Kilograms | -2.75 [-2.95 to -2.56] | -3.17 [-3.39 to -2.95] | -0.65 [-0.85 to -0.44]
Statistical Analysis 1: Comparison: Ertugliflozin 15 mg (Overall Cardiovascular Study) vs Placebo (Overall Cardiovascular Study); Test type: Superiority; p < 0.001, cLDA; cLDA model with fixed effects for treatment, time, baseline eGFR (continuous) and the interaction of time by treatment; Difference in the Least Squares Means = -2.53, 95% CI 2-sided [-2.83 to -2.22]
Statistical Analysis 2: Comparison: Ertugliflozin 5 mg (Overall Cardiovascular Study) vs Placebo (Overall Cardiovascular Study); Test type: Superiority; p < 0.001, cLDA; cLDA model with fixed effects for treatment, time, baseline eGFR (continuous) and the interaction of time by treatment; Difference in the Least Squares Means = -2.11, 95% CI 2-sided [-2.39 to -1.83]

70. Secondary Outcome: Change From Baseline in Body Weight at Month 36 (Overall Cardiovascular Study)
Description: This change from baseline reflects the Month 36 body weight minus the Week 0 body weight. A negative number indicates a reduction in body weight. Participants who met glycemic rescue criteria received glycemic rescue medication.
Time Frame: Baseline and Month 36
Population: The analysis population included all participants who were randomized, received at least one dose of blinded study medication, and have at least one measurement for the analysis endpoint for the specified timepoint(s) at both Baseline and Month 36.
Measure: Mean (95% Confidence Interval); unit: Kilograms
Arm/Group | Ertugliflozin 5 mg (Overall Cardiovascular Study) | Ertugliflozin 15 mg (Overall Cardiovascular Study) | Placebo (Overall Cardiovascular Study)
Number analyzed (Participants) | 1595 | 1578 | 1506
Kilograms | -3.03 [-3.24 to -2.82] | -3.41 [-3.63 to -3.20] | -0.98 [-1.20 to -0.77]

71. Secondary Outcome: Change From Baseline in Body Weight at Month 48 (Overall Cardiovascular Study)
Description: This change from baseline reflects the Month 48 body weight minus the Week 0 body weight. A negative number indicates a reduction in body weight. Participants who met glycemic rescue criteria received glycemic rescue medication.
Time Frame: Baseline and Month 48
Population: The analysis population included all participants who were randomized, received at least one dose of blinded study medication, and had at least one measurement for the analysis endpoint for the specified timepoint(s) at or after baseline).
Measure: Least Squares Mean (95% Confidence Interval); unit: Kilograms
Arm/Group | Ertugliflozin 5 mg (Overall Cardiovascular Study) | Ertugliflozin 15 mg (Overall Cardiovascular Study) | Placebo (Overall Cardiovascular Study)
Number analyzed (Participants) | 2746 | 2746 | 2745
Kilograms | -3.39 [-3.69 to -3.10] | -3.83 [-4.14 to -3.51] | -1.29 [-1.59 to -1.00]
Statistical Analysis 1: Comparison: Ertugliflozin 15 mg (Overall Cardiovascular Study) vs Placebo (Overall Cardiovascular Study); Test type: Superiority; p < 0.001, cLDA; cLDA model with fixed effects for treatment, time, baseline eGFR (continuous) and the interaction of time by treatment; Difference in the Least Squares Means = -2.53, 95% CI 2-sided [-2.97 to -2.10]
Statistical Analysis 2: Comparison: Ertugliflozin 5 mg (Overall Cardiovascular Study) vs Placebo (Overall Cardiovascular Study); Test type: Superiority; p < 0.001, cLDA; cLDA model with fixed effects for treatment, time, baseline eGFR (continuous) and the interaction of time by treatment; Difference in the Least Squares Means = -2.10, 95% CI 2-sided [-2.52 to -1.68]

72. Secondary Outcome: Change From Baseline in Body Weight at Month 60 (Overall Cardiovascular Study)
Description: This change from baseline reflects the Month 60 body weight minus the Week 0 body weight. A negative number indicates a reduction in body weight. Participants who met glycemic rescue criteria received glycemic rescue medication.
Time Frame: Baseline and Month 60
Population: as for outcome 23
Measure: Mean (95% Confidence Interval); unit: Kilograms
Arm/Group | Ertugliflozin 5 mg (Overall Cardiovascular Study) | Ertugliflozin 15 mg (Overall Cardiovascular Study) | Placebo (Overall Cardiovascular Study)
Number analyzed (Participants) | 526 | 530 | 478
Kilograms | -3.66 [-4.11 to -3.20] | -4.58 [-5.06 to -4.11] | -1.21 [-1.63 to -0.78]

73. Secondary Outcome: Change From Baseline in Body Weight at Month 72 (Overall Cardiovascular Study)
Description: This change from baseline reflects the Month 72 body weight minus the Week 0 body weight. A negative number indicates a reduction in body weight. Participants who met glycemic rescue criteria received glycemic rescue medication.
Time Frame: Baseline and Month 72
Population: as for outcome 24
Measure: Mean (95% Confidence Interval); unit: Kilograms
Arm/Group | Ertugliflozin 5 mg (Overall Cardiovascular Study) | Ertugliflozin 15 mg (Overall Cardiovascular Study) | Placebo (Overall Cardiovascular Study)
Number analyzed (Participants) | 13 | 12 | 9
Kilograms | -4.18 [-7.83 to -0.53] | -7.37 [-12.67 to -2.07] | -0.98 [-4.13 to 2.18]

74. Secondary Outcome: Change From Baseline in Estimated Glomerular Filtration Rate (eGFR) at Week 18 (Overall Cardiovascular Study)
Description: This change from baseline reflects the Week 18 eGFR minus the Week 0 eGFR. A negative number indicates a reduction in the eGFR level.
Time Frame: Baseline and Week 18
Population: The analysis population included all participants who were randomized, received at least one dose of blinded study medication, and at least one measurement for the analysis endpoint for the specified timepoint(s) at or after Baseline.
Measure: Least Squares Mean (95% Confidence Interval); unit: mL/min/1.73 m^2
Arm/Group | Ertugliflozin 5 mg (Overall Cardiovascular Study) | Ertugliflozin 15 mg (Overall Cardiovascular Study) | Placebo (Overall Cardiovascular Study)
Number analyzed (Participants) | 2671 | 2667 | 2661
mL/min/1.73 m^2 | -1.22 [-1.66 to -0.77] | -1.81 [-2.26 to -1.36] | -0.03 [-0.48 to 0.42]
Statistical Analysis 1: Comparison: Ertugliflozin 15 mg (Overall Cardiovascular Study); Test type: Superiority; Difference in the Lease Squares Means = -1.78, 95% CI 2-sided [-2.41 to -1.15]; Based on cLDA model with fixed effects for treatment, time, baseline eGFR (continuous) and the interaction of time by treatment. Time was treated as a categorical variable
Statistical Analysis 2: Comparison: Ertugliflozin 5 mg (Overall Cardiovascular Study) vs Placebo (Overall Cardiovascular Study); Test type: Superiority; Difference in the Least Squares Means = -1.19, 95% CI 2-sided [-1.82 to -0.56]; [other analysis details as in outcome 74, analysis 1]

75. Secondary Outcome: Change From Baseline in Estimated Glomerular Filtration Rate (eGFR) at Week 52 (Overall Cardiovascular Study)
Description: This change from baseline reflects the Week 52 eGFR minus the Week 0 eGFR. A negative number indicates a reduction in eGFR level.
Time Frame: Baseline and Week 52
Population: The analysis population included all participants who were randomized, received at least one dose of blinded study medication, and had for the analysis endpoint for the specified timepoint(s) a Baseline measurement and at least one measurement at or after Baseline.
Measure: Least Squares Mean (95% Confidence Interval); unit: mL/min/1.73 m^2
Arm/Group | Ertugliflozin 5 mg (Overall Cardiovascular Study) | Ertugliflozin 15 mg (Overall Cardiovascular Study) | Placebo (Overall Cardiovascular Study)
Number analyzed (Participants) | 2671 | 2669 | 2664
mL/min/1.73 m^2 | -0.51 [-1.01 to -0.02] | -1.18 [-1.67 to -0.68] | -0.30 [-0.80 to 0.20]
Statistical Analysis 1: Comparison: Ertugliflozin 15 mg (Overall Cardiovascular Study); Test type: Superiority; Difference in the Lease Squares Means = -0.88, 95% CI 2-sided [-1.58 to -0.18]; [other analysis details as in outcome 74, analysis 1]
Statistical Analysis 2: Comparison: Ertugliflozin 5 mg (Overall Cardiovascular Study) vs Placebo (Overall Cardiovascular Study); Test type: Superiority; Difference in the Least Squares Means = -0.21, 95% CI 2-sided [-0.91 to 0.49]; [other analysis details as in outcome 74, analysis 1]

76. Secondary Outcome: Change From Baseline in Estimated Glomerular Filtration Rate (eGFR) at Month 24 (Overall Cardiovascular Study)
Description: This change from baseline reflects the Month 24 eGFR minus the Week 0 eGFR. A negative number indicates a reduction in the eGFR level.
Time Frame: Baseline and Month 24
Population: The analysis population included all participants who were randomized, received at least one dose of blinded study medication, and had a measurement for the analysis endpoint for the specified timepoint(s) at both Baseline at or after Baseline.
Measure: Mean (95% Confidence Interval); unit: mL/min/1.73 m^2
Arm/Group | Ertugliflozin 5 mg (Overall Cardiovascular Study) | Ertugliflozin 15 mg (Overall Cardiovascular Study) | Placebo (Overall Cardiovascular Study)
Number analyzed (Participants) | 1576 | 1547 | 1509
mL/min/1.73 m^2 | -1.48 [-2.07 to -0.90] | -2.35 [-2.94 to -1.76] | -2.60 [-3.20 to -2.01]
Statistical Analysis 1: Comparison: Ertugliflozin 15 mg (Overall Cardiovascular Study) vs Placebo (Overall Cardiovascular Study); Test type: Superiority; Difference in the least squares means = 0.25, 95% CI 2-sided [-0.59 to 1.08] — Constrained longitudinal data analysis (cLDA) model with fixed effects for treatment, time, baseline eGFR (continuous) and the interaction of time by treatment. Time was treated as a categorical variable
Statistical Analysis 2: Comparison: Ertugliflozin 5 mg (Overall Cardiovascular Study) vs Placebo (Overall Cardiovascular Study); Test type: Superiority; Difference in the least squares means = 1.12, 95% CI 2-sided [0.28 to 1.95] — [estimate comment as in outcome 76, analysis 1]

77. Secondary Outcome: Change From Baseline in Estimated Glomerular Filtration Rate (eGFR) at Month 36 (Overall Cardiovascular Study)
Description: This change from baseline reflects the Month 36 eGFR minus the Week 0 eGFR. A negative number indicates a reduction in the eGFR level.
Time Frame: Baseline and Month 36
Population: as for outcome 21
Measure: Mean (Standard Deviation); unit: mL/min/1.73 m^2
Arm/Group | Ertugliflozin 5 mg (Overall Cardiovascular Study) | Ertugliflozin 15 mg (Overall Cardiovascular Study) | Placebo (Overall Cardiovascular Study)
Number analyzed (Participants) | 1591 | 1577 | 1504
mL/min/1.73 m^2 | -2.4 (14.0) | -2.3 (13.4) | -3.8 (14.1)

78. Secondary Outcome: Change From Baseline in Estimated Glomerular Filtration Rate (eGFR) at Month 48 (Overall Cardiovascular Study)
Description: This change from baseline reflects the Month 48 eGFR minus the Week 0 eGFR. A negative number indicates a reduction in eGFR level.
Time Frame: Baseline and Month 48
Population: The analysis population included all participants who were randomized, received at least one dose of blinded study medication, and had for the analysis endpoint for the specified timepoint(s) a Baseline measurement and at least one assessment at or after Baseline.
Measure: Least Squares Mean (95% Confidence Interval); unit: mL/min/1.73 m^2
Arm/Group | Ertugliflozin 5 mg (Overall Cardiovascular Study) | Ertugliflozin 15 mg (Overall Cardiovascular Study) | Placebo (Overall Cardiovascular Study)
Number analyzed (Participants) | 2671 | 2669 | 2665
mL/min/1.73 m^2 | -2.75 [-3.56 to -1.94] | -2.93 [-3.73 to -2.13] | -4.41 [-5.27 to -3.55]
Statistical Analysis 1: Comparison: Ertugliflozin 15 mg (Overall Cardiovascular Study); Test type: Superiority; Difference in the Lease Squares Means = 1.48, 95% CI 2-sided [0.31 to 2.66]; [other analysis details as in outcome 74, analysis 1]
Statistical Analysis 2: Comparison: Ertugliflozin 5 mg (Overall Cardiovascular Study) vs Placebo (Overall Cardiovascular Study); Test type: Superiority; Difference in the Least Squares Means = 1.66, 95% CI 2-sided [0.49 to 2.84]; [other analysis details as in outcome 74, analysis 1]

79. Secondary Outcome: Change From Baseline in Estimated Glomerular Filtration Rate (eGFR) at Month 60 (Overall Cardiovascular Study)
Description: This change from baseline reflects the Month 60 eGFR minus the Week 0 eGFR. A negative number indicates a reduction in the eGFR level.
Time Frame: Baseline and Month 60
Population: as for outcome 23
Measure: Mean (Standard Deviation); unit: mL/min/1.73 m^2
Arm/Group | Ertugliflozin 5 mg (Overall Cardiovascular Study) | Ertugliflozin 15 mg (Overall Cardiovascular Study) | Placebo (Overall Cardiovascular Study)
Number analyzed (Participants) | 520 | 529 | 477
mL/min/1.73 m^2 | -2.4 (15.4) | -2.9 (14.1) | -6.8 (14.3)

80. Secondary Outcome: Change From Baseline in Estimated Glomerular Filtration Rate (eGFR) at Month 72 (Overall Cardiovascular Study)
Description: This change from baseline reflects the Month 72 eGFR minus the Week 0 eGFR. A negative number indicates a reduction in the eGFR level.
Time Frame: Baseline and Month 72
Population: as for outcome 66
Measure: Mean (Standard Deviation); unit: mL/min/1.73 m^2
Arm/Group | Ertugliflozin 5 mg (Overall Cardiovascular Study) | Ertugliflozin 15 mg (Overall Cardiovascular Study) | Placebo (Overall Cardiovascular Study)
Number analyzed (Participants) | 12 | 12 | 9
mL/min/1.73 m^2 | 3.7 (12.9) | 0.2 (12.2) | -1.8 (14.1)

81. Secondary Outcome: Baseline Serum Creatinine (Overall Cardiovascular Study)
Description: Baseline reflects Week 0 serum creatinine.
Time Frame: Baseline
Population: The analysis population included all participants who were randomized and had a measurement for the analysis endpoint for the specified timepoint at Baseline.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Ertugliflozin 5 mg (Overall Cardiovascular Study) | Ertugliflozin 15 mg (Overall Cardiovascular Study) | Placebo (Overall Cardiovascular Study) | All Ertugliflozin (Overall Cardiovascular Study)
Number analyzed (Participants) | 2739 | 2740 | 2736 | 5479
mg/dL | 0.992 (0.278) | 0.985 (0.277) | 0.991 (0.281) | 0.998 (0.278)

82. Secondary Outcome: Change From Baseline in Serum Creatinine at Week 18 (Overall Cardiovascular Study)
Description: This change from baseline reflects the Week 18 serum creatinine minus the Week 0 serum creatinine. Participants who met glycemic rescue criteria received glycemic rescue medication.
Time Frame: Baseline and Week 18
Population: The analysis population included all participants who were randomized, received at least one dose of blinded study medication, and had a measurement for the analysis endpoint for the specified timepoint(s) at both Baseline and Week 18.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Ertugliflozin 5 mg (Overall Cardiovascular Study) | Ertugliflozin 15 mg (Overall Cardiovascular Study) | Placebo (Overall Cardiovascular Study)
Number analyzed (Participants) | 2540 | 2520 | 2524
mg/dL | 0.022 (0.154) | 0.032 (0.148) | -0.002 (0.138)

83. Secondary Outcome: Change From Baseline in Serum Creatinine at Week 52 (Overall Cardiovascular Study)
Description: This change from baseline reflects the Week 52 serum creatinine minus the Week 0 serum creatinine. Participants who met glycemic rescue criteria received glycemic rescue medication.
Time Frame: Baseline and Week 52
Population: as for outcome 38
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Ertugliflozin 5 mg (Overall Cardiovascular Study) | Ertugliflozin 15 mg (Overall Cardiovascular Study) | Placebo (Overall Cardiovascular Study)
Number analyzed (Participants) | 2360 | 2344 | 2314
mg/dL | 0.013 (0.166) | 0.023 (0.163) | 0.004 (0.156)

84. Secondary Outcome: Change From Baseline in Serum Creatinine at Month 24 (Overall Cardiovascular Study)
Description: This change from baseline reflects the Month 24 serum creatinine minus the Week 0 serum creatinine. Participants who met glycemic rescue criteria received glycemic rescue medication.
Time Frame: Baseline and Month 24
Population: as for outcome 39
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Ertugliflozin 5 mg (Overall Cardiovascular Study) | Ertugliflozin 15 mg (Overall Cardiovascular Study) | Placebo (Overall Cardiovascular Study)
Number analyzed (Participants) | 1574 | 1548 | 1506
mg/dL | 0.024 (0.176) | 0.035 (0.187) | 0.034 (0.197)

85. Secondary Outcome: Change From Baseline in Serum Creatinine at Month 36 (Overall Cardiovascular Study)
Description: This change from baseline reflects the Month 36 serum creatinine minus the Week 0 serum creatinine. Participants who met glycemic rescue criteria received glycemic rescue medication.
Time Frame: Baseline and Month 36
Population: as for outcome 21
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Ertugliflozin 5 mg (Overall Cardiovascular Study) | Ertugliflozin 15 mg (Overall Cardiovascular Study) | Placebo (Overall Cardiovascular Study)
Number analyzed (Participants) | 1589 | 1575 | 1499
mg/dL | 0.037 (0.194) | 0.035 (0.188) | 0.049 (0.194)

86. Secondary Outcome: Change From Baseline in Serum Creatinine at Month 48 (Overall Cardiovascular Study)
Description: This change from baseline reflects the Month 48 serum creatinine minus the Week 0 serum creatinine. Participants who met glycemic rescue criteria received glycemic rescue medication.
Time Frame: Baseline and Month 48
Population: as for outcome 41
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Ertugliflozin 5 mg (Overall Cardiovascular Study) | Ertugliflozin 15 mg (Overall Cardiovascular Study) | Placebo (Overall Cardiovascular Study)
Number analyzed (Participants) | 875 | 865 | 787
mg/dL | 0.032 (0.206) | 0.036 (0.196) | 0.059 (0.210)

87. Secondary Outcome: Change From Baseline in Serum Creatinine at Month 60 (Overall Cardiovascular Study)
Description: This change from baseline reflects the Month 60 serum creatinine minus the Week 0 serum creatinine. Participants who met glycemic rescue criteria received glycemic rescue medication.
Time Frame: Baseline and Month 60
Population: as for outcome 23
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Ertugliflozin 5 mg (Overall Cardiovascular Study) | Ertugliflozin 15 mg (Overall Cardiovascular Study) | Placebo (Overall Cardiovascular Study)
Number analyzed (Participants) | 518 | 528 | 476
mg/dL | 0.027 (0.202) | 0.042 (0.216) | 0.098 (0.248)

88. Secondary Outcome: Change From Baseline in Serum Creatinine at Month 72 (Overall Cardiovascular Study)
Description: This change from baseline reflects the Month 72 serum creatinine minus the Week 0 serum creatinine. Participants who met glycemic rescue criteria received glycemic rescue medication.
Time Frame: Baseline and Month 72
Population: as for outcome 24
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Ertugliflozin 5 mg (Overall Cardiovascular Study) | Ertugliflozin 15 mg (Overall Cardiovascular Study) | Placebo (Overall Cardiovascular Study)
Number analyzed (Participants) | 12 | 12 | 9
mg/dL | -0.034 (0.176) | 0.001 (0.120) | -0.013 (0.162)

89. Secondary Outcome: Baseline Urinary Albumin/Creatinine Ratio (Overall Cardiovascular Study)
Description: Baseline reflects Week 0 albumin/creatinine ratio.
Time Frame: Baseline
Population: as for outcome 81
Measure: Median (Inter-Quartile Range); unit: mg/g
Arm/Group | Ertugliflozin 5 mg (Overall Cardiovascular Study) | Ertugliflozin 15 mg (Overall Cardiovascular Study) | Placebo (Overall Cardiovascular Study)
Number analyzed (Participants) | 2686 | 2660 | 2684
mg/g | 18.00 [6.00 to 68.00] | 19.00 [6.00 to 69.00] | 19.00 [6.00 to 66.50]

90. Secondary Outcome: Percent Change From Baseline in Urinary Albumin/Creatinine Ratio at Week 18 (Overall Cardiovascular Study)
Description: This percent change relative to baseline reflects the Week 18 albumin/creatinine ratio minus the Week 0 albumin/creatinine ratio. This difference was divided by the baseline to obtain the percent change. A negative number indicates a reduction in the urinary albumin/creatinine ratio. Participants who met glycemic rescue criteria received glycemic rescue medication.
Time Frame: Baseline and Week 18
Population: as for outcome 82
Measure: Median (Inter-Quartile Range); unit: Percent Change
Arm/Group | Ertugliflozin 5 mg (Overall Cardiovascular Study) | Ertugliflozin 15 mg (Overall Cardiovascular Study) | Placebo (Overall Cardiovascular Study)
Number analyzed (Participants) | 2472 | 2450 | 2478
Percent Change | -13.40 [-53.52 to 50.00] | -14.71 [-55.53 to 50.00] | 0.00 [-44.44 to 66.67]

91. Secondary Outcome: Percent Change From Baseline in Urinary Albumin/Creatinine Ratio at Week 52 (Overall Cardiovascular Study)
Description: This percent change relative to baseline reflects the Week 52 albumin/creatinine ratio minus the Week 0 albumin/creatinine ratio. This difference was divided by the baseline to obtain the percent change. A negative number indicates a reduction in the albumin/creatinine ratio. Participants who met glycemic rescue criteria received glycemic rescue medication.
Time Frame: Baseline and Week 52
Population: as for outcome 38
Measure: Median (Inter-Quartile Range); unit: Percent Change
Arm/Group | Ertugliflozin 5 mg (Overall Cardiovascular Study) | Ertugliflozin 15 mg (Overall Cardiovascular Study) | Placebo (Overall Cardiovascular Study)
Number analyzed (Participants) | 2306 | 2277 | 2257
Percent Change | -2.53 [-50.00 to 66.67] | -6.82 [-50.00 to 66.67] | 5.41 [-40.00 to 96.34]

92. Secondary Outcome: Percent Change From Baseline in Urinary Albumin/Creatinine Ratio at Month 24 (Overall Cardiovascular Study)
Description: This percent change relative to baseline reflects the Month 24 albumin/creatinine ratio minus the Week 0 albumin/creatinine ratio. This difference was divided by the baseline to obtain the percent change. A negative number indicates a reduction in urinary albumin/creatinine ratio. Participants who met glycemic rescue criteria received glycemic rescue medication.
Time Frame: Baseline and Month 24
Population: as for outcome 39
Measure: Median (Inter-Quartile Range); unit: Percent Change
Arm/Group | Ertugliflozin 5 mg (Overall Cardiovascular Study) | Ertugliflozin 15 mg (Overall Cardiovascular Study) | Placebo (Overall Cardiovascular Study)
Number analyzed (Participants) | 2125 | 2084 | 2025
Percent Change | -0.73 [-48.96 to 100.00] | 1.06 [-47.78 to 95.26] | 17.14 [-38.00 to 140.00]

93. Secondary Outcome: Percent Change From Baseline in Urinary Albumin/Creatinine Ratio at Month 36 (Overall Cardiovascular Study)
Description: This percent change relative to baseline reflects the Month 36 albumin/creatinine ratio minus the Week 0 albumin/creatinine ratio. This difference was divided by the baseline to obtain the percent change. A negative number indicates a reduction in urinary albumin/creatinine ratio. Participants who met glycemic rescue criteria received glycemic rescue medication.
Time Frame: Baseline and Month 36
Population: as for outcome 21
Measure: Median (Inter-Quartile Range); unit: Percent Change
Arm/Group | Ertugliflozin 5 mg (Overall Cardiovascular Study) | Ertugliflozin 15 mg (Overall Cardiovascular Study) | Placebo (Overall Cardiovascular Study)
Number analyzed (Participants) | 1933 | 1915 | 1841
Percent Change | 13.33 [-49.34 to 120.37] | 3.33 [-49.44 to 100.00] | 27.03 [-38.46 to 177.78]

94. Secondary Outcome: Percent Change From Baseline in Urinary Albumin/Creatinine Ratio at Month 48 (Overall Cardiovascular Study)
Description: This percent change relative to baseline reflects the Month 48 albumin/creatinine ratio minus the Week 0 albumin/creatinine ratio. This difference was divided by the baseline to obtain the percent change. A negative number indicates a reduction in albumin/creatinine ratio. Participants who met glycemic rescue criteria received glycemic rescue medication.
Time Frame: Baseline and Month 48
Population: as for outcome 41
Measure: Median (Inter-Quartile Range); unit: Percent Change
Arm/Group | Ertugliflozin 5 mg (Overall Cardiovascular Study) | Ertugliflozin 15 mg (Overall Cardiovascular Study) | Placebo (Overall Cardiovascular Study)
Number analyzed (Participants) | 825 | 835 | 745
Percent Change | 33.33 [-36.84 to 200.00] | 21.25 [-42.86 to 150.00] | 50.00 [-33.33 to 227.27]

95. Secondary Outcome: Percent Change From Baseline in Urinary Albumin/Creatinine Ratio at Month 60 (Overall Cardiovascular Study)
Description: This percent change relative to baseline reflects the Month 60 albumin/creatinine ratio minus the Week 0 albumin/creatinine ratio. This difference was divided by the baseline to obtain the percent change. A negative number indicates a reduction in albumin/creatinine ratio. Participants who met glycemic rescue criteria received glycemic rescue medication.
Time Frame: Baseline and Month 60
Population: as for outcome 23
Measure: Median (Inter-Quartile Range); unit: Percent Change
Arm/Group | Ertugliflozin 5 mg (Overall Cardiovascular Study) | Ertugliflozin 15 mg (Overall Cardiovascular Study) | Placebo (Overall Cardiovascular Study)
Number analyzed (Participants) | 780 | 771 | 692
Percent Change | 30.99 [-40.00 to 200.00] | 20.00 [-45.83 to 150.00] | 48.53 [-28.57 to 222.41]

96. Secondary Outcome: Percentage of Participants With Albuminuria Progression or Regression at Week 18 (Overall Cardiovascular Study)
Description: Albuminuria progression and regression were assessed relative to the baseline albuminuria category. Progression was defined as either a change from having normal-albuminuria at baseline to micro-albuminuria at the respective visit, or micro-albuminuria at baseline to macro-albuminuria at the respective visit, or normal albuminuria at baseline to macro-albuminuria at the respective visit. Regression was defined as either a change from having micro-albuminuria at baseline to normal albuminuria at the respective visit, or macro-albuminuria at baseline to micro-albuminuria at the respective visit, or macro-albuminuria at baseline to normal albuminuria at the respective visit. Normal albuminuria: urine albumin to urinary creatinine ratio (UACR) <30 (mg/g); Micro-albuminuria: UACR ≥30 and ≤300 (mg/g); Macro-albuminuria: UACR>300 (mg/g).
Time Frame: Week 18
Population: The analysis population included all participants who were randomized, received at least one dose of blinded study medication, had a baseline measurement, and at least one measurement for the analysis endpoint for the specified timepoint at Week 18.
Measure: Number; unit: Percentage of Participants
Arm/Group | Ertugliflozin 5 mg (Overall Cardiovascular Study) | Ertugliflozin 15 mg (Overall Cardiovascular Study) | Placebo (Overall Cardiovascular Study)
Number analyzed (Participants) | 2472 | 2450 | 2478
Percentage of Participants
  Percentage of Participants with albuminuria progression | 7.6 | 7.7 | 10.8
  Percentage of Participants with albuminuria regression | 14.9 | 14.7 | 10.7

97. Secondary Outcome: Percentage of Participants With Albuminuria Progression or Regression at Week 52 (Overall Cardiovascular Study)
Description: Albuminuria progression and regression were assessed relative to the baseline albuminuria category. Progression was defined as either a change from having normal albuminuria at baseline to micro-albuminuria at the respective visit, or micro-albuminuria at baseline to macro-albuminuria at the respective visit, or normal albuminuria at baseline to macro-albuminuria at the respective visit. Regression was defined as either a change from having micro-albuminuria at baseline to normal albuminuria at the respective visit, or macro-albuminuria at baseline to micro-albuminuria at the respective visit, or macro-albuminuria at baseline to normal albuminuria at the respective visit. Normal albuminuria: urine albumin to urinary creatinine ratio (UACR) <30 (mg/g); Micro-albuminuria: UACR ≥30 and ≤300 (mg/g); Macro-albuminuria: UACR>300 (mg/g).
Time Frame: Week 52
Population: The analysis population included all participants who were randomized, received at least one dose of blinded study medication, had a baseline measurement, and at least one measurement for the analysis endpoint for the specified timepoint at Week 52.
Measure: Number; unit: Percentage of Participants
Arm/Group | Ertugliflozin 5 mg (Overall Cardiovascular Study) | Ertugliflozin 15 mg (Overall Cardiovascular Study) | Placebo (Overall Cardiovascular Study)
Number analyzed (Participants) | 2306 | 2277 | 2257
Percentage of Participants
  Percentage of Participants with albuminuria progression | 9.5 | 10.2 | 12.9
  Percentage of Participants with albuminuria regression | 14.6 | 14.8 | 10.2

98. Secondary Outcome: Percentage of Participants With Albuminuria Progression or Regression at Month 24 (Overall Cardiovascular Study)
Description: as for outcome 97
Time Frame: Month 24
Population: The analysis population included all participants who were randomized, received at least one dose of blinded study medication, had a baseline measurement, and at least one measurement for the analysis endpoint for the specified timepoint at Month 24.
Measure: Number; unit: Percentage of Participants
Arm/Group | Ertugliflozin 5 mg (Overall Cardiovascular Study) | Ertugliflozin 15 mg (Overall Cardiovascular Study) | Placebo (Overall Cardiovascular Study)
Number analyzed (Participants) | 2125 | 2084 | 2025
Percentage of Participants
  Percentage of Participants with albuminuria progression | 12.1 | 11.0 | 16.9
  Percentage of Participants with albuminuria regression | 14.3 | 13.8 | 9.9

99. Secondary Outcome: Percentage of Participants With Albuminuria Progression or Regression at Month 36 (Overall Cardiovascular Study)
Description: as for outcome 97
Time Frame: Month 36
Population: The analysis population included all participants who were randomized, received at least one dose of blinded study medication, had a baseline measurement, and at least one measurement for the analysis endpoint for the specified timepoint at Month 36.
Measure: Number; unit: Percentage of Participants
Arm/Group | Ertugliflozin 5 mg (Overall Cardiovascular Study) | Ertugliflozin 15 mg (Overall Cardiovascular Study) | Placebo (Overall Cardiovascular Study)
Number analyzed (Participants) | 1933 | 1915 | 1841
Percentage of Participants
  Participants with albuminuria progression | 14.6 | 12.5 | 18.1
  Participants with albuminuria regression | 13.8 | 14.3 | 11.0

100. Secondary Outcome: Percentage of Participants With Albuminuria Progression or Regression at Month 48 (Overall Cardiovascular Study)
Description: Albuminuria progression and regression were assessed relative to the baseline albuminuria category. Progression was defined as either a change from having normal albuminuria at baseline to micro-albuminuria at the respective visit, or micro-albuminuria at baseline to macro-albuminuria at the respective visit, or normal albuminuria at baseline to macro-albuminuria at the respective visit. Regression was defined as either a change from having micro-albuminuria at baseline to normal albuminuria at the respective visit, or macro-albuminuria at baseline to micro-albuminuria at the respective visit, or macro-albuminuria at baseline and normal albuminuria at the respective visit. Normal albuminuria: urine albumin to urinary creatinine ratio (UACR) <30 (mg/g); Micro-albuminuria: UACR ≥30 and ≤300 (mg/g); Macro-albuminuria: UACR>300 (mg/g).
Time Frame: Month 48
Population: The analysis population included all participants who were randomized, received at least one dose of blinded study medication, had a baseline measurement, and at least one measurement for the analysis endpoint for the specified timepoint at Month 48.
Measure: Number; unit: Percentage of Participants
Arm/Group | Ertugliflozin 5 mg (Overall Cardiovascular Study) | Ertugliflozin 15 mg (Overall Cardiovascular Study) | Placebo (Overall Cardiovascular Study)
Number analyzed (Participants) | 825 | 835 | 745
Percentage of Participants
  Percentage of Participants with albuminuria progression | 19.5 | 14.9 | 21.5
  Percentage of Participants with albuminuria regression | 11.6 | 12.2 | 9.9

101. Secondary Outcome: Percentage of Participants With Albuminuria Progression or Regression at Month 60 (Overall Cardiovascular Study)
Description: Albuminuria progression and regression were assessed relative to the baseline albuminuria category. Progression was defined as either a change from having normal albuminuria at baseline to micro albuminuria at the respective visit, or micro-albuminuria at baseline to macro-albuminuria at the respective visit, or normal albuminuria at baseline to macro-albuminuria at the respective visit. Regression was defined as either a change from having micro-albuminuria at baseline to normal albuminuria at the respective visit, or macro-albuminuria at baseline to micro-albuminuria at the respective visit, or macro-albuminuria at baseline to normal albuminuria at the respective visit. Normal albuminuria: urine albumin to urinary creatinine ratio (UACR) <30 (mg/g); Micro-albuminuria: UACR ≥30 and ≤300 (mg/g); Macro-albuminuria: UACR>300 (mg/g).
Time Frame: Month 60
Population: The analysis population included all participants who were randomized, received at least one dose of blinded study medication, had a baseline measurement, and at least one measurement for the analysis endpoint for the specified timepoint at Month 60.
Measure: Number; unit: Percentage of Participants
Arm/Group | Ertugliflozin 5 mg (Overall Cardiovascular Study) | Ertugliflozin 15 mg (Overall Cardiovascular Study) | Placebo (Overall Cardiovascular Study)
Number analyzed (Participants) | 780 | 771 | 692
Percentage of Participants
  Percentage of Participants with albuminuria progression | 18.6 | 14.7 | 22.1
  Percentage of Participants with albuminuria regression | 11.3 | 14.8 | 10.5

102. Secondary Outcome: Percentage of Participants Experiencing an Adverse Event (AE) (Overall Cardiovascular Study)
Description: An AE is defined as any unfavorable and unintended sign including an abnormal laboratory finding, symptom or disease associated with the use of a medical treatment or procedure, regardless of whether it is considered related to the medical treatment or procedure, that occurs during the course of the study.
Time Frame: Up to approximately 6 years
Population: The analysis population included all participants who were randomized and who received at least one dose of blinded study medication.
Measure: Number; unit: Percentage of Participants
Arm/Group | Ertugliflozin 5 mg (Overall Cardiovascular Study) | Ertugliflozin 15 mg (Overall Cardiovascular Study) | Placebo (Overall Cardiovascular Study)
Number analyzed (Participants) | 2746 | 2747 | 2745
Percentage of Participants | 85.8 | 84.6 | 85.6
Statistical Analysis 1: Comparison: Ertugliflozin 15 mg (Overall Cardiovascular Study) vs Placebo (Overall Cardiovascular Study); Test type: Superiority; Difference in % vs Placebo = -0.9, 95% CI 2-sided [-2.8 to 0.9]; Miettinen & Nurminen method
Statistical Analysis 2: Comparison: Ertugliflozin 5 mg (Overall Cardiovascular Study) vs Placebo (Overall Cardiovascular Study); Test type: Superiority; Difference in % vs Placebo = 0.3, 95% CI 2-sided [-1.6 to 2.1]; Miettinen & Nurminen method

103. Secondary Outcome: Percentage of Participants Experiencing an Adverse Event (AE) (Insulin With or Without Metformin Add-on Glycemic Sub-study)
Description: as for outcome 102
Time Frame: Up to 18 weeks
Population: The analysis population included all participants who were randomized, participated in the Insulin +/- Metformin Glycemic Sub-study, and who received at least one dose of blinded study medication.
Measure: Number; unit: Percentage of Participants
Groups:
- Placebo (Insulin +/- Metformin Glycemic Sub-study): Matching placebo to ertugliflozin administered orally, once daily, for up to 18 weeks
Arm/Group | Ertugliflozin 5 mg (Insulin +/- Metformin Glycemic Sub-study) | Ertugliflozin 15 mg (Insulin +/- Metformin Glycemic Sub-study) | Placebo (Insulin +/- Metformin Glycemic Sub-study)
Number analyzed (Participants) | 348 | 370 | 347
Percentage of Participants | 59.2 | 62.4 | 61.1
Statistical Analysis 1: Comparison: Ertugliflozin 15 mg (Insulin +/- Metformin Glycemic Sub-study) vs Placebo (Insulin +/- Metformin Glycemic Sub-study); Test type: Superiority; Difference in % vs Placebo = 1.3, 95% CI 2-sided [-5.8 to 8.4]; Miettinen & Nurminen method
Statistical Analysis 2: Comparison: Ertugliflozin 5 mg (Insulin +/- Metformin Glycemic Sub-study) vs Placebo (Insulin +/- Metformin Glycemic Sub-study); Test type: Superiority; Difference in % vs Placebo = -1.9, 95% CI 2-sided [-9.2 to 5.4]; Miettinen & Nurminen method

104. Secondary Outcome: Percentage of Participants Experiencing an Adverse Event (AE) (Sulfonylurea Monotherapy Add-on Glycemic Sub-Study)
Description: as for outcome 102
Time Frame: Up to 18 weeks
Population: The analysis population included all participants who were randomized, participated in the Sulfonylurea Monotherapy Glycemic Sub-study, and who received at least one dose of blinded study medication.
Measure: Number; unit: Percentage of Participants
Arm/Group | Ertugliflozin 5 mg (Sulfonylurea Monotherapy Glycemic Sub-study) | Ertugliflozin 15 mg (Sulfonylurea Monotherapy Glycemic Sub-study) | Placebo (Sulfonylurea Monotherapy Glycemic Sub-study)
Number analyzed (Participants) | 55 | 54 | 48
Percentage of Participants | 47.3 | 25.9 | 45.8
Statistical Analysis 1: Comparison: Ertugliflozin 5 mg (Sulfonylurea Monotherapy Glycemic Sub-study) vs Placebo (Sulfonylurea Monotherapy Glycemic Sub-study); Test type: Superiority; Difference in % vs Placebo = 1.4, 95% CI 2-sided [-17.7 to 20.4]; Miettinen and Nurminen method
Statistical Analysis 2: Comparison: Ertugliflozin 15 mg (Sulfonylurea Monotherapy Glycemic Sub-study) vs Placebo (Sulfonylurea Monotherapy Glycemic Sub-study); Test type: Superiority; Difference in % vs Placebo = -19.9, 95% CI 2-sided [-37.5 to -1.2]; Miettinen and Nurminen method

105. Secondary Outcome: Percentage of Participants Experiencing an Adverse Event (AE) (Metformin With Sulfonylurea Add-on Glycemic Sub-study)
Description: as for outcome 102
Time Frame: Up to 18 weeks
Population: The analysis population included all participants who were randomized, participated in the Metformin with Sulfonylurea Glycemic Sub-study, and who received at least one dose of blinded study medication.
Measure: Number; unit: Percentage of Participants
Arm/Group | Ertugliflozin 5 mg (Metformin With Sulfonylurea Glycemic Sub-study) | Ertugliflozin 15 mg (Metformin With Sulfonylurea Glycemic Sub-study) | Placebo (Metformin With Sulfonylurea Glycemic Sub-study)
Number analyzed (Participants) | 100 | 113 | 117
Percentage of Participants | 48.0 | 54.9 | 47.0
Statistical Analysis 1: Comparison: Ertugliflozin 15 mg (Metformin With Sulfonylurea Glycemic Sub-study) vs Placebo (Metformin With Sulfonylurea Glycemic Sub-study); Test type: Superiority; Difference in % vs Placebo = 7.9, 95% CI 2-sided [-5.1 to 20.5]; Based on Miettinen and Nurminen method
Statistical Analysis 2: Comparison: Ertugliflozin 5 mg (Metformin With Sulfonylurea Glycemic Sub-study) vs Placebo (Metformin With Sulfonylurea Glycemic Sub-study); Test type: Superiority; Difference in % vs Placebo = 1.0, 95% CI 2-sided [-12.3 to 14.2]; Miettinen and Nurminen method

106. Secondary Outcome: Percentage of Participants Discontinuing Study Treatment Due to An AE (Overall Cardiovascular Study)
Description: as for outcome 102
Time Frame: Up to approximately 6 years
Population: as for outcome 102
Measure: Number; unit: Percentage of Participants
Arm/Group | Ertugliflozin 5 mg (Overall Cardiovascular Study) | Ertugliflozin 15 mg (Overall Cardiovascular Study) | Placebo (Overall Cardiovascular Study)
Number analyzed (Participants) | 2746 | 2747 | 2745
Percentage of Participants | 7.5 | 7.3 | 6.8

107. Secondary Outcome: Percentage of Participants Discontinuing Study Treatment Due to An AE (Insulin With or Without Metformin Add-on Glycemic Sub-study)
Description: as for outcome 102
Time Frame: Up to 18 weeks
Population: as for outcome 103
Measure: Number; unit: Percentage of Participants
Arm/Group | Ertugliflozin 5 mg (Insulin +/- Metformin Glycemic Sub-study) | Ertugliflozin 15 mg (Insulin +/- Metformin Glycemic Sub-study) | Placebo (Insulin +/- Metformin Glycemic Sub-study)
Number analyzed (Participants) | 348 | 370 | 347
Percentage of Participants | 2.9 | 3.8 | 3.7
Statistical Analysis 1: Comparison: Ertugliflozin 15 mg (Insulin +/- Metformin Glycemic Sub-study) vs Placebo (Insulin +/- Metformin Glycemic Sub-study); Test type: Superiority; Difference in % vs Placebo = 0.0, 95% CI 2-sided [-2.9 to 3.0]; Miettinen & Nurminen method
Statistical Analysis 2: Comparison: Ertugliflozin 5 mg (Insulin +/- Metformin Glycemic Sub-study) vs Placebo (Insulin +/- Metformin Glycemic Sub-study); Test type: Superiority; Difference in % vs Placebo = -1.2, 95% CI 2-sided [-4.0 to 1.6]; Miettinen & Nurminen method

108. Secondary Outcome: Percentage of Participants Discontinuing Study Treatment Due to An AE (Sulfonylurea Monotherapy Add-on Glycemic Sub-Study)
Description: as for outcome 102
Time Frame: Up to 18 weeks
Population: as for outcome 104
Measure: Number; unit: Percentage of Participants
Arm/Group | Ertugliflozin 5 mg (Sulfonylurea Monotherapy Glycemic Sub-study) | Ertugliflozin 15 mg (Sulfonylurea Monotherapy Glycemic Sub-study) | Placebo (Sulfonylurea Monotherapy Glycemic Sub-study)
Number analyzed (Participants) | 55 | 54 | 48
Percentage of Participants | 3.6 | 1.9 | 2.1

109. Secondary Outcome: Percentage of Participants Discontinuing Study Treatment Due to An AE (Metformin With Sulfonylurea Add-on Glycemic Sub-study)
Description: as for outcome 102
Time Frame: Up to 18 weeks
Population: as for outcome 105
Measure: Number; unit: Percentage of Participants
Arm/Group | Ertugliflozin 5 mg (Metformin With Sulfonylurea Glycemic Sub-study) | Ertugliflozin 15 mg (Metformin With Sulfonylurea Glycemic Sub-study) | Placebo (Metformin With Sulfonylurea Glycemic Sub-study)
Number analyzed (Participants) | 100 | 113 | 117
Percentage of Participants | 0 | 2.7 | 1.7

110. Secondary Outcome: Change From Baseline in Fasting Plasma Glucose (FPG) at Week 18 (Excluding Rescue Approach) (Insulin With or Without Metformin Add-on Glycemic Sub-study)
Description: FPG was analyzed after an overnight fast. This change from baseline reflects the Week 18 FPG minus the Week 0 FPG. A negative number indicates a reduction in the FPG. Participants who met glycemic rescue criteria received glycemic rescue medication. "Excluding Rescue" excluded all data following the initiation of rescue in order to avoid the confounding influence of the rescue therapy.
Time Frame: Baseline and Week 18
Population: The analysis population included all participants who were randomized, participated in the Insulin +/- Metformin Glycemic Sub-study, received at least one dose of blinded study medication, and had at least one measurement for the analysis endpoint for the specified timepoint(s) at or after Baseline.
Measure: Least Squares Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Ertugliflozin 5 mg (Insulin +/- Metformin Glycemic Sub-study) | Ertugliflozin 15 mg (Insulin +/- Metformin Glycemic Sub-study) | Placebo (Insulin +/- Metformin Glycemic Sub-study)
Number analyzed (Participants) | 348 | 370 | 347
mg/dL | -26.98 [-32.80 to -21.17] | -33.15 [-38.81 to -27.48] | -7.74 [-13.67 to -1.81]
Statistical Analysis 1: Comparison: Ertugliflozin 15 mg (Insulin +/- Metformin Glycemic Sub-study) vs Placebo (Insulin +/- Metformin Glycemic Sub-study); Test type: Superiority; p < 0.001, CLDA; Model with fixed effects for treatment, time, baseline eGFR, stratum (insulin alone or insulin + metformin) and the interaction of time by treatment; Difference in the Least Squares Means = -25.40, 95% CI 2-sided [-32.84 to -17.96]
Statistical Analysis 2: Comparison: Ertugliflozin 5 mg (Insulin +/- Metformin Glycemic Sub-study) vs Placebo (Insulin +/- Metformin Glycemic Sub-study); Test type: Superiority; p < 0.001, cLDA; [statistical method as in outcome 110, analysis 1]; Difference in the Least Squares Means = -19.24, 95% CI 2-sided [-26.80 to -11.68]

111. Secondary Outcome: Change From Baseline in Body Weight at Week 18 (Excluding Rescue Approach) (Insulin With or Without Metformin Add-on Glycemic Sub-study)
Description: This change from baseline reflects the Week 18 body weight minus the Week 0 body weight. Participants who met glycemic rescue criteria received glycemic rescue medication. "Excluding Rescue" excluded all data following the initiation of rescue in order to avoid the confounding influence of the rescue therapy.
Time Frame: Baseline and Week 18
Population: The analysis population included all participants who were randomized, participated in the Insulin +/- Metformin Glycemic Sub-study, received at least one dose of study medication and had at least one measurement of the analysis endpoint for the specified timepoint(s) at any time from baseline to Week 18.
Measure: Least Squares Mean (95% Confidence Interval); unit: Kilograms
Arm/Group | Ertugliflozin 5 mg (Insulin +/- Metformin Glycemic Sub-study) | Ertugliflozin 15 mg (Insulin +/- Metformin Glycemic Sub-study) | Placebo (Insulin +/- Metformin Glycemic Sub-study)
Number analyzed (Participants) | 348 | 370 | 347
Kilograms | -1.87 [-2.22 to -1.52] | -2.13 [-2.47 to -1.79] | -0.25 [-0.60 to 0.11]
Statistical Analysis 1: Comparison: Ertugliflozin 15 mg (Insulin +/- Metformin Glycemic Sub-study) vs Placebo (Insulin +/- Metformin Glycemic Sub-study); Test type: Superiority; p < 0.001, cLDA; [statistical method as in outcome 110, analysis 1]; Difference in the Least Squares Means = -1.88, 95% CI 2-sided [-2.37 to -1.13]
Statistical Analysis 2: Comparison: Ertugliflozin 5 mg (Insulin +/- Metformin Glycemic Sub-study); Test type: Superiority; p < 0.001, cLDA model; [statistical method as in outcome 110, analysis 1]; Difference in the Least Squares Means = -1.62, 95% CI 2-sided [-2.12 to -1.13]

112. Secondary Outcome: Percentage of Participants With an A1C <7% (<53 mmol/Mol) at Week 18 (Excluding Rescue Approach) (Insulin With or Without Metformin Add-on Glycemic Sub-study)
Description: A1C is a blood marker used to report average blood glucose levels over prolonged periods of time and is reported as a percentage (%). A1C represents the percentage of glycated hemoglobin. Participants who met glycemic rescue criteria received glycemic rescue medication. "Excluding Rescue" excluded all data following the initiation of rescue in order to avoid the confounding influence of the rescue therapy.
Time Frame: Week 18
Population: as for outcome 111
Measure: Number; unit: Percentage of Participants
Arm/Group | Ertugliflozin 5 mg (Insulin +/- Metformin Glycemic Sub-study) | Ertugliflozin 15 mg (Insulin +/- Metformin Glycemic Sub-study) | Placebo (Insulin +/- Metformin Glycemic Sub-study)
Number analyzed (Participants) | 348 | 370 | 347
Percentage of Participants | 20.7 | 21.1 | 10.7
Statistical Analysis 1: Comparison: Ertugliflozin 15 mg (Insulin +/- Metformin Glycemic Sub-study) vs Placebo (Insulin +/- Metformin Glycemic Sub-study); Missing data imputed using the Constrained Longitudinal Data Analysis (cLDA) model fitted with fixed effects as in the primary analysis; Test type: Superiority; p < 0.001, Regression, Logistic; Model fitted with fixed effects for treatment, stratum for insulin sub-study, covariates for baseline A1C and baseline eGFR (continuous); Adjusted Odds Ratio Relative to Placebo = 2.49, 95% CI 2-sided [1.61 to 3.83]
Statistical Analysis 2: Comparison: Ertugliflozin 5 mg (Insulin +/- Metformin Glycemic Sub-study) vs Placebo (Insulin +/- Metformin Glycemic Sub-study); [analysis description as in outcome 112, analysis 1]; Test type: Superiority; p < 0.001, Regression, Logistic; [statistical method as in outcome 112, analysis 1]; Adjusted Odds Ratio Relative to Placebo = 2.60, 95% CI 2-sided [1.64 to 4.12]

113. Secondary Outcome: Change From Baseline in Sitting Systolic Blood Pressure (SBP) at Week 18 (Excluding Rescue Approach) (Insulin With or Without Metformin Add-on Glycemic Sub-study)
Description: This change from baseline reflects the Week 18 SBP minus the Week 0 SBP. A negative number indicates a reduction in SBP. Participants who met glycemic rescue criteria received glycemic rescue medication. "Excluding Rescue" excluded all data following the initiation of rescue in order to avoid the confounding influence of the rescue therapy.
Time Frame: Baseline and Week 18
Population: The analysis population included all participants who were randomized, participated in the Insulin +/- Metformin Glycemic Sub-study, received at least one dose of study medication, and had at least one measurement for the analysis endpoint for the specified timepoint(s) at or after Baseline.
Measure: Least Squares Mean (95% Confidence Interval); unit: mmHg
Arm/Group | Ertugliflozin 5 mg (Insulin +/- Metformin Glycemic Sub-study) | Ertugliflozin 15 mg (Insulin +/- Metformin Glycemic Sub-study) | Placebo (Insulin +/- Metformin Glycemic Sub-study)
Number analyzed (Participants) | 348 | 370 | 347
mmHg | -2.67 [-4.17 to -1.18] | -2.12 [-3.57 to -0.67] | 0.20 [-1.33 to 1.74]
Statistical Analysis 1: Comparison: Ertugliflozin 15 mg (Insulin +/- Metformin Glycemic Sub-study) vs Placebo (Insulin +/- Metformin Glycemic Sub-study); Test type: Superiority; p = 0.025, cLDA; Model with fixed effects for treatment, time, baseline eGFR, stratum (insulin alone or insulin + metformin), and the interaction of time by treatment; Difference in the Least Squares Means = -2.32, 95% CI 2-sided [-4.35 to -0.30]
Statistical Analysis 2: Comparison: Ertugliflozin 5 mg (Insulin +/- Metformin Glycemic Sub-study) vs Placebo (Insulin +/- Metformin Glycemic Sub-study); Test type: Superiority; p = 0.006, cLDA; [statistical method as in outcome 113, analysis 1]; Difference in the Least Squares Means = -2.88, 95% CI 2-sided [-4.94 to -0.82]

114. Secondary Outcome: Change From Baseline in Sitting Diastolic Blood Pressure (DBP) at Week 18 (Excluding Rescue Approach) (Insulin With or Without Metformin Add-on Glycemic Sub-study)
Description: This change from baseline reflects the Week 18 DBP minus the Week 0 BBP. A negative number indicates a reduction in DBP. Participants who met glycemic rescue criteria received glycemic rescue medication. "Excluding Rescue" excluded all data following the initiation of rescue in order to avoid the confounding influence of the rescue therapy.
Time Frame: Baseline and Week 18
Population: as for outcome 113
Measure: Least Squares Mean (95% Confidence Interval); unit: mmHg
Arm/Group | Ertugliflozin 5 mg (Insulin +/- Metformin Glycemic Sub-study) | Ertugliflozin 15 mg (Insulin +/- Metformin Glycemic Sub-study) | Placebo (Insulin +/- Metformin Glycemic Sub-study)
Number analyzed (Participants) | 348 | 370 | 347
mmHg | -0.86 [-1.72 to -0.00] | -0.64 [-1.47 to 0.20] | -0.26 [-1.14 to 0.62]
Statistical Analysis 1: Comparison: Ertugliflozin 15 mg (Insulin +/- Metformin Glycemic Sub-study) vs Placebo (Insulin +/- Metformin Glycemic Sub-study); Test type: Superiority; p = 0.533, cLDA model; [statistical method as in outcome 113, analysis 1]; Difference in the Least Squares Means = -0.38, 95% CI 2-sided [-1.56 to 0.81]
Statistical Analysis 2: Comparison: Ertugliflozin 5 mg (Insulin +/- Metformin Glycemic Sub-study) vs Placebo (Insulin +/- Metformin Glycemic Sub-study); Test type: Superiority; p = 0.326, cLDA model; [statistical method as in outcome 113, analysis 1]; Difference in the Least Squares Means = -0.60, 95% CI 2-sided [-1.81 to 0.60]

115. Secondary Outcome: Baseline Insulin Dose for Participants Receiving Insulin at Baseline - (Insulin With or Without Metformin Add-on Glycemic Sub-study)
Description: Baseline reflects Week 0 insulin dose.
Time Frame: Baseline
Population: The analysis population included all participants who were randomized, participated in the Insulin +/- Metformin Glycemic Sub-study, and received insulin at baseline.
Measure: Mean (Standard Deviation); unit: Unit/day
Arm/Group | Ertugliflozin 5 mg (Insulin +/- Metformin Glycemic Sub-study) | Ertugliflozin 15 mg (Insulin +/- Metformin Glycemic Sub-study) | Placebo (Insulin +/- Metformin Glycemic Sub-study)
Number analyzed (Participants) | 348 | 370 | 347
Unit/day | 70.76 (44.15) | 67.29 (41.23) | 73.20 (49.58)

116. Secondary Outcome: Change From Baseline at Week 18 in Insulin Dose for Participants Receiving Insulin at Baseline - Including Rescue Approach (Insulin With or Without Metformin Add-on Glycemic Sub-study)
Description: This change from baseline reflects the Week 18 insulin dose minus the Week 0 insulin dose. A negative number indicates a decrease in insulin dose. Participants who met glycemic rescue criteria received glycemic rescue medication. "Including rescue", included data following the initiation of rescue therapy.
Time Frame: Baseline and Week 18
Population: The analysis population included all participants who were randomized, participated in the Insulin +/- Metformin Glycemic Sub-study, received at least one dose of study medication and had measurements of the analysis endpoint for the specified timepoint(s) both at Baseline and Week 18, and received insulin at baseline.
Measure: Mean (Standard Deviation); unit: Unit/day
Arm/Group | Ertugliflozin 5 mg (Insulin +/- Metformin Glycemic Sub-study) | Ertugliflozin 15 mg (Insulin +/- Metformin Glycemic Sub-study) | Placebo (Insulin +/- Metformin Glycemic Sub-study)
Number analyzed (Participants) | 347 | 366 | 346
Unit/day | -0.71 (10.14) | -2.14 (10.23) | -0.29 (11.49)

117. Secondary Outcome: Change From Baseline in Fasting Plasma Glucose (FPG) at Week 18 (Excluding Rescue Approach) (Sulfonylurea Monotherapy Add-on Glycemic Sub-Study)
Description: FPG was analyzed after an overnight fast. This change from baseline reflects the Week 18 FPG minus the Week 0 FPG. A negative number indicates a reduction in FPG. Participants who met glycemic rescue criteria received glycemic rescue medication. "Excluding Rescue" excluded all data following the initiation of rescue in order to avoid the confounding influence of the rescue therapy.
Time Frame: Baseline and Week 18
Population: The analysis population included all participants who were randomized, participated in the Sulfonylurea Monotherapy Glycemic Sub-study, received at least one dose of study medication and had at least one measurement of the analysis endpoint for the specified timepoint(s) at any time from baseline to Week 18.
Measure: Least Squares Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Ertugliflozin 5 mg (Sulfonylurea Monotherapy Glycemic Sub-study) | Ertugliflozin 15 mg (Sulfonylurea Monotherapy Glycemic Sub-study) | Placebo (Sulfonylurea Monotherapy Glycemic Sub-study)
Number analyzed (Participants) | 55 | 54 | 48
mg/dL | -28.28 [-39.44 to -17.12] | -26.97 [-38.51 to -15.44] | -14.76 [-26.43 to -3.08]
Statistical Analysis 1: Comparison: Ertugliflozin 15 mg (Sulfonylurea Monotherapy Glycemic Sub-study) vs Placebo (Sulfonylurea Monotherapy Glycemic Sub-study); Test type: Superiority; p = 0.105, cLDA; cLDA model with fixed effects for treatment, time, baseline eGFR (continuous), and the interaction of time by treatment; Difference in the Least Squares Means = -12.22, 95% CI 2-sided [-27.03 to 2.06]
Statistical Analysis 2: Comparison: Ertugliflozin 5 mg (Sulfonylurea Monotherapy Glycemic Sub-study) vs Placebo (Sulfonylurea Monotherapy Glycemic Sub-study); Test type: Superiority; p = 0.068, cLDA; cLDA model with fixed effects for treatment, time, baseline eGFR (continuous), and the interaction of time by treatment; Difference in the Least Squares Means = -13.53, 95% CI 2-sided [-28.06 to 1.00]

118. Secondary Outcome: Change From Baseline in Body Weight at Week 18 (Excluding Rescue Approach) (Sulfonylurea Monotherapy Add-on Glycemic Sub-Study)
Description: as for outcome 67
Time Frame: Baseline and Week 18
Population: as for outcome 117
Measure: Least Squares Mean (95% Confidence Interval); unit: Kilograms
Arm/Group | Ertugliflozin 5 mg (Sulfonylurea Monotherapy Glycemic Sub-study) | Ertugliflozin 15 mg (Sulfonylurea Monotherapy Glycemic Sub-study) | Placebo (Sulfonylurea Monotherapy Glycemic Sub-study)
Number analyzed (Participants) | 55 | 54 | 48
Kilograms | -1.75 [-2.61 to -0.89] | -1.20 [-2.09 to -0.31] | -0.68 [-1.60 to 0.25]
Statistical Analysis 1: Comparison: Ertugliflozin 15 mg (Sulfonylurea Monotherapy Glycemic Sub-study); Test type: Superiority; p = 0.418, cLDA; Model with fixed effects for treatment, time, baseline eGFR (continuous) and the interaction of time by treatment; Difference in the Least Squares Means = -0.52, 95% CI 2-sided [-1.79 to 0.75]
Statistical Analysis 2: Comparison: Ertugliflozin 5 mg (Sulfonylurea Monotherapy Glycemic Sub-study) vs Placebo (Sulfonylurea Monotherapy Glycemic Sub-study); Test type: Superiority; p = 0.092, cLDA model; Model with fixed effects for treatment, time, baseline eGFR (continuous) and the interaction of time by treatment; Difference in the Least Squares Means = -1.07, 95% CI 2-sided [-2.32 to 0.18]

119. Secondary Outcome: Percentage of Participants With an A1C <7% (<53 mmol/Mol) at Week 18 (Excluding Rescue Approach) (Sulfonylurea Monotherapy Add-on Glycemic Sub-Study)
Description: as for outcome 112
Time Frame: Week 18
Population: as for outcome 117
Measure: Number; unit: Percentage of Participants
Arm/Group | Ertugliflozin 5 mg (Sulfonylurea Monotherapy Glycemic Sub-study) | Ertugliflozin 15 mg (Sulfonylurea Monotherapy Glycemic Sub-study) | Placebo (Sulfonylurea Monotherapy Glycemic Sub-study)
Number analyzed (Participants) | 55 | 54 | 48
Percentage of Participants | 32.7 | 27.8 | 25.0
Statistical Analysis 1: Comparison: Ertugliflozin 15 mg (Sulfonylurea Monotherapy Glycemic Sub-study) vs Placebo (Sulfonylurea Monotherapy Glycemic Sub-study); [analysis description as in outcome 112, analysis 1]; Test type: Superiority; p = 0.460, Regression, Logistic; Model fitted with fixed effects for treatment, covariates for baseline A1C and baseline eGFR (continuous); Odds ratio relative to placebo = 1.48, 95% CI 2-sided [0.52 to 4.17]
Statistical Analysis 2: Comparison: Ertugliflozin 5 mg (Sulfonylurea Monotherapy Glycemic Sub-study) vs Placebo (Sulfonylurea Monotherapy Glycemic Sub-study); [analysis description as in outcome 112, analysis 1]; Test type: Superiority; p = 0.335, Regression, Logistic; Model fitted with fixed effects for treatment, covariates for baseline A1C and baseline eGFR (continuous); Odds ratio relative to placebo = 1.62, 95% CI 2-sided [0.61 to 4.35]

120. Secondary Outcome: Change From Baseline in Sitting Systolic Blood Pressure (SBP) at Week 18 (Excluding Rescue Approach) (Sulfonylurea Monotherapy Add-on Glycemic Sub-Study)
Description: as for outcome 113
Time Frame: Baseline and Week 18
Population: as for outcome 117
Measure: Least Squares Mean (95% Confidence Interval); unit: mmHg
Arm/Group | Ertugliflozin 5 mg (Sulfonylurea Monotherapy Glycemic Sub-study) | Ertugliflozin 15 mg (Sulfonylurea Monotherapy Glycemic Sub-study) | Placebo (Sulfonylurea Monotherapy Glycemic Sub-study)
Number analyzed (Participants) | 55 | 54 | 48
mmHg | -0.72 [-4.06 to 2.63] | -0.80 [-4.23 to 2.63] | -3.53 [-7.03 to -0.02]
Statistical Analysis 1: Comparison: Ertugliflozin 15 mg (Sulfonylurea Monotherapy Glycemic Sub-study) vs Placebo (Sulfonylurea Monotherapy Glycemic Sub-study); Test type: Superiority; p = 0.255, cLDA; The model had fixed effects for treatment, time, baseline eGFR (continuous) and the interaction of time by treatment; Difference in the Least Squares Means = 2.73, 95% CI 2-sided [-2.00 to 7.45]
Statistical Analysis 2: Comparison: Ertugliflozin 5 mg (Sulfonylurea Monotherapy Glycemic Sub-study) vs Placebo (Sulfonylurea Monotherapy Glycemic Sub-study); Test type: Superiority; p = 0.235, cLDA; The model had fixed effects for treatment, time, baseline eGFR (continuous) and the interaction of time by treatment; Difference in the Least Squares Means = 2.81, 95% CI 2-sided [-1.85 to 7.48]

121. Secondary Outcome: Change From Baseline in Sitting Diastolic Blood (DBP) Pressure at Week 18 (Excluding Rescue Approach) (Sulfonylurea Monotherapy Add-on Glycemic Sub-Study)
Description: This change from baseline reflects the Week 18 DBP minus the Week 0 DBP. A negative number indicates a reduction in DBP. Participants who met glycemic rescue criteria received glycemic rescue medication. "Excluding Rescue" excluded all data following the initiation of rescue in order to avoid the confounding influence of the rescue therapy.
Time Frame: Baseline and Week 18
Population: as for outcome 117
Measure: Least Squares Mean (95% Confidence Interval); unit: mmHg
Arm/Group | Ertugliflozin 5 mg (Sulfonylurea Monotherapy Glycemic Sub-study) | Ertugliflozin 15 mg (Sulfonylurea Monotherapy Glycemic Sub-study) | Placebo (Sulfonylurea Monotherapy Glycemic Sub-study)
Number analyzed (Participants) | 55 | 54 | 48
mmHg | -1.18 [-3.24 to 0.88] | -0.93 [-3.05 to 1.18] | -2.91 [-5.06 to -0.76]
Statistical Analysis 1: Comparison: Ertugliflozin 15 mg (Sulfonylurea Monotherapy Glycemic Sub-study) vs Placebo (Sulfonylurea Monotherapy Glycemic Sub-study); Test type: Superiority; p = 0.178, cLDA model; [statistical method as in outcome 113, analysis 1]; Difference in the Least Squares Means = 1.98, 95% CI 2-sided [-0.91 to 4.86]
Statistical Analysis 2: Comparison: Ertugliflozin 5 mg (Sulfonylurea Monotherapy Glycemic Sub-study) vs Placebo (Sulfonylurea Monotherapy Glycemic Sub-study); Test type: Superiority; p = 0.230, cLDA; [statistical method as in outcome 113, analysis 1]; Difference in the Least Squares Means = 1.73, 95% CI 2-sided [-1.11 to 4.58]

122. Secondary Outcome: Change From Baseline in Fasting Plasma Glucose (FPG) at Week 18 (Excluding Rescue Approach) (Metformin With Sulfonylurea Add-on Glycemic Sub-study)
Description: as for outcome 117
Time Frame: Baseline and Week 18
Population: The analysis population included all participants who were randomized, participated in the Metformin with Sulfonylurea Glycemic Sub-study, received at least one dose of study medication and had at least one measurement of the analysis endpoint for the specified timepoint(s) at any time from Baseline to Week 18.
Measure: Least Squares Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Ertugliflozin 5 mg (Metformin With Sulfonylurea Glycemic Sub-study) | Ertugliflozin 15 mg (Metformin With Sulfonylurea Glycemic Sub-study) | Placebo (Metformin With Sulfonylurea Glycemic Sub-study)
Number analyzed (Participants) | 100 | 113 | 117
mg/dL | -35.28 [-43.05 to -27.50] | -36.18 [-43.36 to -28.99] | -4.81 [-12.10 to 2.49]
Statistical Analysis 1: Comparison: Ertugliflozin 15 mg (Metformin With Sulfonylurea Glycemic Sub-study); Test type: Superiority; p < 0.001, CLDA; cLDA model with fixed effects for treatment, time, baseline eGFR (continuous), and the interaction of time by treatment; Difference in the Least Squares Means = -31.37, 95% CI 2-sided [-40.68 to -22.07]
Statistical Analysis 2: Comparison: Ertugliflozin 5 mg (Metformin With Sulfonylurea Glycemic Sub-study) vs Placebo (Metformin With Sulfonylurea Glycemic Sub-study); Test type: Superiority; p < 0.001, cLDA; cLDA model with fixed effects for treatment, time, baseline eGFR (continuous), and the interaction of time by treatment; Difference in the Least Squares Means = -30.47, 95% CI 2-sided [-40.23 to -20.72]

123. Secondary Outcome: Change From Baseline in Body Weight at Week 18 (Excluding Rescue Approach) (Metformin With Sulfonylurea Add-on Glycemic Sub-study)
Description: as for outcome 67
Time Frame: Baseline and Week 18
Population: as for outcome 122
Measure: Least Squares Mean (95% Confidence Interval); unit: Kilograms
Arm/Group | Ertugliflozin 5 mg (Metformin With Sulfonylurea Glycemic Sub-study) | Ertugliflozin 15 mg (Metformin With Sulfonylurea Glycemic Sub-study) | Placebo (Metformin With Sulfonylurea Glycemic Sub-study)
Number analyzed (Participants) | 100 | 113 | 117
Kilograms | -2.04 [-2.58 to -1.50] | -2.41 [-2.91 to -1.91] | -0.47 [-0.97 to 0.03]
Statistical Analysis 1: Comparison: Ertugliflozin 15 mg (Metformin With Sulfonylurea Glycemic Sub-study) vs Placebo (Metformin With Sulfonylurea Glycemic Sub-study); Test type: Superiority; p < 0.001, cLDA; Model with fixed effects for treatment, time, baseline eGFR (continuous), and the interaction of time by treatment; Difference in the Least Squares Means = -1.94, 95% CI 2-sided [-2.65 to -1.24]
Statistical Analysis 2: Comparison: Ertugliflozin 5 mg (Metformin With Sulfonylurea Glycemic Sub-study) vs Placebo (Metformin With Sulfonylurea Glycemic Sub-study); Test type: Superiority; p < 0.001, cLDA; Model with fixed effects for treatment, time, baseline eGFR (continuous), and the interaction of time by treatment; Difference in the Least Squares Means = -1.57, 95% CI 2-sided [-2.30 to -0.84]

124. Secondary Outcome: Percentage of Participants With an A1C <7% (<53 mmol/Mol) at Week 18 (Excluding Rescue Approach) (Metformin With Sulfonylurea Add-on Glycemic Sub-study)
Description: as for outcome 112
Time Frame: Week 18
Population: as for outcome 122
Measure: Number; unit: Percentage of Participants
Arm/Group | Ertugliflozin 5 mg (Metformin With Sulfonylurea Glycemic Sub-study) | Ertugliflozin 15 mg (Metformin With Sulfonylurea Glycemic Sub-study) | Placebo (Metformin With Sulfonylurea Glycemic Sub-study)
Number analyzed (Participants) | 100 | 113 | 117
Percentage of Participants | 37.0 | 32.7 | 12.8
Statistical Analysis 1: Comparison: Ertugliflozin 15 mg (Metformin With Sulfonylurea Glycemic Sub-study) vs Placebo (Metformin With Sulfonylurea Glycemic Sub-study); Missing data imputed using the cLDA model fitted with fixed effects as in the primary analysis; Test type: Superiority; p < 0.001, Regression, Logistic; Model fitted with fixed effects for treatment, covariates for baseline A1C and baseline eGFR (continuous); Adjusted odds ratio relative to placebo = 4.10, 95% CI 2-sided [2.00 to 8.42]
Statistical Analysis 2: Comparison: Ertugliflozin 5 mg (Metformin With Sulfonylurea Glycemic Sub-study) vs Placebo (Metformin With Sulfonylurea Glycemic Sub-study); Missing data imputed using the cLDA model fitted with fixed effects as in the primary analysis; Test type: Superiority; p < 0.001, Regression, Logistic; Model fitted with fixed effects for treatment, covariates for baseline A1C and baseline eGFR (continuous); Adjusted odds ratio relative to placebo = 5.97, 95% CI 2-sided [2.86 to 12.49]

125. Secondary Outcome: Change From Baseline in Sitting Systolic Blood Pressure (SBP) at Week 18 (Excluding Rescue Approach) (Metformin With Sulfonylurea Add-on Glycemic Sub-study)
Description: as for outcome 113
Time Frame: Baseline and Week 18
Population: as for outcome 122
Measure: Least Squares Mean (95% Confidence Interval); unit: mmHg
Arm/Group | Ertugliflozin 5 mg (Metformin With Sulfonylurea Glycemic Sub-study) | Ertugliflozin 15 mg (Metformin With Sulfonylurea Glycemic Sub-study) | Placebo (Metformin With Sulfonylurea Glycemic Sub-study)
Number analyzed (Participants) | 100 | 113 | 117
mmHg | -2.26 [-4.78 to 0.25] | -1.54 [-3.85 to 0.77] | -0.70 [-3.04 to 1.64]
Statistical Analysis 1: Comparison: Ertugliflozin 15 mg (Metformin With Sulfonylurea Glycemic Sub-study) vs Placebo (Metformin With Sulfonylurea Glycemic Sub-study); Test type: Superiority; p = 0.597, cLDA; The model had fixed effects for treatment, time, baseline eGFR (continuous) and the interaction of time by treatment; Difference in the Least Squares Means = -0.85, 95% CI 2-sided [-4.00 to 2.30]
Statistical Analysis 2: Comparison: Ertugliflozin 5 mg (Metformin With Sulfonylurea Glycemic Sub-study) vs Placebo (Metformin With Sulfonylurea Glycemic Sub-study); Test type: Superiority; p = 0.351, cLDA; The model had fixed effects for treatment, time, baseline eGFR (continuous) and the interaction of time by treatment; Difference in the Least Squares Means = -1.57, 95% CI 2-sided [-4.87 to 1.73]

126. Secondary Outcome: Change From Baseline in Sitting Diastolic Blood (DBP) Pressure at Week 18 (Excluding Rescue Approach) (Metformin With Sulfonylurea Add-on Glycemic Sub-study)
Description: as for outcome 121
Time Frame: Baseline and Week 18
Population: as for outcome 122
Measure: Least Squares Mean (95% Confidence Interval); unit: mmHg
Arm/Group | Ertugliflozin 5 mg (Metformin With Sulfonylurea Glycemic Sub-study) | Ertugliflozin 15 mg (Metformin With Sulfonylurea Glycemic Sub-study) | Placebo (Metformin With Sulfonylurea Glycemic Sub-study)
Number analyzed (Participants) | 100 | 113 | 117
mmHg | -0.30 [-1.80 to 1.21] | -0.92 [-2.30 to 0.46] | -0.24 [-1.64 to 1.15]
Statistical Analysis 1: Comparison: Ertugliflozin 15 mg (Metformin With Sulfonylurea Glycemic Sub-study) vs Placebo (Metformin With Sulfonylurea Glycemic Sub-study); Test type: Superiority; p = 0.490, cLDA; Model with fixed effects for treatment, time, baseline eGFR (continuous) and the interaction of time by treatment; Difference in the Least Squares Means = -0.68, 95% CI 2-sided [-2.60 to 1.25]
Statistical Analysis 2: Comparison: Ertugliflozin 5 mg (Metformin With Sulfonylurea Glycemic Sub-study) vs Placebo (Metformin With Sulfonylurea Glycemic Sub-study); Test type: Superiority; p = 0.958, cLDA; Model with fixed effects for treatment, time, baseline eGFR (continuous) and the interaction of time by treatment; Difference in the Least Squares Means = -0.05, 95% CI 2-sided [-2.07 to 1.96]

ADVERSE EVENTS:
Time Frame: Overall Cardiovascular study - Up to approximately 6 years 3 Glycemic Sub-studies - Up to 18 weeks
Description: The analysis population for all-cause mortality was all randomized participants and the analysis population for adverse events was all participants who received at least one dose of blinded study medication. The Overall Cardiovascular Study had a follow-up of approximately 6 years whereas the glycemic sub-studies had an 18-week follow-up time.
Groups:
- Ertugliflozin 5 mg (Insulin +/- Metformin Sub-study); Ertugliflozin 5 mg (Sulfonylurea Monotherapy Glycemic Sub-Study); Ertugliflozin 5 mg (Metformin With Sulfonylurea Glycemic Sub-study): Ertugliflozin 5 mg, administered orally, once daily, for up to 18 weeks
Arm/Group | Ertugliflozin 5 mg (Overall Cardiovascular Study) | Ertugliflozin 15 mg (Overall Cardiovascular Study) | Placebo (Overall Cardiovascular Study) | Ertugliflozin 5 mg (Insulin +/- Metformin Sub-study) | Ertugliflozin 15 mg (Insulin +/- Metformin Glycemic Sub-study) | Placebo (Insulin +/- Metformin Glycemic Sub-study) | Ertugliflozin 5 mg (Sulfonylurea Monotherapy Glycemic Sub-Study) | Ertugliflozin 15 mg (Sulfonylurea Monotherapy Glycemic Sub-Study) | Placebo (Sulfonylurea Monotherapy Glycemic Sub-Study) | Ertugliflozin 5 mg (Metformin With Sulfonylurea Glycemic Sub-study) | Ertugliflozin 15 mg (Metformin With Sulfonylurea Glycemic Sub-study) | Placebo (Metformin With Sulfonylurea Glycemic Sub-study)
All-Cause Mortality (participants affected / at risk) | 228/2746 | 233/2747 | 247/2745 | 4/348 | 6/370 | 1/347 | 0/55 | 1/54 | 0/48 | 0/100 | 1/113 | 0/117
Serious Adverse Events (participants affected / at risk) | 958/2746 | 937/2747 | 990/2745 | 33/348 | 27/370 | 37/347 | 4/55 | 1/54 | 2/48 | 7/100 | 8/113 | 6/117
Other Adverse Events (participants affected / at risk) | 1405/2746 | 1389/2747 | 1395/2745 | 127/348 | 144/370 | 135/347 | 10/55 | 4/54 | 9/48 | 24/100 | 32/113 | 26/117
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Ertugliflozin 5 mg (Overall Cardiovascular Study) (N=2746) | Ertugliflozin 15 mg (Overall Cardiovascular Study) (N=2747) | Placebo (Overall Cardiovascular Study) (N=2745) | Ertugliflozin 5 mg (Insulin +/- Metformin Sub-study) (N=348) | Ertugliflozin 15 mg (Insulin +/- Metformin Glycemic Sub-study) (N=370) | Placebo (Insulin +/- Metformin Glycemic Sub-study) (N=347) | Ertugliflozin 5 mg (Sulfonylurea Monotherapy Glycemic Sub-Study) (N=55) | Ertugliflozin 15 mg (Sulfonylurea Monotherapy Glycemic Sub-Study) (N=54) | Placebo (Sulfonylurea Monotherapy Glycemic Sub-Study) (N=48) | Ertugliflozin 5 mg (Metformin With Sulfonylurea Glycemic Sub-study) (N=100) | Ertugliflozin 15 mg (Metformin With Sulfonylurea Glycemic Sub-study) (N=113) | Placebo (Metformin With Sulfonylurea Glycemic Sub-study) (N=117)
Anaemia (Blood and lymphatic system disorders) | 5 (5) | 4 (4) | 3 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood loss anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0/0 (0) | 0/0 (0) | 0/0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemolytic anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Immune thrombocytopenic purpura (Blood and lymphatic system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 (1) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Leukocytosis (Blood and lymphatic system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lymphadenopathy (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lymphadenopathy mediastinal (Blood and lymphatic system disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Microcytic anaemia (Blood and lymphatic system disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Normocytic anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pancytopenia (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Polycythaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thrombotic thrombocytopenic purpura (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute coronary syndrome (Cardiac disorders) | 9 (9) | 6 (6) | 8 (8) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute left ventricular failure (Cardiac disorders) | 3 (3) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 52 (61) | 76 (83) | 73 (80) | 3 | 1 | 1 | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Adams-Stokes syndrome (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Angina pectoris (Cardiac disorders) | 38 (39) | 42 (48) | 49 (54) | 2 | 2 | 3 | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Angina unstable (Cardiac disorders) | 74 (92) | 71 (78) | 89 (106) | 3 | 1 | 1 | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Anginal equivalent (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aortic valve stenosis (Cardiac disorders) | 4 (4) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arrhythmia (Cardiac disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arrhythmia supraventricular (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arteriosclerosis coronary artery (Cardiac disorders) | 3 (3) | 2 (2) | 3 (3) | 0 | 0 | 1 | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 30 (33) | 31 (38) | 37 (40) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Atrial flutter (Cardiac disorders) | 11 (12) | 9 (9) | 9 (11) | 1 | 0 | 0 | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Atrial tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Atrioventricular block (Cardiac disorders) | 1 (1) | 3 (3) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Atrioventricular block complete (Cardiac disorders) | 3 (3) | 2 (2) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Atrioventricular block first degree (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Atrioventricular block second degree (Cardiac disorders) | 5 (5) | 5 (5) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bradyarrhythmia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bradycardia (Cardiac disorders) | 1 (1) | 5 (5) | 5 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bundle branch block left (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bundle branch block right (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardiac arrest (Cardiac disorders) | 7 (7) | 15 (15) | 13 (13) | 0 | 0 | 2 | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardiac asthma (Cardiac disorders) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardiac disorder (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardiac failure (Cardiac disorders) | 35 (39) | 34 (36) | 43 (58) | 0 | 0 | 1 | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardiac failure acute (Cardiac disorders) | 7 (7) | 7 (7) | 8 (11) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardiac failure chronic (Cardiac disorders) | 16 (20) | 10 (12) | 14 (17) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 19 (23) | 28 (37) | 35 (42) | 0 (0) | 0 (0) | 0 | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardiac tamponade (Cardiac disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardiac ventricular thrombosis (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardio-respiratory arrest (Cardiac disorders) | 4 (4) | 5 (5) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardiogenic shock (Cardiac disorders) | 3 (3) | 4 (4) | 8 (8) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardiomyopathy (Cardiac disorders) | 2 (2) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardiopulmonary failure (Cardiac disorders) | 1 (1) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardiovascular disorder (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardiovascular insufficiency (Cardiac disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chronic left ventricular failure (Cardiac disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Conduction disorder (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Coronary artery disease (Cardiac disorders) | 35 (43) | 34 (36) | 38 (42) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Coronary artery insufficiency (Cardiac disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Coronary artery occlusion (Cardiac disorders) | 2 (2) | 5 (6) | 5 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Coronary artery stenosis (Cardiac disorders) | 14 (14) | 20 (22) | 16 (18) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Coronary ostial stenosis (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertensive cardiomyopathy (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ischaemic cardiomyopathy (Cardiac disorders) | 1 (1) | 4 (4) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Left ventricular dysfunction (Cardiac disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Left ventricular failure (Cardiac disorders) | 2 (2) | 4 (4) | 6 (6) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Microvascular coronary artery disease (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mitral valve incompetence (Cardiac disorders) | 2 (2) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mitral valve stenosis (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myocardial infarction (Cardiac disorders) | 39 (39) | 49 (52) | 37 (41) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Myocardial ischaemia (Cardiac disorders) | 17 (17) | 13 (14) | 18 (21) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nodal arrhythmia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pericardial effusion (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pericarditis (Cardiac disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Postinfarction angina (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Silent myocardial infarction (Cardiac disorders) | 1 (1) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinoatrial block (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinus bradycardia (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinus node dysfunction (Cardiac disorders) | 4 (4) | 3 (3) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Stress cardiomyopathy (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Supraventricular tachyarrhythmia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 3 (5) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Systolic dysfunction (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Torsade de pointes (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tricuspid valve incompetence (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Trifascicular block (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ventricular arrhythmia (Cardiac disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ventricular extrasystoles (Cardiac disorders) | 2 (2) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ventricular failure (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ventricular fibrillation (Cardiac disorders) | 3 (3) | 5 (5) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ventricular tachycardia (Cardiac disorders) | 2 (2) | 13 (13) | 7 (8) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Atrial septal defect (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hydrocele (Congenital, familial and genetic disorders) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Phimosis (Congenital, familial and genetic disorders) | 6 (6) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute vestibular syndrome (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Deafness neurosensory (Ear and labyrinth disorders) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Deafness unilateral (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Meniere's disease (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Middle ear inflammation (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 4 (4) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vertigo positional (Ear and labyrinth disorders) | 2 (2) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vestibular disorder (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Adrenal haematoma (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Adrenal mass (Endocrine disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Adrenocortical insufficiency acute (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Goitre (Endocrine disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypothyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thyroid mass (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Angle closure glaucoma (Eye disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blindness unilateral (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cataract (Eye disorders) | 8 (9) | 13 (17) | 17 (22) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cataract nuclear (Eye disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diabetic retinal oedema (Eye disorders) | 2 (2) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diabetic retinopathy (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diplopia (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eyelid ptosis (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Glaucoma (Eye disorders) | 1 (1) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Keratitis (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Macular degeneration (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Macular fibrosis (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Macular hole (Eye disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Macular oedema (Eye disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Retinal artery embolism (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Retinal artery occlusion (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Retinal detachment (Eye disorders) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Retinal disorder (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Retinal haemorrhage (Eye disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Retinal tear (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Retinal vein thrombosis (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rhegmatogenous retinal detachment (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tractional retinal detachment (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Uveitis (Eye disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vitreoretinal traction syndrome (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vitreous adhesions (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vitreous haemorrhage (Eye disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal hernia (Gastrointestinal disorders) | 1 (1) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 5 (5) | 3 (3) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal wall haematoma (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anal fissure (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anal fistula (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anal incontinence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anogenital dysplasia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ascites (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Buccal polyp (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chronic gastritis (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Colitis ischaemic (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 5 (5) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diabetic gastroparesis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diverticulum (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diverticulum intestinal (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diverticulum intestinal haemorrhagic (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Duodenal perforation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Duodenal ulcer (Gastrointestinal disorders) | 2 (2) | 3 (3) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Enterocolitis (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Erosive duodenitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Erosive oesophagitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastric haemorrhage (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastric ulcer (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastric ulcer perforation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 4 (4) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastritis erosive (Gastrointestinal disorders) | 4 (4) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastritis haemorrhagic (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 6 (6) | 6 (6) | 6 (7) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 3 (3) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Haematemesis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haematochezia (Gastrointestinal disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ileus (Gastrointestinal disorders) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ileus paralytic (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Incarcerated inguinal hernia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 4 (5) | 5 (5) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intestinal ischaemia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intestinal mass (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intestinal perforation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intestinal stenosis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Irritable bowel syndrome (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Large intestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Large intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Large intestinal stenosis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Large intestinal ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Large intestine perforation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Large intestine polyp (Gastrointestinal disorders) | 2 (2) | 4 (4) | 3 (4) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Melaena (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mesenteric panniculitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Obstructive pancreatitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oedematous pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oesophageal achalasia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oesophageal ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oesophagitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pancreatic cyst (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pancreatic duct dilatation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 4 (4) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pancreatitis acute (Gastrointestinal disorders) | 6 (7) | 7 (7) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pancreatitis chronic (Gastrointestinal disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pancreatitis haemorrhagic (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peptic ulcer (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peptic ulcer haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Proctitis haemorrhagic (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rectal polyp (Gastrointestinal disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Salivary gland calculus (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 2 (2) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Small intestinal perforation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Strangulated umbilical hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Subileus (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Umbilical hernia (Gastrointestinal disorders) | 1 (1) | 7 (7) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 (2) | 6 (6) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Accidental death (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Asthenia (General disorders) | 1 (1) | 3 (3) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Catheter site haemorrhage (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Catheter site phlebitis (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chest discomfort (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chest pain (General disorders) | 17 (19) | 8 (9) | 8 (8) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Death (General disorders) | 35 (35) | 22 (22) | 25 (25) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hanging (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Inflammation (General disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Multiple organ dysfunction syndrome (General disorders) | 4 (4) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Non-cardiac chest pain (General disorders) | 26 (29) | 16 (18) | 22 (23) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Physical deconditioning (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Polyp (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 3 (4) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Stent-graft endoleak (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sudden cardiac death (General disorders) | 4 (4) | 3 (3) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sudden death (General disorders) | 2 (2) | 0 (0) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ulcer (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vascular stent occlusion (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vascular stent stenosis (General disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Autoimmune hepatitis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bile duct obstruction (Hepatobiliary disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bile duct stenosis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bile duct stone (Hepatobiliary disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Biliary colic (Hepatobiliary disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Biliary dilatation (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cholangitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cholangitis chronic (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 2 (2) | 7 (7) | 6 (6) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 11 (11) | 4 (4) | 11 (11) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cholecystitis chronic (Hepatobiliary disorders) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 5 (5) | 9 (9) | 6 (6) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cholelithiasis obstructive (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Drug-induced liver injury (Hepatobiliary disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gallbladder necrosis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gallbladder rupture (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatic cirrhosis (Hepatobiliary disorders) | 3 (3) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatic steatosis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatitis acute (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatitis cholestatic (Hepatobiliary disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Jaundice (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Liver injury (Hepatobiliary disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Portal vein thrombosis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Post cholecystectomy syndrome (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anaphylactic shock (Immune system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Drug hypersensitivity (Immune system disorders) | 1 (1) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypersensitivity (Immune system disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sarcoidosis (Immune system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal wall abscess (Infections and infestations) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abscess jaw (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abscess limb (Infections and infestations) | 3 (3) | 5 (5) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abscess neck (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abscess of salivary gland (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Actinomycosis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Amoebic colitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Amoebic dysentery (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anal abscess (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Appendicitis (Infections and infestations) | 1 (1) | 3 (3) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arteriosclerotic gangrene (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aspergilloma (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Atypical pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bacterial sepsis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Beta haemolytic streptococcal infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 5 (5) | 6 (6) | 11 (11) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bronchitis bacterial (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bronchitis viral (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bursitis infective (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Campylobacter gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Carbuncle (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 21 (23) | 31 (33) | 21 (26) | 0 (0) | 3 (3) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cholecystitis infective (Infections and infestations) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chronic tonsillitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Clostridium difficile colitis (Infections and infestations) | 2 (2) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Colonic abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cystitis (Infections and infestations) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Device related sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diabetic foot infection (Infections and infestations) | 2 (2) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diabetic gangrene (Infections and infestations) | 2 (2) | 4 (6) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diverticulitis (Infections and infestations) | 0 (0) | 2 (2) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Endocarditis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Endotoxic shock (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Epididymitis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Erysipelas (Infections and infestations) | 2 (2) | 4 (4) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Escherichia bacteraemia (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Escherichia sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Escherichia urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Extradural abscess (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gallbladder empyema (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gangrene (Infections and infestations) | 16 (18) | 16 (20) | 8 (8) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gas gangrene (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 5 (5) | 4 (4) | 5 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis bacterial (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 | 0 | 0 | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis clostridial (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis norovirus (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis rotavirus (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Graft infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Groin abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Groin infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haematoma infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Helicobacter infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatitis C (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Herpes zoster (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infected skin ulcer (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infective exacerbation of bronchiectasis (Infections and infestations) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infective thrombosis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 2 (2) | 2 (2) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Klebsiella bacteraemia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Klebsiella sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Labyrinthitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Laryngitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Liver abscess (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Localised infection (Infections and infestations) | 4 (4) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 1 (1) | 2 (2) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lyme disease (Infections and infestations) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lymph node tuberculosis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Meningitis aseptic (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Meningitis viral (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Meningoencephalitis bacterial (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Metapneumovirus infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscle abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ophthalmic herpes zoster (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Orchitis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Osteomyelitis (Infections and infestations) | 14 (15) | 10 (11) | 6 (8) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Otitis externa (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Paraspinal abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Paronychia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Perihepatic abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Periorbital cellulitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peritonitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peritonsillar abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pharyngeal abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pharyngitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pharyngitis streptococcal (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumococcal sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 51 (58) | 46 (48) | 45 (49) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia bacterial (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia influenzal (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia parainfluenzae viral (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia pseudomonal (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia staphylococcal (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Post procedural sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Postoperative abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Postoperative wound infection (Infections and infestations) | 3 (3) | 4 (4) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pseudomonas infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pulmonary tuberculosis (Infections and infestations) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyelonephritis (Infections and infestations) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyelonephritis acute (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyelonephritis chronic (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyoderma (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory syncytial virus infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory tract infection (Infections and infestations) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rhinovirus infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Scrotal abscess (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 22 (23) | 12 (12) | 7 (7) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Septic embolus (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Septic encephalopathy (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Septic shock (Infections and infestations) | 2 (2) | 8 (8) | 6 (6) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Spinal cord infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Staphylococcal bacteraemia (Infections and infestations) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Staphylococcal infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Staphylococcal sepsis (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Staphylococcal skin infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Streptococcal bacteraemia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Streptococcal sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Systemic candida (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tonsillitis (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tracheobronchitis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tropical ulcer (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tuberculosis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tuberculosis of eye (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 2 (2) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 16 (24) | 10 (10) | 14 (15) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection bacterial (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection fungal (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urosepsis (Infections and infestations) | 2 (2) | 1 (1) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vestibular neuronitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Viral infection (Infections and infestations) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Viral upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Wound infection (Infections and infestations) | 0 (0) | 2 (2) | 3 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Wound infection bacterial (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Wound sepsis (Infections and infestations) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Accident (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Accidental overdose (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anastomotic leak (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ankle fracture (Injury, poisoning and procedural complications) | 3 (3) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Arterial bypass occlusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arterial bypass stenosis (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arterial bypass thrombosis (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arteriovenous graft site stenosis (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Avulsion fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Back injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Brain contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardiac contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Comminuted fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Concussion (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Confusion postoperative (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 3 (3) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Coronary vascular graft occlusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Craniocerebral injury (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ear canal injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Epiphyseal fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eye contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Facial bones fracture (Injury, poisoning and procedural complications) | 2 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Femoral neck fracture (Injury, poisoning and procedural complications) | 3 (3) | 3 (3) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 6 (6) | 2 (2) | 5 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fibula fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Foot fracture (Injury, poisoning and procedural complications) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Forearm fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Foreign body in respiratory tract (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fracture displacement (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal stoma complication (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hand fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Head injury (Injury, poisoning and procedural complications) | 3 (3) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Heat exhaustion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 4 (4) | 3 (3) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Humerus fracture (Injury, poisoning and procedural complications) | 4 (4) | 2 (2) | 6 (6) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Incisional hernia (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injury corneal (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intentional overdose (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Jaw fracture (Injury, poisoning and procedural complications) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Joint dislocation (Injury, poisoning and procedural complications) | 2 (3) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Joint injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ligament sprain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Limb crushing injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Limb injury (Injury, poisoning and procedural complications) | 4 (4) | 3 (4) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Limb traumatic amputation (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lower limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 2 (4) | 1 (4) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Median nerve injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Meniscus injury (Injury, poisoning and procedural complications) | 2 (2) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nerve injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nerve root injury cervical (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Osteoradionecrosis (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Paranasal sinus injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Patella fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pelvic fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Periprocedural myocardial infarction (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Post procedural bile leak (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Post procedural discharge (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Post procedural haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Post procedural myocardial infarction (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Postoperative respiratory failure (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Postoperative thoracic procedure complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Postoperative wound complication (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Postpericardiotomy syndrome (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Procedural nausea (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Radius fracture (Injury, poisoning and procedural complications) | 1 (1) | 3 (3) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 2 (7) | 5 (13) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Road traffic accident (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin laceration (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skull fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skull fractured base (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 (1) | 5 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Spinal cord injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Spinal fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Stab wound (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sternal fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Subdural haematoma (Injury, poisoning and procedural complications) | 4 (4) | 4 (4) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Subdural haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tendon rupture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thermal burn (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 2 (3) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tibia fracture (Injury, poisoning and procedural complications) | 4 (4) | 6 (6) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tooth injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Toxicity to various agents (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Traumatic haematoma (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Traumatic intracranial haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Traumatic lung injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ulna fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper limb fracture (Injury, poisoning and procedural complications) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vascular access site haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vascular injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Wound (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Wound dehiscence (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Wound haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anticoagulation drug level above therapeutic (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Antipsychotic drug level increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood creatinine increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood glucose fluctuation (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood glucose increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood pressure increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Creatinine renal clearance decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Glomerular filtration rate decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatic enzyme increased (Investigations) | 3 (3) | 3 (3) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Liver function test increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oxygen saturation decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Transaminases increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Troponin T increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardiometabolic syndrome (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 2 (2) | 3 (3) | 5 (5) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diabetes mellitus (Metabolism and nutrition disorders) | 5 (6) | 1 (1) | 6 (6) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 12 (12) | 6 (7) | 14 (14) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 4 (5) | 5 (5) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diabetic metabolic decompensation (Metabolism and nutrition disorders) | 4 (6) | 4 (4) | 5 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fluid overload (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gout (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 3 (4) | 4 (5) | 8 (8) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 2 (2) | 4 (4) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperosmolar state (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 12 (17) | 9 (9) | 14 (14) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypovolaemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Insulin-requiring type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ketoacidosis (Metabolism and nutrition disorders) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ketosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lactic acidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Metabolic acidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Obesity (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 2 (4) | 2 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 (4) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 4 (4) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 4 (4) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bone cyst (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bursitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Connective tissue inflammation (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Costochondritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Foot deformity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gouty arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Groin pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (2) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intervertebral disc displacement (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 2 (2) | 3 (3) | 6 (6) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Joint contracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Loose body in joint (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Meniscal degeneration (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscle fatigue (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 10 (11) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myositis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Osteitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Osteitis deformans (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 22 (25) | 16 (18) | 21 (23) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Osteochondrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Periarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Polyarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Polymyalgia rheumatica (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 4 (4) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 6 (6) | 3 (3) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Spinal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Spondyloarthropathy (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Synovial cyst (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Systemic lupus erythematosus (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tenosynovitis stenosans (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Undifferentiated connective tissue disease (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute promyelocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Adenocarcinoma gastric (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 4 (4) | 5 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Adenocarcinoma pancreas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Adrenal adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Atypical fibroxanthoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
B-cell small lymphocytic lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 20 (21) | 25 (30) | 16 (21) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Basosquamous carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Basosquamous carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Benign lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 (5) | 4 (4) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bladder cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bladder neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bladder papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bladder transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 3 (3) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bladder transitional cell carcinoma stage II (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bone cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bone giant cell tumour malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bowen's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Brain neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Brain neoplasm benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Brain neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Breast cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Breast cancer stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bronchial carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Carcinoma in situ of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardiac myxoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cholangiocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chronic lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Clear cell endometrial carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Clear cell renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Colon adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4) | 4 (4) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Colon cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Colorectal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diffuse large B-cell lymphoma stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ductal adenocarcinoma of pancreas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Endometrial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Endometrial cancer stage III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Follicular thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gallbladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastric neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Glioblastoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Glioblastoma multiforme (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Glioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemangioma of liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hair follicle tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatic cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatic cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
High-grade B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intestinal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intraductal papillary-mucinous carcinoma of pancreas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intraductal proliferative breast lesion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Keratoacanthoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Large cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Leiomyosarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Liposarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lung adenocarcinoma stage 0 (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 3 (3) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lung carcinoma cell type unspecified stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 (5) | 3 (3) | 5 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lung squamous cell carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 4 (4) | 5 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Malignant melanoma in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Malignant neoplasm of ampulla of Vater (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Malignant neoplasm of renal pelvis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mantle cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Marginal zone lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Meningioma benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mesothelioma malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Metastases to abdominal cavity (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Metastases to peritoneum (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Metastases to spine (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Metastatic gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Metastatic lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Metastatic malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Metastatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Metastatic squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neoplasm of orbit (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neuroendocrine carcinoma of the skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neuroendocrine tumour of the lung metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Non-small cell lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oesophageal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oesophageal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oral neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 3 (3) | 4 (4) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pancreatic carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 1 (1) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pancreatic carcinoma recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Papillary renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Papillary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Paranasal sinus benign neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Paranasal sinus neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Penis carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Plasma cell myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 16 (16) | 10 (10) | 11 (11) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Prostate cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Prostate cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Prostate cancer stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Prostate cancer stage II (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rectal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 3 (3) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rectal adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rectal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Renal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Renal oncocytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Seborrhoeic keratosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 | 0 | 0 | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Small cell lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Small intestine carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 7 (8) | 8 (8) | 10 (12) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Squamous cell carcinoma of lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 (6) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Squamous cell carcinoma of the cervix (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Squamous cell carcinoma of the tongue (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Testicular cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tongue cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tongue neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tongue neoplasm malignant stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tonsil cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tumour of ampulla of Vater (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Uterine cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vulval cancer stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Altered state of consciousness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Amyotrophic lateral sclerosis (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aphasia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ataxia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Basal ganglia infarction (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Brain hypoxia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Brain injury (Nervous system disorders) | 4 (4) | 4 (4) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Brain stem haemorrhage (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Brain stem infarction (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Brain stem stroke (Nervous system disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Carotid arteriosclerosis (Nervous system disorders) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Carotid artery occlusion (Nervous system disorders) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Carotid artery stenosis (Nervous system disorders) | 11 (12) | 13 (13) | 12 (14) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Carpal tunnel syndrome (Nervous system disorders) | 2 (3) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Central nervous system lesion (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cerebellar infarction (Nervous system disorders) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cerebellar stroke (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cerebral arteriosclerosis (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cerebral circulatory failure (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cerebral haemorrhage (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cerebral infarction (Nervous system disorders) | 6 (6) | 13 (13) | 5 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 | 0
Cerebral ischaemia (Nervous system disorders) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 | 0
Cerebral small vessel ischaemic disease (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cerebral venous thrombosis (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 27 (27) | 25 (30) | 22 (23) | 2 (2) | 3 (3) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cerebrovascular disorder (Nervous system disorders) | 1 (1) | 3 (3) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cerebrovascular insufficiency (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cervical cord compression (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cervical radiculopathy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cervicobrachial syndrome (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chronic inflammatory demyelinating polyradiculoneuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cognitive disorder (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dementia Alzheimer's type (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diabetic encephalopathy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diabetic neuropathy (Nervous system disorders) | 5 (7) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 2 (2) | 2 (2) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysarthria (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyskinesia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Embolic cerebral infarction (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Embolic stroke (Nervous system disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Encephalopathy (Nervous system disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Epilepsy (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Essential tremor (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Facial paralysis (Nervous system disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemorrhagic cerebral infarction (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemorrhagic stroke (Nervous system disorders) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 2 (2) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hemiparaesthesia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hemiparesis (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatic encephalopathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hydrocephalus (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypersomnia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertensive encephalopathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoxic-ischaemic encephalopathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intraventricular haemorrhage (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ischaemic cerebral infarction (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ischaemic stroke (Nervous system disorders) | 29 (31) | 40 (40) | 41 (45) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lacunar infarction (Nervous system disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lacunar stroke (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Leukoencephalopathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Loss of consciousness (Nervous system disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lumbar radiculopathy (Nervous system disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lumbosacral radiculopathy (Nervous system disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Memory impairment (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Metabolic encephalopathy (Nervous system disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Migraine (Nervous system disorders) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mixed dementia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Motor dysfunction (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myasthenia gravis (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myelitis transverse (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myelopathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neuralgia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neuralgic amyotrophy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neuritis (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neuropathy peripheral (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Normal pressure hydrocephalus (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Paralysis (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Paraparesis (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peripheral paralysis (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Polyneuropathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Presyncope (Nervous system disorders) | 4 (4) | 2 (2) | 5 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Radiculopathy (Nervous system disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Reversible ischaemic neurological deficit (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Seizure (Nervous system disorders) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Subarachnoid haemorrhage (Nervous system disorders) | 1 (1) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 8 (10) | 10 (10) | 8 (9) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tension headache (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thalamic infarction (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thrombotic cerebral infarction (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 19 (20) | 14 (14) | 23 (25) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Trigeminal neuralgia (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
VIth nerve paralysis (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vascular dementia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vascular encephalopathy (Nervous system disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vertebral artery stenosis (Nervous system disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vertebrobasilar insufficiency (Nervous system disorders) | 2 (2) | 2 (2) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Device breakage (Product Issues) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Device malfunction (Product Issues) | 1 (1) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Device occlusion (Product Issues) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Device stimulation issue (Product Issues) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Adjustment disorder (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bipolar I disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Completed suicide (Psychiatric disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Confusional state (Psychiatric disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Delirium (Psychiatric disorders) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hallucination, visual (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Major depression (Psychiatric disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mania (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mental disorder (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mental status changes (Psychiatric disorders) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mood disorder due to a general medical condition (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Paranoia (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Stress (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Suicidal ideation (Psychiatric disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Suicide attempt (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 24 (24) | 18 (18) | 22 (24) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Azotaemia (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bladder dysplasia (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bladder neck obstruction (Renal and urinary disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bladder outlet obstruction (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bladder tamponade (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Calculus bladder (Renal and urinary disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Calculus urinary (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chronic kidney disease (Renal and urinary disorders) | 1 (1) | 6 (6) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cystitis haemorrhagic (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diabetic nephropathy (Renal and urinary disorders) | 2 (5) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
End stage renal disease (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haematuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemorrhage urinary tract (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hydronephrosis (Renal and urinary disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 4 (4) | 2 (2) | 6 (7) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nephropathy (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nephropathy toxic (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neurogenic bladder (Renal and urinary disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Proteinuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Renal artery stenosis (Renal and urinary disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Renal colic (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Renal cyst (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Renal failure (Renal and urinary disorders) | 4 (4) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Renal haemorrhage (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Renal impairment (Renal and urinary disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Renal tubular necrosis (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Stag horn calculus (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Stress urinary incontinence (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tubulointerstitial nephritis (Renal and urinary disorders) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ureteric stenosis (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ureterolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0) | 3 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urethral stenosis (Renal and urinary disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary incontinence (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary retention (Renal and urinary disorders) | 2 (2) | 4 (5) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract obstruction (Renal and urinary disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acquired hydrocele (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acquired phimosis (Reproductive system and breast disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 10 (10) | 12 (12) | 7 (7) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cystocele (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Genital haemorrhage (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Metrorrhagia (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Orchitis noninfective (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ovarian cyst (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Prostatic dysplasia (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Prostatitis (Reproductive system and breast disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Prostatomegaly (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Testicular mass (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Uterine prolapse (Reproductive system and breast disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vaginal prolapse (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 8 (8) | 7 (7) | 9 (9) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (2) | 4 (7) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Asthma-chronic obstructive pulmonary disease overlap syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bronchial hyperreactivity (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 11 (22) | 6 (10) | 14 (19) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chronic respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (3) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Emphysema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 2 (2) | 0 | 0 | 0 | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Laryngeal oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lower respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasal polyps (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasal septum deviation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Paranasal cyst (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 4 (4) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 3 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumothorax spontaneous (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 11 (11) | 4 (4) | 6 (6) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pulmonary granuloma (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pulmonary infarction (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2) | 6 (7) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 9 (9) | 6 (6) | 11 (11) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Angioedema (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (3) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diabetic foot (Skin and subcutaneous tissue disorders) | 10 (10) | 9 (9) | 13 (14) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diabetic ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ischaemic skin ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lichen sclerosus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Psoriasis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin necrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin ulcer (Skin and subcutaneous tissue disorders) | 5 (8) | 7 (7) | 4 (4) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Stasis dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Atrial appendage closure (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Accelerated hypertension (Vascular disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aortic aneurysm (Vascular disorders) | 7 (7) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aortic aneurysm rupture (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aortic stenosis (Vascular disorders) | 2 (2) | 3 (3) | 6 (6) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aortic thrombosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arteriosclerosis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arteriovenous fistula (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood pressure inadequately controlled (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Brachiocephalic artery stenosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Circulatory collapse (Vascular disorders) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 4 (4) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Embolism arterial (Vascular disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Extremity necrosis (Vascular disorders) | 2 (3) | 6 (8) | 4 (5) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Femoral artery aneurysm (Vascular disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haematoma (Vascular disorders) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haemorrhage (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemorrhagic vasculitis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 2 (2) | 5 (5) | 11 (12) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertensive crisis (Vascular disorders) | 4 (6) | 0 (0) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertensive emergency (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertensive urgency (Vascular disorders) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 4 (4) | 2 (2) | 10 (10) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypovolaemic shock (Vascular disorders) | 1 (1) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Iliac artery occlusion (Vascular disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Iliac artery rupture (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Iliac artery stenosis (Vascular disorders) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intermittent claudication (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Leriche syndrome (Vascular disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Orthostatic hypotension (Vascular disorders) | 5 (5) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peripheral arterial occlusive disease (Vascular disorders) | 16 (19) | 20 (23) | 22 (25) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peripheral artery aneurysm (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peripheral artery occlusion (Vascular disorders) | 3 (4) | 3 (3) | 8 (9) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Peripheral artery stenosis (Vascular disorders) | 1 (1) | 5 (7) | 5 (5) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peripheral artery thrombosis (Vascular disorders) | 3 (3) | 2 (2) | 4 (4) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peripheral embolism (Vascular disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peripheral ischaemia (Vascular disorders) | 17 (18) | 13 (18) | 10 (10) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peripheral vascular disorder (Vascular disorders) | 4 (4) | 3 (5) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peripheral venous disease (Vascular disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Shock haemorrhagic (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Subclavian artery occlusion (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Subclavian artery stenosis (Vascular disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thrombosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Varicose ulceration (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Varicose vein (Vascular disorders) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Venous thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Venous thrombosis limb (Vascular disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ertugliflozin 5 mg (Overall Cardiovascular Study) (N=2746) | Ertugliflozin 15 mg (Overall Cardiovascular Study) (N=2747) | Placebo (Overall Cardiovascular Study) (N=2745) | Ertugliflozin 5 mg (Insulin +/- Metformin Sub-study) (N=348) | Ertugliflozin 15 mg (Insulin +/- Metformin Glycemic Sub-study) (N=370) | Placebo (Insulin +/- Metformin Glycemic Sub-study) (N=347) | Ertugliflozin 5 mg (Sulfonylurea Monotherapy Glycemic Sub-Study) (N=55) | Ertugliflozin 15 mg (Sulfonylurea Monotherapy Glycemic Sub-Study) (N=54) | Placebo (Sulfonylurea Monotherapy Glycemic Sub-Study) (N=48) | Ertugliflozin 5 mg (Metformin With Sulfonylurea Glycemic Sub-study) (N=100) | Ertugliflozin 15 mg (Metformin With Sulfonylurea Glycemic Sub-study) (N=113) | Placebo (Metformin With Sulfonylurea Glycemic Sub-study) (N=117)
Diarrhoea (Gastrointestinal disorders) | 132 (163) | 138 (161) | 126 (153) | 7 (7) | 9 (11) | 8 (8) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 3 (3) | 0 (0)
Nasopharyngitis (Infections and infestations) | 178 (249) | 204 (272) | 186 (244) | 4 (4) | 13 (13) | 11 (12) | 1 (1) | 0 (0) | 2 (4) | 2 (2) | 5 (5) | 3 (3)
Upper respiratory tract infection (Infections and infestations) | 197 (277) | 177 (257) | 203 (324) | 8 (8) | 10 (11) | 9 (9) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 2 (2) | 4 (4)
Urinary tract infection (Infections and infestations) | 256 (378) | 262 (354) | 211 (301) | 8 (8) | 9 (10) | 7 (7) | 1 (2) | 1 (1) | 0 (0) | 1 (1) | 4 (5) | 3 (4)
Hyperglycaemia (Metabolism and nutrition disorders) | 106 (158) | 96 (201) | 178 (283) | 5 (7) | 9 (13) | 6 (7) | 0 (0) | 0 (0) | 2 (2) | 3 (3) | 2 (2) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 883 (10056) | 854 (9474) | 884 (11591) | 101 (400) | 112 (541) | 109 (559) | 3 (4) | 3 (3) | 0 (0) | 13 (23) | 19 (110) | 14 (49)
Back pain (Musculoskeletal and connective tissue disorders) | 133 (144) | 138 (157) | 143 (160) | 2 (2) | 2 (2) | 2 (2) | 2 (2) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 2 (2)
Dizziness (Nervous system disorders) | 139 (174) | 141 (179) | 89 (107) | 8 (8) | 9 (10) | 4 (4) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 4 (4) | 1 (1)
Hypertension (Vascular disorders) | 133 (218) | 148 (272) | 168 (343) | 5 (5) | 4 (4) | 2 (2) | 2 (2) | 0 (0) | 2 (2) | 4 (4) | 2 (2) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Investigator will provide manuscripts, abstracts, or the full text of any other intended disclosure to the sponsor at least 30 days before they are submitted for publication or otherwise disclosed. If any patent action is required to protect intellectual property rights, investigator agrees to delay the disclosure for an additional 60 days. Investigator will, on request, remove any previously undisclosed Confidential Information (other than the Study results themselves) before disclosure.

DOCUMENTS (2):
  • Study Protocol (2016-03-11): https://cdn.clinicaltrials.gov/large-docs/81/NCT01986881/Prot_000.pdf
  • Statistical Analysis Plan (2020-03-20): https://cdn.clinicaltrials.gov/large-docs/81/NCT01986881/SAP_001.pdf